Comparative effectiveness of tirzepatide vs sitagliptin in individuals at cardiovascular risk

NCT07203677

15<sup>th</sup> October 2025

# 1. Title Page

| Title | Comparative effectiveness of tirzepatide vs |
|---|---|
| Title | |
| December working & Objectives | sitagliptin in individuals at cardiovascular risk. |
| Research question & Objectives | The aim of this study is to assess the |
| | comparative effectiveness of tirzepatide vs |
| | sitagliptin in preventing atherosclerotic |
| | cardiovascular events in patients with type 2 |
| | diabetes and atherosclerotic cardiovascular |
| | disease. |
| Protocol version | Version 2 |
| Last update date | October 15, 2025 |
| Contributors | Primary investigators contact information: |
| | Dr. Nils Krüger, nkruger1@bwh.harvard.edu |
| | Dr. Shirley Wang, swang1@bwh.harvard.edu |
| | Contributor names: |
| | Dr. Krüger implemented the study design in the |
| | Aetion Evidence Platform. He is responsible for |
| | the validity of the design and analytic choices. |
| | All implementation steps are recorded and the |
| | implementation history is archived in the |
| | platform. |
| Study registration | Site: ClinicalTrials.gov and Open Science |
| | Framework |
| | Identifier: NCT07203677, osf.io/zmfke |
| Sponsor | Organization: N/A |
| • | Contact: N/A |
| Conflict of interest | Dr. Krüger has no conflict of interest. |
| | Dr. Wang has consulted for Cytel Incs, Exponent |
| | Inc, and MITRE an FFRDC for Centers for |
| | Medicare and Medicaid for unrelated work. |

## **Table of contents**

| Title Page | 1 |
|---|---|
| 2. Abstract | 4 |
| 3. Amendments and updates | 4 |
| 1. Rationale and background | 5 |
| 5. Research question and objectives | 5 |
| Table 2. Research questions and objectives | 5 |
| 5. Research methods | 7 |
| 6.1 Study design | 7 |
| 6.2 Study design diagram (Figure 1). | 8 |
| 6.3 Setting | 9 |
| 6.3.1 Context and rationale for definition of time 0 (and other primary time anchors) for entry to the study population | 9 |
| 6.3.2 Context and rationale for study inclusion criteria: | 9 |
| 6.3.3 Context and rationale for study exclusion criteria | 9 |
| 6.4 Variables | 9 |
| 6.4.1 Context and rationale for exposure(s) of interest | 9 |
| 6.4.2 Context and rationale for outcome(s) of interest | 9 |
| 6.4.3 Context and rationale for follow-up | 10 |
| Table 1. Operational definitions of follow-up | 10 |
| 6.4.4 Context and rationale for covariates (confounding variables and effect modifiers, e.g. risk factors, comorbidities, comedications) | 11 |
| Table 2. Operational definitions of covariates | 11 |
| 6.5 Data analysis | 40 |
| 6.5.1 Context and rationale for analysis plan | 40 |
| Table 3. Analysis specification | 40 |
| Table 4. Sensitivity analyses – rationale, strengths and limitations | 42 |
| 6.6 Data sources | 43 |
| 6.6.1 Context and rationale for data sources | 43 |
| Table 5. Metadata about data sources and software | 44 |
| 6.7 Data management | 44 |
| 6.8 Quality control | 46 |
| 6.9 Study size and feasibility | 47 |
| 7. Limitation of the methods | 47 |
| 3. Protection of human subjects | 47 |

| 9. References | 47 |
|---|---|
| 10. Appendices | 49 |
| 1 Target Trial Framework, Operational Definitions, and Data Fitness Assessment | 49 |
| 2 Code algorithms | 49 |
| 3 Flowchart for cohort assembly | 49 |
| 4 1st feasibility assessment | 49 |
| 5 2nd feasibility assessment | 49 |
| 6 Balance Assessment - PS Distribution and C-Statistic | 49 |
| 7 Balance Assessment - Table 1 | 49 |

## 2. Abstract

This is a non-randomized, non-interventional study that is part of the *Randomized Controlled Trials Duplicated Using Prospective Longitudinal Insurance Claims: Applying Techniques of Epidemiology* (RCT-DUPLICATE) initiative (www.rctduplicate.org) of the Brigham and Women's Hospital, Harvard Medical School. It is intended to assess the comparative effectiveness of tirzepatide vs sitagliptin as a placebo proxy, after the pivotal RCT SURPASS-CVOT (NCT04255433) and its emulation (NCT07088718) demonstrated non-inferiority, leaving both regulators and clinical guideline committees uncertain whether to approve and recommend tirzepatide for a cardiovascular indication. This comparative effectiveness target trial described below draws from eligibility criteria from the SURPASS-CVOT trial and its emulation. Although many features of the target trial cannot be directly replicated in healthcare claims, key design features, including outcomes, exposures, and inclusion/exclusion criteria, were selected to proxy those features from the target trial. Randomization cannot be achieved in healthcare claims data but was proxied through a statistical balancing of measured covariates according to standard practice.

The database study will be a new-user active-comparative study, conducted using 2 national United States claims databases, where we compare the effect of tirzepatide vs sitagliptin in preventing atherosclerotic cardiovascular events. Clinical guidelines during the study period recommended both agents under investigation as second-line options for glucose lowering and were similarly costly.

The study will use two data sources: Optum Clinformatics and Merative MarketScan. Optum: Study period between May 13, 2022 to May 31, 2025.

MarketScan: Study period between May 13, 2022 to December 31, 2023.

# 3. Amendments and updates

| Version date | Version number | Section of protocol | Amendment or update | Reason |
|---|---|---|---|---|
| 1 | September 22,<br>2025 | | | |
| 2 | October 15,<br>2025 | 6.5.1 | Added subgroups for sex and age. | Exploratory analyses investigating potential effect measure modification by sex and age. |

## 4. Rationale and background

The purpose of this protocol is to specify the target trial assessing the comparative effectiveness of the dual glucose-dependent insulinotropic polypeptide (GIP) and glucagon-like peptide-1 receptor agonist (GLP-1-RA) tirzepatide vs the dipeptidyl peptidase-4 inhibitors (DPP4i) sitagliptin on atherosclerotic cardiovascular end points in patients with type 2 diabetes and atherosclerotic cardiovascular disease.

The GIP/GLP-1-RA tirzepatide became available on May 13, 2022, when it was approved to treat T2DM.<sup>1</sup> A year later, on November 8, 2023 tirzepatide was approved for chronic weight management in adults with obesity or overweight who also have at least one weight-related comorbid condition, such as hypertension, dyslipidemia, T2DM, obstructive sleep apnea, or CVD. On December 20 2024, tirzepatide was approved to treat moderate to severe obstructive sleep apnea (OSA) in adults with obesity, to be used in combination with a reduced-calorie diet and increased physical activity.

Sitagliptin was specifically chosen as an active comparator that could proxy for placebo because a major randomized controlled trial on cardiovascular outcomes demonstrated that it does not affect the cardiovascular outcomes under investigation.<sup>2</sup> This contrasts with other DPP4i such as saxagliptin, which has raised concerns regarding potential increased risks of heart failure, <sup>3-6</sup> and linagliptin, which is commonly prescribed for patients with renal impairment because it does not require dose modifications based on kidney function, potentially leading to increased confounding compared to sitagliptin.<sup>7,8</sup> Sodium-glucose cotransporter-2 (SGLT2) inhibitors would not be a neutral comparator, as they significantly reduce clinically important kidney events, kidney failure, and cardiovascular events.<sup>9-12</sup> Sulfonylureas (SUs), though inexpensive and widely used, are a poor comparator in cardiovascular outcome studies due to their association with hypoglycemia, weight gain, and channeling bias, as they are often prescribed to elderly, lower socioeconomic status patients with higher baseline cardiovascular risk, making direct comparisons to GLP-1-RAs less reliable.<sup>13</sup>

Due to the ongoing discussion about tirzepatide's role in preventing atherosclerotic cardiovascular events, we will focus on the end points of myocardial infarction, stroke, coronary revascularization, and unstable angina in this study. In prior emulations of the SURPASS-CVOT and SUSTAIN-6 trials using the same real-world data sources, design, and analytic infrastructure, results were benchmarked against those of the reference trials, demonstrating highly concordant results for these non-fatal atherosclerotic cardiovascular outcomes. This provided support for the ability to validly evaluate these outcomes in the present study. All-cause mortality will not be included as an end point in this study, as the emulation of SUSTAIN-6 showed divergent results for mortality that were suggestive of residual confounding and informed the development of the current protocol.

## 5. Research question and objectives

Table 2. Research questions and objectives

# A. Research questions and objectives

| Objective: | To evaluate the comparative effect of tirzepatide vs sitagliptin at preventing myocardial |
|---|---|
| | infarction in patients with type 2 diabetes and atherosclerotic cardiovascular disease when |
| | following the inclusion and exclusion criteria of the SURPASS-CVOT trial. |
| Hypothesis: | We hypothesize that tirzepatide will be superior to sitagliptin at preventing myocardial |
| | infarction in patients with type 2 diabetes and atherosclerotic cardiovascular disease. |
| Population (mention key inclusion-exclusion | Individuals aged 40 years or older with T2DM and atherosclerotic cardiovascular disease. |
| criteria): | |
| Exposure: | Tirzepatide. |
| Comparator: | Sitagliptin. |
| Outcome: | Myocardial infarction. |
| Time (when follow-up begins and ends): | 1 day after cohort entry date until the first of outcome, disenrollment, end of study period, discontinuation (45 days grace and risk window), switch between the arms, nursing home admission, 365 days after cohort entry, or start of any other GLP-1-RA. |
| Setting: | The outcome will be measured from inpatient hospitalizations. |
| Main measure of effect: | Hazard ratio. |

| Objective: | To evaluate the comparative effect of tirzepatide vs sitagliptin at preventing stroke in patients with type 2 diabetes and atherosclerotic cardiovascular disease when following the inclusion |
|---|---|
| | and exclusion criteria of the SURPASS-CVOT trial. |
| Hypothesis: | We hypothesize that tirzepatide will be superior to sitagliptin at preventing stroke in patients with type 2 diabetes and atherosclerotic cardiovascular disease. |
| Population (mention key inclusion-exclusion criteria): | Individuals aged 40 years or older with T2DM and atherosclerotic cardiovascular disease. |
| Exposure: | Tirzepatide. |
| Comparator: | Sitagliptin. |
| Outcome: | Stroke. |
| Time (when follow-up begins and ends): | 1 day after cohort entry date until the first of outcome, disenrollment, end of study period, discontinuation (45 days grace and risk window), switch between the arms, nursing home admission, 365 days after cohort entry, or start of any other GLP-1-RA. |
| Setting: | The outcome will be measured from inpatient hospitalizations. |
| Main measure of effect: | Hazard ratio. |

| Objective: | To evaluate the comparative effect of tirzepatide vs sitagliptin on the composite of myocardial infarction or stroke in patients with type 2 diabetes and atherosclerotic cardiovascular disease when following the inclusion and exclusion criteria of the SURPASS-CVOT trial. |
|---|---|
| Hypothesis: | We hypothesize that tirzepatide will be superior to sitagliptin at preventing myocardial infarction or stroke in patients with type 2 diabetes and atherosclerotic cardiovascular disease. |
| Population (mention key inclusion-exclusion criteria): | Individuals aged 40 years or older with T2DM and atherosclerotic cardiovascular disease. |
| Exposure: | Tirzepatide. |
| Comparator: | Sitagliptin. |
| Outcome: | Composite of myocardial infarction or stroke. |
| Time (when follow-up begins and ends): | 1 day after cohort entry date until the first of outcome, disenrollment, end of study period, discontinuation (45 days grace and risk window), switch between the arms, nursing home admission, 365 days after cohort entry, or start of any other GLP-1-RA. |
| Setting: | The outcome will be measured from inpatient hospitalizations. |
| Main measure of effect: | Hazard ratio. |

| Objective: | To evaluate the comparative effect of tirzepatide vs sitagliptin on the composite of myocardial infarction, stroke, coronary revascularization, or hospitalization for unstable angina in patients with type 2 diabetes and atherosclerotic cardiovascular disease when following the inclusion and exclusion criteria of the SURPASS-CVOT trial. |
|---|---|
| Hypothesis: | We hypothesize that tirzepatide will be superior to sitagliptin at preventing myocardial infarction, stroke, coronary revascularization, or hospitalization for unstable angina in patients with type 2 diabetes and atherosclerotic cardiovascular disease. |
| Population (mention key inclusion-exclusion criteria): | Individuals aged 40 years or older with T2DM and atherosclerotic cardiovascular disease. |
| Exposure: | Tirzepatide. |
| Comparator: | Sitagliptin. |
| Outcome: | Composite of myocardial infarction, stroke, coronary revascularization, or hospitalization for unstable angina. |
| Time (when follow-up begins and ends): | 1 day after cohort entry date until the first of outcome, disenrollment, end of study period, discontinuation (45 days grace and risk window), switch between the arms, nursing home admission, 365 days after cohort entry, or start of any other GLP-1-RA. |

| Setting: | The outcome will be measured from inpatient hospitalizations. |
|---|---|
| Main measure of effect: | Hazard ratio. |

## **B.** Research questions for negative controls

| Objective: | To evaluate the effect of tirzepatide vs sitagliptin on negative control outcomes, including (1) hernia and (2) lumbar radiculopathy in patients with type 2 diabetes and atherosclerotic cardiovascular disease when following the inclusion and exclusion criteria of the SURPASS-CVOT trial. |
|---|---|
| Hypothesis: | We hypothesize that tirzepatide will not have a different effect from sitagliptin. |
| Population (mention key inclusion-exclusion criteria): | Individuals aged 40 years or older with T2DM and atherosclerotic cardiovascular disease. In addition, patients will be excluded with recent hernia or lumbar radiculopathy prior to the follow-up time window (30 days) when studying the negative outcome hernia or lumbar radiculopathy, respectively. |
| Exposure: | Tirzepatide. |
| Comparator: | Sitagliptin. |
| Outcome: | Separate analyses for hernia and lumbar radiculopathy. |
| Time (when follow-up begins and ends): | 1 day after cohort entry date until the first of outcome, disenrollment, end of study period, discontinuation (45 days grace and risk window), switch between the arms, nursing home admission, 365 days after cohort entry, or start of any other GLP-1-RA. |
| Setting: | The outcome will be measured using diagnosis codes in an inpatient or outpatient setting. |
| Main measure of effect: | Hazard ratio. |

## 6. Research methods

## 6.1 Study design

Research design (e.g. cohort, case-control, etc.): New user active-comparator cohort study.

**Rationale for study design choice:** The new user active-comparator design is a powerful design that may be able to address confounding by indication. It accomplishes this, in large part, through judicious selection of an appropriate active-comparator group. While selection of an appropriate comparator in the design phase is crucial, cohort studies often require additional adjustment of measurable confounders. A common method for adjusting for confounding is via a propensity score.

## **6.2 Study design diagram** (Figure 1).

Figure 1. Exposure-based cohort entry where the cohort entry date is selected after application of exclusion criteria



### 6.3 Setting

#### 6.3.1 Context and rationale for definition of time 0 (and other primary time anchors) for entry to the study population

Time 0 in the database study was defined to emulate randomization to tirzepatide vs sitagliptin in the trial design. See appendix tables 1 and 2a for operational definitions and detailed code algorithms.

### **6.3.2** Context and rationale for study inclusion criteria:

Study inclusion criteria were defined to emulate the inclusion criteria for the trial. See appendix tables 1 and 2 for operational definitions and detailed code algorithms. A flowchart of the study cohort assembly is provided in appendix 3.

#### 6.3.3 Context and rationale for study exclusion criteria

Study exclusion criteria were defined to emulate the exclusion criteria for the trial. See appendix tables 1 and 2 for operational definitions and detailed code algorithms. A flowchart of the study cohort assembly is provided in appendix 3.

#### 6.4 Variables

#### 6.4.1 Context and rationale for exposure(s) of interest

The exposure and comparator were defined to emulate the agents compared for the trial, tirzepatide vs sitagliptin (active-comparator). See appendix tables 1 and 2 for operational definitions and detailed code algorithms.

#### Algorithm to define duration of exposure effect:

Assuming the effect of the drug lasts for 45 days after the last day's supply, we allow a 45 days gap between the dispensation (grace period) and also add 45 days at the end of the last day's supply (exposure risk window).

## 6.4.2 Context and rationale for outcome(s) of interest

The outcomes for the database study were defined to emulate the outcomes of the target trial, i.e., myocardial infarction, stroke, coronary revascularization, or unstable angina. See appendix tables 1 and 2 for operational definitions and detailed code algorithms. PPV for myocardial infarction using ICD9 codes was 94%. PPV for ischemic stroke using ICD9 codes was 95%. Both of the above ICD9 codes were mapped to ICD10. 19

Control outcomes of interest include:

- 1. Hernia (excluding patients with recent outcome prior to the follow-up time window). This is a negative control outcome where no difference in effect is expected for tirzepatide vs sitagliptin.
- 2. Lumbar radiculopathy (excluding patients with recent outcome prior to the follow-up time window). This is a negative control outcome where no difference in effect is expected for tirzepatide vs sitagliptin.

#### 6.4.3 Context and rationale for follow-up

Both on-treatment (OT) and intention-to-treat (ITT) analyses will be conducted. Adherence in clinical practice databases is expected to be much worse than in the trial, therefore the OT analysis will be the primary analysis. The OT analysis targets the relative hazard of outcomes while on treatment and may more closely emulate the effect observed in highly adherent trial participants. Both OT and ITT analyses will be conducted with up to 1-year follow-up.

**Table 1. Operational Definitions of follow-up** 

| follow-up start | Day 1 | |
|---|---|---|
| follow-up end <sup>1</sup> | Select<br>all that<br>apply | Specify |
| Date of outcome | Yes | |
| Date of death | Yes | |
| End of observation in data | Yes | Date of disenrollment. |
| <b>Day X following index date</b> (specify day) | Yes | Day 365. |
| End of study period (specify date) | Yes | Different dates for different databases (Optum: May 31, 2025; MarketScan: December 31, 2023). |
| End of exposure<br>(specify operational details,<br>e.g. stockpiling algorithm, grace<br>period) | Yes | 45 days grace window and 45 days risk window. |
| Date of add to/switch from exposure (specify algorithm) | Yes | Date of augmentation or switching from an exposure to a comparator and vice versa. |
| Other date (specify) | Yes | Censor upon nursing home admission or starting any other GLP-1-RA. |

## 6.4.4 Context and rationale for covariates (confounding variables and effect modifiers, e.g. risk factors, comorbidities, comedications)

We identified a series of covariates that were likely confounders due to being strong risk factors for the primary outcome that were associated with choice of treatment. These include demographics, disease severity related variables, comorbid conditions, comedications, frailty, healthcare utilization and markers of health seeking behaviour.

**Table 2. Operational Definitions of Covariates** 

| Characteristics | Details | Type of variable | Assessmen<br>t window | Care<br>Settings <sup>1</sup> | Code Type <sup>2</sup> | Diagnosi<br>s<br>Position <sup>3</sup> | Applied to study populations: | Measurement<br>characteristics<br>/<br>validation | Source for algorithm |
|---|---|---|---|---|---|---|---|---|---|
| Demographics | | | | | | | | | |
| Age | Cohort entry year – year of birth, (last observed value in the baseline) | Continuous | [0, 0] | n/a | n/a | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Sitagliptin | n/a | n/a |
| Gender | Male, Female<br>(last observed<br>value in the<br>baseline) | Categorical | [0, 0] | n/a | n/a | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Sitagliptin | n/a | n/a |
| Race* | White, Black,<br>Other (Asian,<br>Hispanic),<br>Missing/Unkn<br>own (last<br>observed<br>value in the<br>baseline) | Categorical | [0, 0] | n/a | n/a | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Sitagliptin | n/a | n/a |

<sup>&</sup>lt;sup>1</sup> follow-up ends at the first occurrence of any of the selected criteria that end follow-up.


| Characteristics | Details | Type of<br>variable | Assessmen<br>t window | Care<br>Settings <sup>1</sup> | Code Type <sup>2</sup> | Diagnosi<br>s<br>Position <sup>3</sup> | Applied to study populations: | Measurement<br>characteristics<br>/<br>validation | Source for algorithm |
|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | Reference:<br>Sitagliptin | | |
| Bowel obstruction | | Binary | [-365, 0] | Inpatient | ICD-10-CM | Primary | Exposure: Tirzepatide Reference: Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Gastroparesis | | Binary | [-365, 0] | Any | ICD-10-CM | Any | Exposure:<br>Tirzepatide<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Diabetes medication | ons | | | | | | | | |
| Number of antidiabetic drugs on CED | | Continuous | [0,0] | n/a | generic | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Concomitant use or initiation of metformin | | Binary | [0, 0] | n/a | generic | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Concomitant use or initiation of insulin | | Binary | [0, 0] | n/a | generic | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Concomitant use or initiation of sulfonylureas | | Binary | [0, 0] | n/a | generic | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Concomitant use or initiation of DPP4i except sitagliptin | | Binary | [0, 0] | n/a | generic | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Concomitant use or initiation of SGLT2i | | Binary | [0, 0] | n/a | generic | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |

| Characteristics | Details | Type of<br>variable | Assessmen<br>t window | Care<br>Settings <sup>1</sup> | Code Type <sup>2</sup> | Diagnosi<br>s<br>Position <sup>3</sup> | Applied to study populations: | Measurement<br>characteristics<br>/<br>validation | Source for algorithm |
|---|---|---|---|---|---|---|---|---|---|
| Concomitant use or initiation of other glucose-lowering drugs | | Binary | [0, 0] | n/a | generic | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Past use of metformin | | Binary | [-365, -1] | n/a | generic | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Past use of insulin | | Binary | [-365, -1] | n/a | generic | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Past use of sulfonylureas | | Binary | [-365, -1] | n/a | generic | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Past use of DPP4i<br>except sitagliptin | | Binary | [-365, -1] | n/a | generic | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Past use of SGLT2i | | Binary | [-365, -1] | n/a | generic | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Past use of other glucose-lowering drugs | | Binary | [-365, -1] | n/a | generic | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Heart failure medic | cations | | | | | | | | |
| ACEi / ARB | | Binary | [-365, 0] | n/a | generic | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |

| Characteristics | Details | Type of variable | Assessmen<br>t window | Care<br>Settings <sup>1</sup> | Code Type <sup>2</sup> | Diagnosi<br>s<br>Position <sup>3</sup> | Applied to study populations: | Measurement characteristics / validation | Source for algorithm |
|---|---|---|---|---|---|---|---|---|---|
| ARNI | | Binary | [-365, 0] | n/a | generic | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Thiazides | | Binary | [-365, 0] | n/a | generic | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Beta-blockers | | Binary | [-365, 0] | n/a | generic | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Calcium channel<br>blockers | | Binary | [-365, 0] | n/a | generic | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Digoxin / Digitoxin | | Binary | [-365, 0] | n/a | generic | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Loop diuretics | | Binary | [-365, 0] | n/a | generic | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Other diuretics | | Binary | [-365, 0] | n/a | generic | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Intravenous diuretics | | Binary | [-365, 0] | n/a | generic | n/a | Exposure: Tirzepatide Reference: Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Nitrates | | Binary | [-365, 0] | n/a | generic | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |

| Characteristics | Details | Type of<br>variable | Assessmen<br>t window | Care<br>Settings <sup>1</sup> | Code Type <sup>2</sup> | Diagnosi<br>s<br>Position <sup>3</sup> | Applied to study populations: | Measurement<br>characteristics<br>/<br>validation | Source for algorithm |
|---|---|---|---|---|---|---|---|---|---|
| Other medications | | | | | | | | | |
| Anti-arrhythmics | | Binary | [-365, 0] | n/a | generic | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Statins | | Binary | [-365, 0] | n/a | generic | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| PCSK9 inhibitors<br>and other<br>lipid-lowering<br>drugs | | Binary | [-365, 0] | n/a | generic | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Antiplatelet agents | | Binary | [-365, 0] | n/a | generic | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Oral<br>anticoagulants | | Binary | [-365, 0] | n/a | generic | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| COPD/Asthma<br>medication | | Binary | [-365, 0] | n/a | generic | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| NSAIDs | | Binary | [-365, 0] | n/a | generic | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Oral corticosteroids | | Binary | [-365, 0] | n/a | generic | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |

| Characteristics | Details | Type of variable | Assessmen<br>t window | Care<br>Settings <sup>1</sup> | Code Type <sup>2</sup> | Diagnosi<br>s<br>Position <sup>3</sup> | Applied to study populations: | Measurement characteristics / validation | Source for algorithm |
|---|---|---|---|---|---|---|---|---|---|
| Osteoporosis<br>agents (incl.<br>bisphosphonates) | | Binary | [-365, 0] | n/a | generic | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Opioids | | Binary | [-365, 0] | n/a | generic | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Anti-depressants | | Binary | [-365, 0] | n/a | generic | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Antipsychotics | | Binary | [-365, 0] | n/a | generic | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Anxiolytics/hypnot ics, benzodiazepines | | Binary | [-365, 0] | n/a | generic | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Medication for dementia | | Binary | [-365, 0] | n/a | generic | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Urinary tract infections antibiotics | | Binary | [-365, 0] | n/a | generic | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Laxatives | | Binary | [-365, 0] | n/a | generic | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Healthcare utilizat | ion markers | | | | | | | | |
| Number of distinct medications, | | Continuous | [-365, 0] | n/a | n/a | n/a | Exposure:<br>Tirzepatide | n/a | Appendix,<br>Covariate –<br>Algorithm |

| Characteristics | Details | Type of<br>variable | Assessmen<br>t window | Care<br>Settings <sup>1</sup> | Code Type <sup>2</sup> | Diagnosi<br>s<br>Position <sup>3</sup> | Applied to study populations: | Measurement<br>characteristics<br>/<br>validation | Source for algorithm |
|---|---|---|---|---|---|---|---|---|---|
| median (iqr), mean<br>(sd) | | | | | | | Reference:<br>Sitagliptin | | |
| Number of office<br>visits, median (iqr),<br>mean (sd) | | Continuous | [-365, 0] | n/a | n/a | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Number of<br>endocrinologist<br>visits, median (iqr),<br>mean (sd) | | Continuous | [-365, 0] | n/a | n/a | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Number of<br>cardiologist visits,<br>median (iqr), mean<br>(sd) | | Continuous | [-365, 0] | n/a | n/a | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Number of internal<br>medicine/family<br>medicine visits,<br>median (iqr), mean<br>(sd) | | Continuous | [-365, 0] | n/a | n/a | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Number of<br>Electrocardiogram<br>s, median (iqr),<br>mean (sd) | | Continuous | [-365, 0] | n/a | n/a | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Number of<br>Echocardiograms,<br>median (iqr), mean<br>(sd) | | Continuous | [-365, 0] | n/a | n/a | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Pharmacy<br>out-of-pocket<br>cost, median (iqr), | | Continuous | [-365, 0] | n/a | n/a | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |

| Characteristics | Details | Type of variable | Assessmen<br>t window | Care<br>Settings <sup>1</sup> | Code Type <sup>2</sup> | Diagnosi<br>s<br>Position <sup>3</sup> | Applied to study populations: | Measurement characteristics / validation | Source for algorithm |
|---|---|---|---|---|---|---|---|---|---|
| mean (sd) | | | | | | | | | |
| Unique brand<br>medications,<br>median (iqr), mean<br>(sd)** | | Continuous | [-365, 0] | n/a | n/a | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Unique generic<br>medications,<br>median (iqr), mean<br>(sd)** | | Continuous | [-365, 0] | n/a | n/a | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Ratio of unique<br>brand to generic<br>medications,<br>median (iqr), mean<br>(sd) | | Continuous | [-365, 0] | n/a | n/a | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Healthy behavior n | narkers | | | | | | | | |
| Colonoscopy /<br>Sigmoidoscopy | | Binary | [-365, 0] | Any | CPT/HCPCS | Any | Exposure:<br>Tirzepatide<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Flu vaccine /<br>Pneumococcal<br>vaccine | | Binary | [-365, 0] | Any | CPT/HCPCS | Any | Exposure:<br>Tirzepatide<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Pap smear test | | Binary | [-365, 0] | Any | CPT/HCPCS | Any | Exposure:<br>Tirzepatide<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| PSA test | | Binary | [-365, 0] | Any | CPT/HCPCS | Any | Exposure:<br>Tirzepatide<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |

| Characteristics | Details | Type of variable | Assessmen<br>t window | Care<br>Settings <sup>1</sup> | Code Type <sup>2</sup> | Diagnosi<br>s<br>Position <sup>3</sup> | Applied to study populations: | Measurement<br>characteristics<br>/<br>validation | Source for algorithm |
|---|---|---|---|---|---|---|---|---|---|
| Fecal occult blood test | | Binary | [-365, 0] | Any | CPT/HCPCS | Any | Exposure:<br>Tirzepatide<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Bone mineral density tests | | Binary | [-365, 0] | Any | CPT/HCPCS | Any | Exposure:<br>Tirzepatide<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Mammograms | | Binary | [-365, 0] | Any | CPT/HCPCS | Any | Exposure:<br>Tirzepatide<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Telemedicine | | Binary | [-365, 0] | Any | CPT/HCPCS | Any | Exposure:<br>Tirzepatide<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Laboratory and dia | gnostic tests | | | | | | | | |
| Number of HbA1c<br>tests, median (iqr),<br>mean (sd) | | Continuous | [-365, 0] | Any | CPT/HCPCS | Any | Exposure:<br>Tirzepatide<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Number of lipid<br>panels, median<br>(iqr), mean (sd) | | Continuous | [-365, 0] | Any | CPT/HCPCS | Any | Exposure:<br>Tirzepatide<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Number of<br>creatinine tests,<br>median (iqr), mean<br>(sd) | | Continuous | [-365, 0] | Any | CPT/HCPCS | Any | Exposure:<br>Tirzepatide<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Number of<br>natriuretic peptide<br>tests, median (iqr),<br>mean (sd) | | Continuous | [-365, 0] | Any | CPT/HCPCS | Any | Exposure:<br>Tirzepatide<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |

| Characteristics | Details | Type of variable | Assessmen<br>t window | Care<br>Settings <sup>1</sup> | Code Type <sup>2</sup> | Diagnosi<br>s<br>Position <sup>3</sup> | Applied to study populations: | Measurement characteristics / validation | Source for algorithm |
|---|---|---|---|---|---|---|---|---|---|
| Number of urine<br>tests, median (iqr),<br>mean (sd) | | Continuous | [-365, 0] | Any | CPT/HCPCS | Any | Exposure:<br>Tirzepatide<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Lab values | | | | | | | | | |
| HbA1c** | | Continuous | [-365, 0] | n/a | n/a | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Glucose** | | Continuous | [-365, 0] | n/a | n/a | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Creatinine** | | Continuous | [-365, 0] | n/a | n/a | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Systolic blood pressure** | | Continuous | [-365, 0] | n/a | n/a | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Heart rate** | | Continuous | [-365, 0] | n/a | n/a | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| BMI** | | Continuous | [-365, 0] | n/a | n/a | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| eGFR** | | Continuous | [-365, 0] | n/a | n/a | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| LDL** (mg/dl;<br>mean, sd) | | Continuous | [-365, 0] | n/a | n/a | n/a | Exposure:<br>Tirzepatide | n/a | Appendix,<br>Covariate –<br>Algorithm |

| Characteristics | Details | Type of variable | Assessmen<br>t window | Care<br>Settings <sup>1</sup> | Code Type <sup>2</sup> | Diagnosi<br>s<br>Position <sup>3</sup> | Applied to study populations: | Measurement<br>characteristics<br>/<br>validation | Source for algorithm |
|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | Reference:<br>Sitagliptin | | |
| HDL** (mg/dl;<br>mean, sd) | | Continuous | [-365, 0] | n/a | n/a | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Total cholesterol**<br>(mg/dl; mean, sd) | | Continuous | [-365, 0] | n/a | n/a | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Triglyceride**<br>(mg/dl; mean, sd) | | Continuous | [-365, 0] | n/a | n/a | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Burden of comorbi | dities | | | | | | | | |
| Combined comorbidity score | | Continuous | [-365, 0] | Any | ICD10-CM | Any | Exposure:<br>Tirzepatide<br>Reference:<br>Sitagliptin | n/a | Gagne et al.,<br>Sun et al. <sup>20,21</sup> |
| Frailty score | | Continuous | [-365, 0] | Any | ICD10-CM | Any | Exposure:<br>Tirzepatide<br>Reference:<br>Sitagliptin | n/a | Kim et al. <sup>22</sup> |
| Baseline hospitaliz | ations and hospit | al metrics | | | | | | | |
| Number of any<br>hospitalization,<br>median (iqr), mean<br>(sd) | | Continuous | [-365, 0] | n/a | n/a | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Any hospitalization<br>within prior 91<br>days; n (%) | | Binary | [-91, 0] | n/a | n/a | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |

| Characteristics | Details | Type of variable | Assessmen<br>t window | Care<br>Settings <sup>1</sup> | Code Type <sup>2</sup> | Diagnosi<br>s<br>Position <sup>3</sup> | Applied to study populations: | Measurement characteristics / validation | Source for algorithm |
|---|---|---|---|---|---|---|---|---|---|
| Any hospitalization<br>within prior<br>92-365 days; n (%) | | Binary | [-365, -92] | n/a | n/a | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| 0, 1, >1<br>hospitalizations<br>(any) | | Continuous | [-365, 0] | n/a | n/a | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Hospitalization for heart failure | | Binary | [-365, 0] | n/a | n/a | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Emergency<br>department visits | | Binary | [-365, 0] | n/a | n/a | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Sitagliptin | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Calendar year of co | hort entry | | | | | | | | |
| 2022 | | Categorical | [0, 0] | n/a | n/a | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Sitagliptin | n/a | n/a |
| 2023 | | Categorical | [0, 0] | n/a | n/a | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Sitagliptin | n/a | n/a |
| 2024 | | Categorical | [0, 0] | n/a | n/a | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Sitagliptin | n/a | n/a |
| 2025 | | Categorical | [0, 0] | n/a | n/a | n/a | Exposure: Tirzepatide Reference: Sitagliptin | n/a | n/a |

 $<sup>^{1}</sup>$ IP = inpatient, OP = outpatient, ED = emergency department, OT = other, n/a = not applicable

<sup>&</sup>lt;sup>2</sup>See appendix for listing of clinical codes for each study parameter
<sup>3</sup>Specify whether a diagnosis code is required to be in the primary position (main reason for encounter)

## 6.5 Data analysis

#### **6.5.1** Context and rationale for analysis plan

The study will use a propensity score based overlap weighting method. The propensity score will be estimated as the probability of initiating tirzepatide vs sitagliptin given the baseline patient characteristics using multivariable logistic regression models. As diagnostics for PS models, the study will evaluate distributional covariate balance using standardized differences and c-statistics post-matching. The study will estimate the hazard ratio for tirzepatide vs sitagliptin in preventing atherosclerotic cardiovascular events in the weighted population using a Cox proportional hazards model with robust standard errors.

## **Table 3. Analysis specification**

### A. Analyses

| Hypothesis: | Tirzepatide does not increase the risk of myocardial infarction in patients with T2DM and an established CVD |
|---|---|
| | when following the eligibility criteria of the SURPASS-CVOT trial. |
| Exposure contrast: | Tirzepatide vs sitagliptin. |
| Outcome: | Myocardial infarction. |
| Analytic software: | Aetion, SAS 9.4, R.4.4.0, Python 3.13.3 |
| Model(s): | Outcome model: Cox proportional hazards |
| (provide details or code) | Follow-up time * status(0) = exposure |
| Confounding adjustment method | Name method and provide relevant details, e.g. bivariate, multivariable, propensity score weighting (specify weighting algorithm ratio and caliper), propensity score weighting (specify weight formula, trimming, truncation), propensity score stratification (specify strata definition), other. |
| | Overlap weighting based on the propensity score. |
| Missing data methods | Name method and provide relevant details, e.g. missing indicators, complete case, last value carried forward, multiple imputation (specify model/variables), other. |
| | Assumption that if no relevant claims diagnoses/procedures are present, the condition is not present. |
| Subgroup Analyses | List all subgroups |
| | Individuals <70, Individuals ≥70, Male, Female (exploratory analyses). |

<sup>\*</sup>Available for Optum Clinformatics and Medicare

<sup>\*\*</sup>Not used in the PS model

| Hypothesis: | Tirzepatide does not increase the risk of stroke in patients with T2DM and an established CVD when following the eligibility criteria of the SURPASS-CVOT trial. |
|---|---|
| Exposure contrast: | Tirzepatide vs sitagliptin. |
| Outcome: | Stroke. |
| Analytic software: | Aetion, SAS 9.4, R.4.4.0, Python 3.13.3 |
| Model(s): | Outcome model: Cox proportional hazards |
| (provide details or code) | Follow-up time * status(0) = exposure |
| Confounding adjustment method | Name method and provide relevant details, e.g. bivariate, multivariable, propensity score weighting (specify weighting algorithm ratio and caliper), propensity score weighting (specify weight formula, trimming, truncation), propensity score stratification (specify strata definition), other. |
| | Overlap weighting based on the propensity score. |
| Missing data methods | Name method and provide relevant details, e.g. missing indicators, complete case, last value carried forward, multiple |
| wildsing data methods | imputation (specify model/variables), other. |
| iviissing data methods | |
| Subgroup Analyses | imputation (specify model/variables), other. |

| Hypothesis: | Tirzepatide does not increase the risk of a composite of myocardial infarction or stroke in patients with T2DM |
|---|---|
| | and an established CVD when following the eligibility criteria of the SURPASS-CVOT trial. |
| Exposure contrast: | Tirzepatide vs sitagliptin. |
| Outcome: | Composite of myocardial infarction or stroke. |
| Analytic software: | Aetion, SAS 9.4, R.4.4.0, Python 3.13.3 |
| Model(s): | Outcome model: Cox proportional hazards |
| (provide details or code) | Follow-up time * status(0) = exposure |
| Confounding adjustment method | Name method and provide relevant details, e.g. bivariate, multivariable, propensity score weighting (specify weighting |
| | algorithm ratio and caliper), propensity score weighting (specify weight formula, trimming, truncation), propensity score stratification (specify strata definition), other. |
| | Overlap weighting based on the propensity score. |
| Missing data methods | Name method and provide relevant details, e.g. missing indicators, complete case, last value carried forward, multiple imputation (specify model/variables), other. |
| | Assumption that if no relevant claims diagnoses/procedures are present, the condition is not present. |
| Subgroup Analyses | List all subgroups |
| | Individuals <70, Individuals ≥70, Male, Female (exploratory analyses). |

| Hypothesis: | Tirzepatide does not increase the risk of a composite of myocardial infarction, stroke, coronary |
|---|---|
| | revascularization, or instable angina in patients with T2DM and an established CVD when following the eligibility criteria of the SURPASS-CVOT trial. |
| Exposure contrast: | Tirzepatide vs sitagliptin. |
| Outcome: | Composite of myocardial infarction, stroke, coronary revascularization, or instable angina. |
| Analytic software: | Aetion, SAS 9.4, R.4.4.0, Python 3.13.3 |
| Model(s): | Outcome model: Cox proportional hazards |
| (provide details or code) | Follow-up time * status(0) = exposure |
| Confounding adjustment method | Name method and provide relevant details, e.g. bivariate, multivariable, propensity score weighting (specify weighting |
| | algorithm ratio and caliper), propensity score weighting (specify weight formula, trimming, truncation), propensity score stratification (specify strata definition), other. |
| | Overlap weighting based on the propensity score. |
| Missing data methods | Name method and provide relevant details, e.g. missing indicators, complete case, last value carried forward, multiple |
| | imputation (specify model/variables), other. |
| | Assumption that if no relevant claims diagnoses/procedures are present, the condition is not present. |
| Subgroup Analyses | List all subgroups |
| | Individuals <70, Individuals ≥70, Male, Female (exploratory analyses). |

# **B.** Negative Control Analyses

| Hypothesis: | Tirzepatide vs sitagliptin has no effect on risk of negative control outcomes compared to sitagliptin. Negative |
|---|---|
| | control outcomes include (1) hernia and (2) lumbar radiculopathy. |
| Exposure contrast: | Tirzepatide vs sitagliptin. |
| Outcome: | Separate analyses for each negative control outcome, including hernia and lumbar radiculopathy |
| Analytic software: | Aetion, SAS 9.4, R.4.4.0, Python 3.13.3 |
| Model(s): | Outcome model: Cox proportional hazards |
| (provide details or code) | Follow-up time*status(0) = exposure |
| Confounding adjustment method | Name method and provide relevant details, e.g. bivariate, multivariable, propensity score weighting (specify weighting algorithm ratio and caliper), propensity score weighting (specify weight formula, trimming, truncation), propensity score stratification (specify strata definition), other. |
| | Overlap weighting based on the propensity score. |
| Missing data methods | Name method and provide relevant details, e.g. missing indicators, complete case, last value carried forward, multiple imputation (specify model/variables), other. |
| | Assumption that if no relevant claims diagnoses/procedures are present, the condition is not present. |
| Subgroup Analyses | List all subgroups |
| | N/A. |
**Table 4. Sensitivity analyses – rationale, strengths and limitations** 

| | What is being varied? How? | Why?<br>(What do you expect to<br>learn?) | Strengths of the sensitivity analysis compared to the primary | Limitations of the sensitivity analysis compared to the primary |
|---|---|---|---|---|
| Negative control<br>outcomes,<br>including hernia,<br>lumbar<br>radiculopathy | We evaluate negative control outcomes of hernia and lumbar radiculopathy, where no causal effect is expected from tirzepatide, or sitagliptin. | We will evaluate the potential impact of residual confounding on this outcome for which there is not expected to be a causal effect | The evaluates the robustness of the interpretation of the primary analysis by evaluating the potential magnitude of unmeasured confounding | This analysis assumes that the confounding structure is the same or similar for the negative control outcome as the outcome of interest |
| Accounting for the competing event of death. | We will account for the competing event of death in our primary outcome model by using the Fine-Gray method. | To assess the impact of the competing event of death on the primary end point. | Accounts for the fact that death is a competing event, yielding clinically relevant cumulative incidence estimates and avoiding bias from treating death as non-informative censoring. | Targets a slightly different estimand than Cox, may have lower power, and interpretation can be difficult if treatment also affects death or confounding affects death differently than the primary end point. |
| As-started analyses (observational analogue to intention-to-treat) to address potential informative censoring. | To address potential informative censoring. | We will consider the first-used medication for 365 days without considering drug discontinuation or switching, mimicking an "intention-to-treat" approach. | Reflects follow-up regimen of RCT. | Persistence of drug use is shorter in clinical practice whereas adherence is typically higher in RCTs. Therefore, we expect the estimated effects will be diluted toward the null, underestimating the true treatment effect had patients remained on therapy. |

### **6.6 Data sources**

#### **6.6.1** Context and rationale for data sources

**Reason for selection:** The study will be conducted in 2 US health care claims databases: Optum Clinformatics (2022-2025), and Merative MarketScan (2022-2023). Data from the Merative MarketScan database will only be included if sufficient sample size can be accrued.

**Strengths of data source(s):** Each data source contains deidentified, longitudinal, date-stamped information on patient enrollment, demographics, inpatient/outpatient diagnosis and procedures, admission and discharge dates, and medication dispensation. The death data is captured in the Optum database from inpatient discharge status, social security death master file, and deaths scraped from obituaries or other sources. The death data in MarketScan is captured from the social security death master file and inpatient discharge status. It is recognized that the social security death master file has high specificity and positive predictive value for deaths. While this data resource has under captured deaths since 2011, the capture of deaths is not expected to be differential between compared exposure groups.

Limitations of data source(s): Patient healthcare encounters are only observable when they are enrolled in an insurance plan that contributes to the database. Patients may change insurance plans for multiple reasons. Both Optum Clinformatics and Merative MarketScan are primarily employer based insurance databases where patients may disenroll with job changes. In claims data, dispensing data for inpatient medication is unavailable. Diagnoses reflect billing practices, therefore algorithms (preferably validated) are needed for accurate phenotyping of patient conditions. Services that are not covered by insurance do not appear in the data. The trial evaluated cardiovascular deaths, however we will evaluate all-cause mortality in the emulation because most deaths in this cohort of patients at high cardiovascular risk will be related to cardiovascular reasons, the cause of death is not recorded for databases not linked to NDI, and the performance of NDI at identifying cardiovascular causes of death may be suboptimal. <sup>23</sup>

#### **Data source provenance/curation:**

Information about Optum Clinformatics and Merative MarketScan can be found in data dictionaries and user guides that are provided to clients.

Table 5. Metadata about data sources and software

| | Data 1 | Data 2 |
|---|---|---|
| Data Source(s): | Optum Clinformatics | Merative MarketScan |
| Study Period: | 13 <sup>th</sup> May 2022 | 13 <sup>th</sup> May 2022 |
| Eligible Cohort Entry Period: | May 31, 2025 | December 31, 2023 |
| Data Version (or date of last update): | April 2025 | Mortality Cut Set A<br>Received 2024-03-01 |
| Data sampling/extraction criteria: | n/a | n/a |
| Type(s) of data: | Administrative claims | Administrative claims |
| Data linkage: | n/a | n/a |
| Conversion to CDM*: | n/a | n/a |

Software for data management:

| Aetion Evidence Platform® | Aetion Evidence Platform® |
|---------------------------|---------------------------|
| (2025) | (2025) |

\*CDM = Common Data Model

#### **6.7 Data management**

<u>Tracking data:</u> The Data Use Agreement (DUA) Custodian (Principal Investigator) and the Division Operations Manager (Winta Tekle) are responsible for receiving and creating a record of new data associated with the given request. The Operations Manager is responsible for all indexing and archiving of documents and electronic media related to data that the Division receives and will log data location, data contents, and associated DUA and Institutional Review Board (IRB) numbers in the Division's centralized tracking system.

<u>Handling and storage:</u> In-scope data will be stored utilizing Mass General Brigham approved information systems – i.e., Division servers and Mass General Brigham network storage.

<u>Archiving</u>: Data retention and any removal will be executed by the Division Operations Manager (Winta Tekle) and Data Manager (Todd MacGarvey). The Division follows Mass General Brigham enterprise record retention policies and follow the terms of the agreement through which the in-scope data was received.

Information security: The Division follows Mass General Brigham's Enterprise Information Security Program (EISP). The EISP helps by providing assurance that Mass General Brigham information and information systems are protected from unauthorized access, use, disclosure, duplication, modification, or destruction in order to maintain their confidentiality, integrity, and availability. To that end, the EISP policies, standards and procedures create an information security framework that is aligned with the recommendations of the International Organization for Standardization's (ISO) publication 27001 and the National Institute of Standards and Technology's (NIST) publication 800-53 Family of Controls and MGB regulatory and legal requirements (as a HIPAA covered entity).

Mass General Brigham workforce members are required to complete new workforce privacy and information security training upon hire and annually thereafter. Refresh training is provided as appropriate. Mass General Brigham workforce members are required to review and sign a Confidentiality Agreement upon hire and annually thereafter. Additionally, we follow Enterprise Information Security and Privacy policies, including Managing Workforce Members Information Security Responsibilities Policy, which was developed to help assure that Mass General Brigham workforce members are competent and eligible to support the information security responsibilities associated with their role. Mass General Brigham workforce, including Division staff, are required to comply with Enterprise Information Security and Privacy Policies.

<u>Facilities:</u> The research team uses a highly secure, state-of-the-art, computing facility housed at Mass General Brigham's Corporate Data Centers in Needham and Marlborough, Massachusetts as well as Amazon Web Services (AWS). We maintain redundant storage for maximal data integrity and high-speed data access.

The Division uses Mass General Brigham corporate provisioned servers to analyze and store data in connection with this project. There are strict access controls enforced by technical means to ensure that only study staff who have been approved to conduct data analyses and contracted data engineers

are able to access data (e.g., Mass General Brigham Authentication (Active Directory) utilized; auditing, logging, and monitoring enabled; firewalls enabled; etc.). All Division servers used in this study are accessible to only authorized staff only through the MGB network and utilizing VPN as appropriate (i.e., users must be on the network and logged into VPN to access). Mass General Brigham has a network information security monitoring team and in-scope servers are enrolled in enterprise security tools (e.g., vulnerability scanning service, antivirus, etc.).

The Division also uses AWS. In-scope AWS services / resources have undergone review and assessment by Mass General Brigham's Information Security Risk Assessment Team/ InfoSec Risk Management Team as required and in alignment with NIST 800-30: Guide for Conducting Risk Assessments. In-scope AWS servers are for our exclusive use (reserved instances), are covered under our organization's Business Associate Agreement with AWS. In-scope servers are housed in anonymous facilities that are not branded as AWS facilities. Physical access is strictly controlled both at the perimeter and at building ingress points by professional security staff utilizing video surveillance, intrusion detection systems, and other electronic means.

Security attributes and controls for the Division's use of in-scope AWS in connection with this project include: encryption at rest and in transit (industry standard AES-256 encryption, SSL/TSL), anti-malware, latest OS updates and patches as well as anti-virus; multi-factor authentication (MFA), Identity and Access Management, including SSO; auditing and logging; principle of least privilege, including for traffic and ports (e.g., deny all default configurations), use of VPC enabled Step functions, etc.; separation between environments; minimum necessary (out of the box AWS roles are not used as they can be overly permissive); all data would reside in the US domestic regions – use only US east HIPAA compliant region; performance monitoring enabled and reviewed as per internal processes; passwords compliant with enterprise password policy and, as appropriate, more protective password requirements; etc. Our Division's AWS use is also subject to ongoing evaluation and monitoring as well – e.g., vulnerability scanning and management, access review, etc.

A data file list will be maintained in Amazon S3 and tracked through Cloudtrail and Cloudwatch. Reporting of data file availability for any file stored in an S3 bucket will be controlled by MGB.

Amazon EC2, Amazon EBS, and Amazon VPC are integrated with AWS CloudTrail, a service that provides a record of actions taken by a user, role, or an AWS service in Amazon EC2, Amazon EBS, and Amazon VPC. CloudTrail captures all API calls for Amazon EC2, Amazon EBS, and Amazon VPC as events, including calls from the console and from code calls to the APIs. MGB IT/security staff have full access to CloudTrail to ensure that CloudTrail monitoring is available at all times. Amazon CloudWatch Events delivers a near-real-time stream of system events that describe changes in AWS resources. Amazon CloudTrail can log, continuously monitor, and retain account activity related to actions across the MGB AWS infrastructure. CloudTrail provides event history of MGB AWS account activity. This event history simplifies security analysis, resource change tracking, and troubleshooting and complies with requirements to ensure the data file inventory is controlled by MGB.

<u>Backups</u>: Backups are created using industry recognized Cryptographic mechanisms (e.g., 256-bit AES encryption) as appropriate and required. Data are backed up within the MGB network from the MGB Needham data center to the MGB Marlborough data center via replication/mirroring and volume-level snapshots. AWS Backup supports both instance-level backups as Amazon Machine Images (AMIs) and volume-level backups as separate snapshots based on the resource tags. AMIs allow MGB IT and security staff to create backups of all S3 and EC2 instances.

In addition to the safeguards listed above, the Division follows enterprise privacy and information security policies and maintains internally procedures in connection with this project to safeguard the data in connection with this project as appropriate and required including: Physical Security and

Environmental Controls for Electronic Information Policy; IT Access Control Standards for Users policy; Safeguarding Fax Copiers Printers Telephone Use and Pagers; Physical Removal and Transport of Protected Health Information and Personal Information policy, etc.

### 6.8 Quality control

Senior Programmers and Research Specialists perform QA/QC on raw or common data model converted data via SAS/R/Aetion software. The protocol will be iteratively developed and pre-specified data checks including feasibility counts and balance on baseline covariates will be conducted with outputs reviewed by MGB team members. Team members will review code lists to ensure fidelity to intended algorithms.

#### 6.9 Study size and feasibility

See appendix 4 and appendix 5 (feasibility, weighting on age, sex, comorbidity score as well as all predefined propensity score variables). Propensity score distribution plots with c-statistics are available in appendix 6. Table 1 showing prevalence of baseline characteristics and standardized differences in distribution are available in appendix 7. Additional diagnostic evaluations, including balance assessments of laboratory and clinical examination test results not included in the propensity score as well as assessment of heart failure-related medication after follow-up, will be conducted to assess potential residual confounding and divergence of treatment over time.

#### 7. Limitation of the methods

As we are using secondary data and the data were not collected for research purposes, some important variables may not be collected or will be measured imperfectly. We have selected validated algorithms when possible and we have created proxies for important variables that are not directly captured in the data to reduce confounding by unmeasured factors.

When comparing results from an RCT to a database study that emulates the design, we assume that the findings from the single RCT are internally valid.

Although we plan to emulate the important features of each trial as closely as possible in healthcare claims, there may be some elements of the RCT design that are not emulable with a database study, which means that the real-world evidence obtained from the database study and trial will address slightly different clinical questions. For example, in routine clinical care, adherence to treatment is typically not as high as it is in an RCT with strong measures in place to encourage adherence to the study protocol. This means that there is more discontinuation and short-term medication use in the patients identified in claims databases than trial participants.

Apparent agreement between RCT and database study results could occur if the effects of multiple factors (chance, emulation differences, bias) cancel each other out.

# 8. Protection of human subjects

This study has been approved by the Brigham and Women's Hospital Institutional Review Board.

## 9. References

- 1. FDA approves Lilly's Mounjaro™ (tirzepatide) injection, the first and only GIP and GLP-1 receptor agonist for the treatment of adults with type 2 diabetes | Eli Lilly and Company. Accessed July 18, 2025. https://investor.lilly.com/news-releases/news-release-details/fda-approves-lillys-mounjarotm-tirzepatide-injection-first-and
- 2. Green JB, Bethel MA, Armstrong PW, et al. Effect of Sitagliptin on Cardiovascular Outcomes in Type 2 Diabetes. *N Engl J Med*. 2015;373(3):232-242. doi:10.1056/NEJMoa1501352
- 3. Scirica BM, Bhatt DL, Braunwald E, et al. Saxagliptin and Cardiovascular Outcomes in Patients with Type 2 Diabetes Mellitus. *N Engl J Med*. 2013;369(14):1317-1326. doi:10.1056/NEJMoa1307684
- 4. Heart Failure, Saxagliptin, and Diabetes Mellitus: Observations from the SAVOR-TIMI 53 Randomized Trial. doi:10.1161/CIRCULATIONAHA.114.010389
- 5. A Multicenter Observational Study of Incretin-based Drugs and Heart Failure | New England Journal of Medicine. Accessed December 2, 2024. https://www-nejm-org.emedien.ub.uni-muenchen.de/doi/10.1056/NEJMoa1506115
- 6. Risk for Hospitalized Heart Failure Among New Users of Saxagliptin, Sitagliptin, and Other Antihyperglycemic Drugs: A Retrospective Cohort Study: Annals of Internal Medicine: Vol 164, No 11. Accessed December 2, 2024. https://www.acpjournals.org/doi/10.7326/M15-2568
- 7. Patorno E, Gopalakrishnan C, Bartels DB, Brodovicz KG, Liu J, Schneeweiss S. Preferential prescribing and utilization trends of diabetes medications among patients with renal impairment: Emerging role of linagliptin and other dipeptidyl peptidase 4 inhibitors. *Endocrinol Diabetes Metab*. 2018;1(1):e00005. doi:10.1002/edm2.5
- 8. Gallwitz B. Safety and efficacy of linagliptin in type 2 diabetes patients with common renal and cardiovascular risk factors. *Ther Adv Endocrinol Metab*. 2013;4(3):95-105. doi:10.1177/2042018813486165
- 9. Packer M, Anker SD, Butler J, et al. Cardiovascular and Renal Outcomes with Empagliflozin in Heart Failure. *N Engl J Med*. 2020;383(15):1413-1424. doi:10.1056/NEJMoa2022190
- 10. Solomon SD, McMurray JJV, Claggett B, et al. Dapagliflozin in Heart Failure with Mildly Reduced or Preserved Ejection Fraction. *N Engl J Med*. 2022;387(12):1089-1098. doi:10.1056/NEJMoa2206286
- 11. Anker SD, Butler J, Filippatos G, et al. Empagliflozin in Heart Failure with a Preserved Ejection Fraction. *N Engl J Med*. 2021;385(16):1451-1461. doi:10.1056/NEJMoa2107038
- 12. McMurray JJV, Solomon SD, Inzucchi SE, et al. Dapagliflozin in Patients with Heart Failure and Reduced Ejection Fraction. N Engl J Med. 2019;381(21):1995-2008. doi:10.1056/NEJMoa1911303
- 13. Mohan V, Saboo B, Khader J, et al. Position of Sulfonylureas in the Current ERA: Review of National and International Guidelines. Clin Med Insights Endocrinol

- 14. Schneeweiss S. A basic study design for expedited safety signal evaluation based on electronic healthcare data. *Pharmacoepidemiol Drug Saf.* 2010;19(8):858-868. doi:10.1002/pds.1926
- 15. Ray WA. Evaluating medication effects outside of clinical trials: new-user designs. Am J Epidemiol. 2003;158(9):915-920. doi:10.1093/aje/kwg231
- 16. Kiyota Y, Schneeweiss S, Glynn RJ, Cannuscio CC, Avorn J, Solomon DH. Accuracy of medicare claims-based diagnosis of acute myocardial infarction: estimating positive predictive value on the basis of review of hospital records. *Am Heart J*. 2004;148(1):99-104. doi:10.1016/j.ahj.2004.02.013
- 17. Andrade SE, Harrold LR, Tjia J, et al. A systematic review of validated methods for identifying cerebrovascular accident or transient ischemic attack using administrative data. *Pharmacoepidemiol Drug Saf.* 2012;21 Suppl 1(Suppl 1):100-128. doi:10.1002/pds.2312
- 18. Roumie CL, Mitchel E, Gideon PS, Varas-Lorenzo C, Castellsague J, Griffin MR. Validation of ICD-9 codes with a high positive predictive value for incident strokes resulting in hospitalization using Medicaid health data. *Pharmacoepidemiol Drug Saf.* 2008;17(1):20-26. doi:10.1002/pds.1518
- 19. Wahl PM, Rodgers K, Schneeweiss S, et al. Validation of claims-based diagnostic and procedure codes for cardiovascular and gastrointestinal serious adverse events in a commercially-insured population. *Pharmacoepidemiol Drug Saf.* 2010;19(6):596-603. doi:10.1002/pds.1924
- 20. Gagne JJ, Glynn RJ, Avorn J, Levin R, Schneeweiss S. A combined comorbidity score predicted mortality in elderly patients better than existing scores. *J Clin Epidemiol*. 2011;64(7):749-759. doi:10.1016/j.jclinepi.2010.10.004
- 21. Sun JW, Rogers JR, Her Q, et al. Adaptation and Validation of the Combined Comorbidity Score for ICD-10-CM. *Med Care*. 2017;55(12):1046-1051. doi:10.1097/MLR.0000000000000824
- 22. Kim DH, Schneeweiss S, Glynn RJ, Lipsitz LA, Rockwood K, Avorn J. Measuring Frailty in Medicare Data: Development and Validation of a Claims-Based Frailty Index. *J Gerontol A Biol Sci Med Sci*. 2018;73(7):980-987. doi:10.1093/gerona/glx229
- 23. Olubowale OT, Safford MM, Brown TM, et al. Comparison of Expert Adjudicated Coronary Heart Disease and Cardiovascular Disease Mortality With the National Death Index: Results From the REasons for Geographic And Racial Differences in Stroke (REGARDS) Study. *J Am Heart Assoc.* 2017;6(5):e004966. doi:10.1161/JAHA.116.004966

## 10. Appendices

See accompanying excel files that specify the cohort study.

- 1 Target Trial Framework, Operational Definitions, and Data Fitness Assessment
- 2 Code algorithms
  - 2a Exposure
  - 2a Inclusion

- 2c Exclusion
- 2d Outcome
- **3 Flowchart for cohort assembly**
- 4 1st feasibility assessment
- 5 2nd feasibility assessment
- 6 Balance Assessment PS Distribution and C-Statistic
- 7 Balance Assessment Table 1
- **8 Covariate Algorithm Sources**

| | TIRZSITA-CVOT | OPTUM | MARKETSCAN | Notes/Questions | Color coding |
|---|---|---|---|---|---|
| | International, double-blind, randomized, active- | Non-randomized initiation of treatment Tirzepatide vs Sitagliptin | Non-randomized initiation of treatment Tirzepatide vs Sitagliptin | | |
| | Tirzepatide (subcutaneously | ordose Assessment window: N/A Source of algorithm: N/A | (first eligible entry to study population) Code type: RX Care settling: N/A Diagnosis position: N/A Washout window: [-183,-1] Incident with respect to: Tirzepatide and sitagliptininany formulation or dose Assessment window: N/A Source of algorithm: N/A | | |
| Exposure | | ordose Assessment window: N/A | Measurement characteristics: N/A Code type: RX Care setting: N/A Diagnosis position: N/A Washout window: [-183, -1] Incident with respect to: Tirzepatide and sitagliptininany formulation or dose Assessment window: N/A | | Good proxy definition |
| Comparator | | Source of algorithm: N/A Measurement characteristics: N/A Code type: DX, PX Care setting: Inpatient for MI, stroke, unstable angina. Any for coronary revascularization Diagnosis position: Primary Washout window: Source of algorithm: See below. Measurement characteristics: PPV for MI using ICD9 codes was 88.4% and 94%. | Source of algorithm: N/A Measurement characteristics: N/A Code type: DX, PX Care setting: Inpatient for MI, stroke, unstable angina. Any for coronary revascularization Diagnosis position: Primary Washout window: Source of algorithm: See below. Measurement characteristics: PPV for MI using ICD9 codes was 88.4% and 94%. | | Moderate proxy definition |
| Outcomes to be emulated<br>Follow up start | Atheroscelrotic cardiovascular events, i.e., myocardial infarction, stroke, coronary revasularization, unstable angina | PPV for ischemic stroke using ICD9 codes was 88% and 95% Both of the above ICD9 codes were mapped to ICD10, but no validation study was performed. One day after initiation of treatment with tirzepatide or sitagliptin | PPV for ischemic stroke using ICD9 codes was 88% and 95%. Both of the above ICD9 codes were mapped to ICD10, but no validation study was performed. One day after initiation of treatment with tirzepatide or sitagliptin | | Poorly measured in database |
| | Expected mean follow-up:1 year | Earliest of: Outcome, end of observation in data, end of study period (365 days), discontinuation of study drug (45 days grace window and risk-window), switch to other GLP-1-RA, nursing home admission | Earliest of: Outcome, end of observation in data, end of study period (365 days), discontinuation of study drug (45 days grace window and risk-window), switch to other GLP-1-RA, nursing home admission | Algorithm detail: Adherence in clinical practice databases is | |
| | Intention-to-treat effect Cox proportional hazards model | On-treatment effect Cox proportional hazards regression model | On-treatment effect Cox proportional hazards regression model | expected to be much worse than in the trial, therefore the on-<br>treatment analysis at 1 year follow-up will be the primary<br>analysis. | |
| | Men and women aged 40 years or older | Applied before/after selection of index date: Before Assessment window: [0,0] Code type: N/A Care setting: N/A Diagnosis position: N/A Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-365,0] Code type: DX Care setting: Any Diagnosis position: Any | Applied before/after selection of index date: Before Assessment window: [0, 0] Code type: N/A Care setting: N/A Diagnosis position: N/A Source of algorithm: N/A Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-365, 0] Code type: DX Care setting: Any Diagnosis position: Any Diagnosis position: Any | | |
| 2 | Type 2 diabetes mellitus | Source of algorithm: PROMISE team Measurement characteristics: N/A | Source of algorithm: PROMISE team<br>Measurement characteristics: N/A | | |
| 3 | HbA1c ≥7% and ≤ 10.5% | Applied before/after selection of index date: Before Assessment window: [-120, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-730, 0] Code type: DX, LOINC Care setting: Any Diagnosis position: Any Source of algorithm: Validation of obesity-related diagnosis codes in claims data: Validation of hot passing index (FMM): Prelated (ICD-9-CM) and ICD-10-CM and indistrate diagnosis codes recorded in IIS Calaims. | Applied before/after selection of index date: Before Assessment window: [-120,0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-730,0] Code type: DX, LOINC Care setting: Any Diagnosis position: Any Source of algorithm: Yallidation of obesity-related diagnosis codes in claims data: Yallidation of hody mass index (RMM)-related ICD-9-CM and ICD-10-CM administrative diagnosis codes recorded in US: Calaims. | Algorithm detail: Not considered in the main cohort due to high missingness of HbAIc measurements. A sensitivity analyses on a subset of the cohort with HbAIc measurements will be conducted in the cohort from the Optum database, including the last recorded value in the propensity score. | |
| | D | data | data | Algorithm detail: If BMI measurement via LOINC code is | |
| 5 | BMI ≥ 25kg/m2 Established atherosclerotic cardiovascular disease Coronary artery disease, either one of: | Applied before/after selection of index date: Before Assessment window: [all available data, 0] | Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] | below 10 or above 100 then measurent is set to missing. | |
| 51.1 | Documented history of myocardial infarction | Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A | Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A | | |

| 5.1.3 | ≥50% stenosis in ≥1 major coronary arteries determined by invasive angiography ≥50% stenosis in 2 or more major coronary arteries History of surgical or percutaneous coronary revascularization procedure | Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX, PX Care setting: Any Diagnosis position: N/A Source of algorithm: N/A Measurement characteristics: N/A | Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX, PX Care setting: Any Diagnosis position: N/A Source of algorithm: N/A Measurement characteristics: N/A Measurement characteristics: N/A | Algorithm detail: ≥50% stenosis was proxied by ICD-10 codes, based on the premise that most patients are coded only after surpassing the symptomatic threshold of 50-70%. |
|---|---|---|---|---|
| 5.2 | Cerebrovascular disease, either one of: Documented history of ischemic stroke | Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] | Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] | |
| 5.2.2 | Carotid arterial disease with ≥50% stenosis, documented by carotid ultrasound, MRI, or angiography | Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] | Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] | See 5.1.2 |
| 5.2.3 | History of carotid stenting or surgical revascularization Peripheral arterial disease, either one of: | Code type: DX, PX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before | Code type: DX, PX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before | |
| 5.3.1 | Intermittent claudication and ankle-brachial index < 0.9 | Applied before/after selection of index date: Before | Assessment window: [-all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before | Algorithm detail: Intermittent claudication was proxied by ICD-10-CM codes for peripheral vascular disease. |
| 5.3.2 | Prior nontraumatic amputation or peripheral vascular procedure (eg., stenting or surgical revascularization), due to peripheral arterial ischemia | Assessment window: [all available data, 0] Code tyne: DX, PX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A | Assessment window: [all available data, 0] Code type: DX, PX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A | |
| clusion criteria | | Applied before/after selection of index date: Before | Applied before/after selection of index date: Before | |
| | HbA1c>10.5% Planning treatment for diabetic retinopathy and/or | Assessment window: [-120, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-365, 0] Code type: PX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team | Assessment window: [-120,0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-365,0] Code type: PX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team | Algorithm detail: Not considered in the main cohort due to high missingness of HbALc measurements. A sensitivity analyses on a subset of the cohort with HbALc measurements will be conducted in the cohort from the Optum database, including the last recorded value in the propensity score. Algorithm detail: Planned treatment will be proxied by a history of treatment (e.g. codes for intravitreal injection of |
| | macular edema Hospitalized for chronic heart failure within 2 months prior to screening | Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-60, 0] for HF diagnosis or HHF Code type: DX, RX Care setting: Inpatient Diagnosis position: Primary Source of algorithm: DUPLICATE team, investigator reviewed codes Measurement characteristics: N/A | Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-60, 0] for HF diagnosis or HHF Code type: DX, RX Care setting: Inpatient Diagnosis position: Primary Source of algorithm: DUPLICATE team, investigator reviewed codes Measurement characteristics: N/A | anti-VEGFi OR photocoagulation.) |

| | Chronic New York Heart Association Functional | | | Algorithm detail: A proportion of patients with NYHA class |
|---|---|---|---|---|
| 9 | Classification IV heart failure | Can't be measured in claims. | Can't be measured in claims. | IV will be excluded from the cohort by exclusion criterion 8. |
| | Planned coronary, carotid, or peripheral artery | | | |
| 10 | revascularization | Can't be measured in claims. | Can't be measured in claims. | |
| | | Applied before/after selection of index date: Before | Applied before/after selection of index date: Before | |
| | | Assessment window: [-183,0] | Assessment window: [-183, 0] | |
| | | Code type: DX | Code type: DX | |
| | | Care setting: Any | Care setting: Any | |
| | | Diagnosis position: Any | Diagnosis position: Any | |
| | | Source of algorithm: PROMISE team | Source of algorithm: PROMISE team | |
| 11 | History of chronic or acute pancreatitis | Measurement characteristics: N/A | Measurement characteristics: N/A | |
| | | Applied before/after selection of index date: Before | Applied before/after selection of index date: Before | |
| | | Assessment window: [-365, 0] | Assessment window: [-365, 0] | |
| | | Code type: DX, | Code type: DX, | |
| | | Care setting: Inpatient | Care setting: Inpatient | |
| | | Diagnosis position: Any | Diagnosis position: Any | |
| | | Source of algorithm: PROMISE team, | Source of algorithm: PROMISE team, | |
| | | https://pubmed.ncbi.nlm.nih.gov/35857336/, Investigator reviewed | https://pubmed.nchi.nlm.nih.gov/35857336/. Investigator reviewed | |
| | Known clinically significant gastric emptying | codes | codes | |
| 12 | abnormality or bariatric surgery | Measurement characteristics: N/A | Measurement characteristics: N/A | See SUMMIT |
| | ability of bandare bangery | Applied before/after selection of index date: Before | Applied before/after selection of index date: Before | 000 00 1111111 |
| | | Assessment window: [-183,0] | Assessment window: [-183, 0] | |
| | | Code type: DX,PX | Code type: DX,PX | |
| | | Care setting: Any | Care setting: Any | |
| | | Diagnosis position: Any | Diagnosis position: Any | |
| | Liver disease (not including non-alcoholic fatty liver | Source of algorithm: Investigator reviewed codes | Source of algorithm: Investigator reviewed codes | Algorithm detail: Based on diagnostic codes rather than |
| 12 | disease [NAFLD]) or ALT level ≥3X the ULN | Measurement characteristics: N/A | Measurement characteristics: N/A | laboratory values. |
| 13 | disease [NATED]) of ALT level 23X the OLIV | Applied before/after selection of index date: Before | Applied before/after selection of index date: Before | laboratory values. |
| | | Assessment window: [-365,0] | Assessment window: [-365,0] | |
| | | Code type: DX, PX | Code type: DX, PX | |
| | | Care setting: Any | Care setting: Any | |
| | | Diagnosis position: Any | Diagnosis position: Any | Algorithm datail Proving by ICD 10 CM and an for abronia |
| | | Source of algorithm: PROMISE team | Source of algorithm: PROMISE team | Algorithm detail: Proxied by ICD-10-CM codes for chronic kidney disease stage 5 OR end-stage renal disease OR ICD- |
| | -OFR -15 I (Mi-/172 2 | Measurement characteristics: N/A | Measurement characteristics: N/A | |
| 14 | eGFR <15 mL/Min/1.73 m2 or on chronic dialysis | | | 10-CM procedure codes for dialysis. |
| | | Applied before/after selection of index date: Before Assessment window: [all available data, 0] | Applied before/after selection of index date: Before Assessment window: [all available data, 0] | |
| | | Code type: DX | Code type: DX | |
| | | Care setting: Any Diagnosis position: Any | Care setting: Any Diagnosis position: Any | |
| | Family or personal history of multiple endocrine | Source of algorithm: PROMISE team | Source of algorithm: PROMISE team | |
| 4.5 | | Measurement characteristics: N/A | Measurement characteristics: N/A | |
| | neoplasia or medullary thyroid carcinoma | | | |
| 16 | Elevated serum calcitonin level | Can't be measured in claims. | Can't be measured in claims. | |
| | | Applied before/after selection of index date: Before | Applied before/after selection of index date: Before | |
| | | Assessment window: [-60, 0] for all except unstable angina [-30, 0] | Assessment window: [-60, 0] for all except unstable angina [-30, 0] | |
| | | Code type: DX, PX Core cotting: Innation / ED for MI Strake TIA innation for proceedures | Code type: DX, PX Core actions Innation / ED for MI Strake TIA innation for proceedures | |
| | | Care setting: Inpatient/ED for MI, Stroke, TIA, inpatient for procedures<br>Diagnosis position: Any | Care setting: Inpatient/ED for MI, Stroke, TIA, inpatient for procedures<br>Diagnosis position: Any | |
| | 0 11 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 | | | |
| | | Source of algorithm: PROMISE team, Investigator reviewed codes | Source of algorithm: PROMISE team, Investigator reviewed codes | |
| 17 | screening | Measurement characteristics: N/A | Measurement characteristics: N/A | |
| | | Applied before/after selection of index date: Before | Applied before/after selection of index date: Before | |
| | | Assessment window: [-183, 0] | Assessment window: [-183, 0] | |
| | | Code type: RX | Code type: RX | |
| | | Care setting: N/A | Care setting: N/A | |
| | CLD 1 DAintid-tttuithi 2 | Diagnosis position: N/A | Diagnosis position: N/A | |
| | | Source of algorithm: N/A | Source of algorithm: N/A | |
| 18 | prior to Visit 1 | Measurement characteristics: n/a | Measurement characteristics: n/a | |
| | | Applied before/after selection of index date: Before | Applied before/after selection of index date: Before | |
| | | Assessment window: [-365, 0] | Assessment window: [-365, 0] | |
| | | Code type: DX | Code type: DX | |
| | | Code type: DX Care setting: Any | Care setting: Any | |
| | | Code type: DX<br>Care setting: Any<br>Diagnosis position: Any | Care setting: Any Diagnosis position: Any | Alassidas datail Davidado (OD 10 CM andre) |
| 10 | Women who are pregnant or breastfeeding | Code type: DX Care setting: Any | Care setting: Any | Algorithm detail: Proxied by ICD-10-CM codes indicative of pregnancy at baseline. |


| <b>5.1.4</b> History of surgical or percutaneous coronary revascularization procedure | 21009C PX | BYPASS CORONARY ARTERY, ONE ARTERY FROM THORACIC ARTERY WITH AUTOLOGOUS VENOUS TISSUE, OPEN APPROACH |
|---|---|---|
| <b>5.1.4</b> History of surgical or percutaneous coronary revascularization procedure | 21009F PX | BYPASS CORONARY ARTERY, ONE ARTERY FROM ABDOMINAL ARTERY WITH AUTOLOGOUS VENOUS TISSUE, OPEN APPROACH |
| <b>5.1.4</b> History of surgical or percutaneous coronary revascularization procedure | 21009W PX | BYPASS CORONARY ARTERY, ONE ARTERY FROM AORTA WITH AUTOLOGOUS VENOUS TISSUE, OPEN APPROACH |
| <b>5.1.4</b> History of surgical or percutaneous coronary revascularization procedure | 2100A3 PX | BYPASS CORONARY ARTERY, ONE ARTERY FROM CORONARY ARTERY WITH AUTOLOGOUS ARTERIAL TISSUE, OPEN APPROACH |
| <b>5.1.4</b> History of surgical or percutaneous coronary revascularization procedure | 2100A8 PX | BYPASS CORONARY ARTERY, ONE ARTERY FROM RIGHT INTERNAL MAMMARY WITH AUTOLOGOUS ARTERIAL TISSUE, OPEN APPROACH |
| <b>5.1.4</b> History of surgical or percutaneous coronary revascularization procedure | 2100A9 PX | BYPASS CORONARY ARTERY, ONE ARTERY FROM LEFT INTERNAL MAMMARY WITH AUTOLOGOUS ARTERIAL TISSUE, OPEN APPROACH |
| <b>5.1.4</b> History of surgical or percutaneous coronary revascularization procedure | 2100AC PX | BYPASS CORONARY ARTERY, ONE ARTERY FROM THORACIC ARTERY WITH AUTOLOGOUS ARTERIAL TISSUE, OPEN APPROACH |
| <b>5.1.4</b> History of surgical or percutaneous coronary revascularization procedure | 2100AF PX | BYPASS CORONARY ARTERY, ONE ARTERY FROM ABDOMINAL ARTERY WITH AUTOLOGOUS ARTERIAL TISSUE, OPEN APPROACH |
| <b>5.1.4</b> History of surgical or percutaneous coronary revascularization procedure | 2100AW PX | BYPASS CORONARY ARTERY, ONE ARTERY FROM AORTA WITH AUTOLOGOUS ARTERIAL TISSUE, OPEN APPROACH |
| <b>5.1.4</b> History of surgical or percutaneous coronary revascularization procedure | 2100J3 PX | BYPASS CORONARY ARTERY, ONE ARTERY FROM CORONARY ARTERY WITH SYNTHETIC SUBSTITUTE, OPEN APPROACH |
| <b>5.1.4</b> History of surgical or percutaneous coronary revascularization procedure | 2100J8 PX | BYPASS CORONARY ARTERY, ONE ARTERY FROM RIGHT INTERNAL MAMMARY WITH SYNTHETIC SUBSTITUTE, OPEN APPROACH |
| <b>5.1.4</b> History of surgical or percutaneous coronary revascularization procedure | 2100J9 PX | BYPASS CORONARY ARTERY, ONE ARTERY FROM LEFT INTERNAL MAMMARY WITH SYNTHETIC SUBSTITUTE, OPEN APPROACH |
| <b>5.1.4</b> History of surgical or percutaneous coronary revascularization procedure | 2100JC PX | BYPASS CORONARY ARTERY, ONE ARTERY FROM THORACIC ARTERY WITH SYNTHETIC SUBSTITUTE, OPEN APPROACH |
| <b>5.1.4</b> History of surgical or percutaneous coronary revascularization procedure | 2100JF PX | BYPASS CORONARY ARTERY, ONE ARTERY FROM ABDOMINAL ARTERY WITH SYNTHETIC SUBSTITUTE, OPEN APPROACH |
| <b>5.1.4</b> History of surgical or percutaneous coronary revascularization procedure | 2100JW PX | BYPASS CORONARY ARTERY, ONE ARTERY FROM AORTA WITH SYNTHETIC SUBSTITUTE, OPEN APPROACH |
| <b>5.1.4</b> History of surgical or percutaneous coronary revascularization procedure | 2100K3 PX | BYPASS CORONARY ARTERY, ONE ARTERY FROM CORONARY ARTERY WITH NONAUTOLOGOUS TISSUE SUBSTITUTE, OPEN APPROACH |
| <b>5.1.4</b> History of surgical or percutaneous coronary revascularization procedure | 2100K8 PX | $ \verb BYPASS CORONARY ARTERY, ONE ARTERY FROM RIGHT INTERNAL MAMMARY WITH NONAUTOLOGOUS TISSUE SUBSTITUTE, OPEN APPROACH \\$ |
| <b>5.1.4</b> History of surgical or percutaneous coronary revascularization procedure | 2100K9 PX | BYPASS CORONARY ARTERY, ONE ARTERY FROM LEFT INTERNAL MAMMARY WITH NONAUTOLOGOUS TISSUE SUBSTITUTE, OPEN APPROACH |
| <b>5.1.4</b> History of surgical or percutaneous coronary revascularization procedure | 2100KC PX | BYPASS CORONARY ARTERY, ONE ARTERY FROM THORACIC ARTERY WITH NONAUTOLOGOUS TISSUE SUBSTITUTE, OPEN APPROACH |
| <b>5.1.4</b> History of surgical or percutaneous coronary revascularization procedure | 2100KF PX | BYPASS CORONARY ARTERY, ONE ARTERY FROM ABDOMINAL ARTERY WITH NONAUTOLOGOUS TISSUE SUBSTITUTE, OPEN APPROACH |
| <b>5.1.4</b> History of surgical or percutaneous coronary revascularization procedure | 2100KW PX | BYPASS CORONARY ARTERY, ONE ARTERY FROM AORTA WITH NONAUTOLOGOUS TISSUE SUBSTITUTE, OPEN APPROACH |


| <b>5.1.4</b> History of surgical or percutaneous 0211 coronary revascularization procedure | .489 PX | BYPASS CORONARY ARTERY, TWO ARTERIES FROM LEFT INTERNAL MAMMARY WITH ZOOPLASTIC TISSUE, PERCUTANEOUS ENDOSCOPIC APPROACH |
|---|---|---|
| <b>5.1.4</b> History of surgical or percutaneous 0211 coronary revascularization procedure | .48C PX | BYPASS CORONARY ARTERY, TWO ARTERIES FROM THORACIC ARTERY WITH ZOOPLASTIC TISSUE, PERCUTANEOUS ENDOSCOPIC APPROACH |
| <b>5.1.4</b> History of surgical or percutaneous o211 coronary revascularization procedure | .48F PX | BYPASS CORONARY ARTERY, TWO ARTERIES FROM ABDOMINAL ARTERY WITH ZOOPLASTIC TISSUE, PERCUTANEOUS ENDOSCOPIC APPROACH |
| <b>5.1.4</b> History of surgical or percutaneous coronary revascularization procedure | 48W PX | BYPASS CORONARY ARTERY, TWO ARTERIES FROM AORTA WITH ZOOPLASTIC TISSUE, PERCUTANEOUS ENDOSCOPIC APPROACH |
| <b>5.1.4</b> History of surgical or percutaneous coronary revascularization procedure | 493 PX | BYPASS CORONARY ARTERY, TWO ARTERIES FROM CORONARY ARTERY WITH AUTOLOGOUS VENOUS TISSUE, PERCUTANEOUS ENDOSCOPIC APPROACH |
| <b>5.1.4</b> History of surgical or percutaneous coronary revascularization procedure | 498 PX | BYPASS CORONARY ARTERY, TWO ARTERIES FROM RIGHT INTERNAL MAMMARY WITH AUTOLOGOUS VENOUS TISSUE, PERCUTANEOUS ENDOSCOPIC APPROACH |
| <b>5.1.4</b> History of surgical or percutaneous coronary revascularization procedure | 499 PX | BYPASS CORONARY ARTERY, TWO ARTERIES FROM LEFT INTERNAL MAMMARY WITH AUTOLOGOUS VENOUS TISSUE, PERCUTANEOUS ENDOSCOPIC APPROACH |
| <b>5.1.4</b> History of surgical or percutaneous coronary revascularization procedure | 49C PX | BYPASS CORONARY ARTERY, TWO ARTERIES FROM THORACIC ARTERY WITH AUTOLOGOUS VENOUS TISSUE, PERCUTANEOUS ENDOSCOPIC APPROACH |
| <b>5.1.4</b> History of surgical or percutaneous coronary revascularization procedure | 49F PX | BYPASS CORONARY ARTERY, TWO ARTERIES FROM ABDOMINAL ARTERY WITH AUTOLOGOUS VENOUS TISSUE, PERCUTANEOUS ENDOSCOPIC APPROACH |
| <b>5.1.4</b> History of surgical or percutaneous coronary revascularization procedure | 49W PX | BYPASS CORONARY ARTERY, TWO ARTERIES FROM AORTA WITH AUTOLOGOUS VENOUS TISSUE, PERCUTANEOUS ENDOSCOPIC APPROACH |
| <b>5.1.4</b> History of surgical or percutaneous coronary revascularization procedure | 4A3 PX | BYPASS CORONARY ARTERY, TWO ARTERIES FROM CORONARY ARTERY WITH AUTOLOGOUS ARTERIAL TISSUE, PERCUTANEOUS ENDOSCOPIC APPROACH |
| <b>5.1.4</b> History of surgical or percutaneous coronary revascularization procedure | .4A8 PX | BYPASS CORONARY ARTERY, TWO ARTERIES FROM RIGHT INTERNAL MAMMARY WITH AUTOLOGOUS ARTERIAL TISSUE, PERCUTANEOUS ENDOSCOPIC APPROACH |
| <b>5.1.4</b> History of surgical or percutaneous coronary revascularization procedure | .4A9 PX | BYPASS CORONARY ARTERY, TWO ARTERIES FROM LEFT INTERNAL MAMMARY WITH AUTOLOGOUS ARTERIAL TISSUE, PERCUTANEOUS ENDOSCOPIC APPROACH |
| <b>5.1.4</b> History of surgical or percutaneous coronary revascularization procedure | .4AC PX | BYPASS CORONARY ARTERY, TWO ARTERIES FROM THORACIC ARTERY WITH AUTOLOGOUS ARTERIAL TISSUE, PERCUTANEOUS ENDOSCOPIC APPROACH |
| <b>5.1.4</b> History of surgical or percutaneous coronary revascularization procedure | .4AF PX | BYPASS CORONARY ARTERY, TWO ARTERIES FROM ABDOMINAL ARTERY WITH AUTOLOGOUS ARTERIAL TISSUE, PERCUTANEOUS ENDOSCOPIC APPROACH |
| <b>5.1.4</b> History of surgical or percutaneous coronary revascularization procedure | .4AW PX | BYPASS CORONARY ARTERY, TWO ARTERIES FROM AORTA WITH AUTOLOGOUS ARTERIAL TISSUE, PERCUTANEOUS ENDOSCOPIC APPROACH |
| <b>5.1.4</b> History of surgical or percutaneous 0211 coronary revascularization procedure | 4D4 PX | BYPASS CORONARY ARTERY, TWO ARTERIES FROM CORONARY VEIN WITH INTRALUMINAL DEVICE, PERCUTANEOUS ENDOSCOPIC APPROACH |
| <b>5.1.4</b> History of surgical or percutaneous 0211 coronary revascularization procedure | 4J3 PX | BYPASS CORONARY ARTERY, TWO ARTERIES FROM CORONARY ARTERY WITH SYNTHETIC SUBSTITUTE, PERCUTANEOUS ENDOSCOPIC APPROACH |
| <b>5.1.4</b> History of surgical or percutaneous coronary revascularization procedure | .4J8 PX | BYPASS CORONARY ARTERY, TWO ARTERIES FROM RIGHT INTERNAL MAMMARY WITH SYNTHETIC SUBSTITUTE, PERCUTANEOUS ENDOSCOPIC APPROACH |
| <b>5.1.4</b> History of surgical or percutaneous coronary revascularization procedure | 4J9 PX | BYPASS CORONARY ARTERY, TWO ARTERIES FROM LEFT INTERNAL MAMMARY WITH SYNTHETIC SUBSTITUTE, PERCUTANEOUS ENDOSCOPIC APPROACH |
| <b>5.1.4</b> History of surgical or percutaneous coronary revascularization procedure | 4JC PX | BYPASS CORONARY ARTERY, TWO ARTERIES FROM THORACIC ARTERY WITH SYNTHETIC SUBSTITUTE, PERCUTANEOUS ENDOSCOPIC APPROACH |

| <b>5.1.4</b> History of surgical or percutaneous 02114 coronary revascularization procedure | IJF PX | BYPASS CORONARY ARTERY, TWO ARTERIES FROM ABDOMINAL ARTERY WITH SYNTHETIC SUBSTITUTE, PERCUTANEOUS ENDOSCOPIC APPROACH |
|---|---|---|
| <b>5.1.4</b> History of surgical or percutaneous o2114 coronary revascularization procedure | IJW PX | BYPASS CORONARY ARTERY, TWO ARTERIES FROM AORTA WITH SYNTHETIC SUBSTITUTE, PERCUTANEOUS ENDOSCOPIC APPROACH |
| <b>5.1.4</b> History of surgical or percutaneous coronary revascularization procedure 02114 | IK3 PX | BYPASS CORONARY ARTERY, TWO ARTERIES FROM CORONARY ARTERY WITH NONAUTOLOGOUS TISSUE SUBSTITUTE, PERCUTANEOUS ENDOSCOPIC APPROACH |
| <b>5.1.4</b> History of surgical or percutaneous coronary revascularization procedure 02114 | IK8 PX | BYPASS CORONARY ARTERY, TWO ARTERIES FROM RIGHT INTERNAL MAMMARY WITH NONAUTOLOGOUS TISSUE SUBSTITUTE, PERCUTANEOUS ENDOSCOPIC APPROACH |
| <b>5.1.4</b> History of surgical or percutaneous coronary revascularization procedure | IK9 PX | BYPASS CORONARY ARTERY, TWO ARTERIES FROM LEFT INTERNAL MAMMARY WITH NONAUTOLOGOUS TISSUE SUBSTITUTE, PERCUTANEOUS ENDOSCOPIC APPROACH |
| <b>5.1.4</b> History of surgical or percutaneous coronary revascularization procedure | IKC PX | BYPASS CORONARY ARTERY, TWO ARTERIES FROM THORACIC ARTERY WITH NONAUTOLOGOUS TISSUE SUBSTITUTE, PERCUTANEOUS ENDOSCOPIC APPROACH |
| <b>5.1.4</b> History of surgical or percutaneous coronary revascularization procedure | IKF PX | BYPASS CORONARY ARTERY, TWO ARTERIES FROM ABDOMINAL ARTERY WITH NONAUTOLOGOUS TISSUE SUBSTITUTE, PERCUTANEOUS ENDOSCOPIC APPROACH |
| <b>5.1.4</b> History of surgical or percutaneous coronary revascularization procedure | IKW PX | BYPASS CORONARY ARTERY, TWO ARTERIES FROM AORTA WITH NONAUTOLOGOUS TISSUE SUBSTITUTE, PERCUTANEOUS ENDOSCOPIC APPROACH |
| <b>5.1.4</b> History of surgical or percutaneous coronary revascularization procedure | Z3 PX | BYPASS CORONARY ARTERY, TWO ARTERIES FROM CORONARY ARTERY, PERCUTANEOUS ENDOSCOPIC APPROACH |
| <b>5.1.4</b> History of surgical or percutaneous coronary revascularization procedure | 728 PX | BYPASS CORONARY ARTERY, TWO ARTERIES FROM RIGHT INTERNAL MAMMARY, PERCUTANEOUS ENDOSCOPIC APPROACH |
| <b>5.1.4</b> History of surgical or percutaneous coronary revascularization procedure 02114 | Z9 PX | BYPASS CORONARY ARTERY, TWO ARTERIES FROM LEFT INTERNAL MAMMARY, PERCUTANEOUS ENDOSCOPIC APPROACH |
| <b>5.1.4</b> History of surgical or percutaneous ocronary revascularization procedure | ZC PX | BYPASS CORONARY ARTERY, TWO ARTERIES FROM THORACIC ARTERY, PERCUTANEOUS ENDOSCOPIC APPROACH |
| <b>5.1.4</b> History of surgical or percutaneous coronary revascularization procedure | ZF PX | BYPASS CORONARY ARTERY, TWO ARTERIES FROM ABDOMINAL ARTERY, PERCUTANEOUS ENDOSCOPIC APPROACH |
| <b>5.1.4</b> History of surgical or percutaneous coronary revascularization procedure | 33 PX | BYPASS CORONARY ARTERY, THREE ARTERIES FROM CORONARY ARTERY WITH ZOOPLASTIC TISSUE, OPEN APPROACH |
| <b>5.1.4</b> History of surgical or percutaneous coronary revascularization procedure | 38 PX | BYPASS CORONARY ARTERY, THREE ARTERIES FROM RIGHT INTERNAL MAMMARY WITH ZOOPLASTIC TISSUE, OPEN APPROACH |
| <b>5.1.4</b> History of surgical or percutaneous coronary revascularization procedure | 39 PX | BYPASS CORONARY ARTERY, THREE ARTERIES FROM LEFT INTERNAL MAMMARY WITH ZOOPLASTIC TISSUE, OPEN APPROACH |
| <b>5.1.4</b> History of surgical or percutaneous o2120 coronary revascularization procedure | D8C PX | BYPASS CORONARY ARTERY, THREE ARTERIES FROM THORACIC ARTERY WITH ZOOPLASTIC TISSUE, OPEN APPROACH |
| <b>5.1.4</b> History of surgical or percutaneous 02120 coronary revascularization procedure | D8F PX | BYPASS CORONARY ARTERY, THREE ARTERIES FROM ABDOMINAL ARTERY WITH ZOOPLASTIC TISSUE, OPEN APPROACH |
| <b>5.1.4</b> History of surgical or percutaneous 02120 coronary revascularization procedure | D8W PX | BYPASS CORONARY ARTERY, THREE ARTERIES FROM AORTA WITH ZOOPLASTIC TISSUE, OPEN APPROACH |
| <b>5.1.4</b> History of surgical or percutaneous 21209 coronary revascularization procedure | 93 PX | BYPASS CORONARY ARTERY, THREE ARTERIES FROM CORONARY ARTERY WITH AUTOLOGOUS VENOUS TISSUE, OPEN APPROACH |
| <b>5.1.4</b> History of surgical or percutaneous 21209 coronary revascularization procedure | 98 PX | BYPASS CORONARY ARTERY, THREE ARTERIES FROM RIGHT INTERNAL MAMMARY WITH AUTOLOGOUS VENOUS TISSUE, OPEN APPROACH |


| <b>5.1.4</b> History of surgical or percutaneous 0271 coronary revascularization procedure | 1076 PX | DILATION OF CORONARY ARTERY, TWO ARTERIES, BIFURCATION, WITH FOUR OR MORE DRUG-ELUTING INTRALUMINAL DEVICES, OPEN APPROACH |
|---|---|---|
| <b>5.1.4</b> History of surgical or percutaneous 0271 coronary revascularization procedure | 107Z PX | DILATION OF CORONARY ARTERY, TWO ARTERIES WITH FOUR OR MORE DRUG-ELUTING INTRALUMINAL DEVICES, OPEN APPROACH |
| <b>5.1.4</b> History of surgical or percutaneous 0271 coronary revascularization procedure | LOD6 PX | DILATION OF CORONARY ARTERY, TWO ARTERIES, BIFURCATION, WITH INTRALUMINAL DEVICE, OPEN APPROACH |
| <b>5.1.4</b> History of surgical or percutaneous 0271 coronary revascularization procedure | LODZ PX | DILATION OF CORONARY ARTERY, TWO ARTERIES WITH INTRALUMINAL DEVICE, OPEN APPROACH |
| <b>5.1.4</b> History of surgical or percutaneous coronary revascularization procedure | 10E6 PX | DILATION OF CORONARY ARTERY, TWO ARTERIES, BIFURCATION, WITH TWO INTRALUMINAL DEVICES, OPEN APPROACH |
| <b>5.1.4</b> History of surgical or percutaneous coronary revascularization procedure | LOEZ PX | DILATION OF CORONARY ARTERY, TWO ARTERIES WITH TWO INTRALUMINAL DEVICES, OPEN APPROACH |
| <b>5.1.4</b> History of surgical or percutaneous 0271 coronary revascularization procedure | LOF6 PX | DILATION OF CORONARY ARTERY, TWO ARTERIES, BIFURCATION, WITH THREE INTRALUMINAL DEVICES, OPEN APPROACH |
| <b>5.1.4</b> History of surgical or percutaneous 0271 coronary revascularization procedure | LOFZ PX | DILATION OF CORONARY ARTERY, TWO ARTERIES WITH THREE INTRALUMINAL DEVICES, OPEN APPROACH |
| <b>5.1.4</b> History of surgical or percutaneous 0271 coronary revascularization procedure | LOG6 PX | DILATION OF CORONARY ARTERY, TWO ARTERIES, BIFURCATION, WITH FOUR OR MORE INTRALUMINAL DEVICES, OPEN APPROACH |
| <b>5.1.4</b> History of surgical or percutaneous coronary revascularization procedure | LOGZ PX | DILATION OF CORONARY ARTERY, TWO ARTERIES WITH FOUR OR MORE INTRALUMINAL DEVICES, OPEN APPROACH |
| <b>5.1.4</b> History of surgical or percutaneous 0271 coronary revascularization procedure | L0T6 PX | DILATION OF CORONARY ARTERY, TWO ARTERIES, BIFURCATION, WITH RADIOACTIVE INTRALUMINAL DEVICE, OPEN APPROACH |
| <b>5.1.4</b> History of surgical or percutaneous coronary revascularization procedure | LOTZ PX | DILATION OF CORONARY ARTERY, TWO ARTERIES WITH RADIOACTIVE INTRALUMINAL DEVICE, OPEN APPROACH |
| <b>5.1.4</b> History of surgical or percutaneous 0271 coronary revascularization procedure | 10Z6 PX | DILATION OF CORONARY ARTERY, TWO ARTERIES, BIFURCATION, OPEN APPROACH |
| <b>5.1.4</b> History of surgical or percutaneous coronary revascularization procedure | LOZZ PX | DILATION OF CORONARY ARTERY, TWO ARTERIES, OPEN APPROACH |
| <b>5.1.4</b> History of surgical or percutaneous coronary revascularization procedure | 1346 PX | DILATION OF CORONARY ARTERY, TWO ARTERIES, BIFURCATION, WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTANEOUS APPROACH |
| <b>5.1.4</b> History of surgical or percutaneous coronary revascularization procedure | 134Z PX | DILATION OF CORONARY ARTERY, TWO ARTERIES WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTANEOUS APPROACH |
| <b>5.1.4</b> History of surgical or percutaneous coronary revascularization procedure | 1356 PX | DILATION OF CORONARY ARTERY, TWO ARTERIES, BIFURCATION, WITH TWO DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH |
| <b>5.1.4</b> History of surgical or percutaneous 0271 coronary revascularization procedure | 135Z PX | DILATION OF CORONARY ARTERY, TWO ARTERIES WITH TWO DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH |
| <b>5.1.4</b> History of surgical or percutaneous coronary revascularization procedure | 1366 PX | DILATION OF CORONARY ARTERY, TWO ARTERIES, BIFURCATION, WITH THREE DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH |
| <b>5.1.4</b> History of surgical or percutaneous coronary revascularization procedure | 136Z PX | DILATION OF CORONARY ARTERY, TWO ARTERIES WITH THREE DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH |
| <b>5.1.4</b> History of surgical or percutaneous coronary revascularization procedure | 1376 PX | DILATION OF CORONARY ARTERY, TWO ARTERIES, BIFURCATION, WITH FOUR OR MORE DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH |

| <b>5.1.4</b> History of surgical or percutaneous coronary revascularization procedure | 137Z PX | DILATION OF CORONARY ARTERY, TWO ARTERIES WITH FOUR OR MORE DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH |
|---|---|---|
| <b>5.1.4</b> History of surgical or percutaneous coronary revascularization procedure | 13D6 PX | DILATION OF CORONARY ARTERY, TWO ARTERIES, BIFURCATION, WITH INTRALUMINAL DEVICE, PERCUTANEOUS APPROACH |
| <b>5.1.4</b> History of surgical or percutaneous 027 coronary revascularization procedure | 13DZ PX | DILATION OF CORONARY ARTERY, TWO ARTERIES WITH INTRALUMINAL DEVICE, PERCUTANEOUS APPROACH |
| <b>5.1.4</b> History of surgical or percutaneous 027 coronary revascularization procedure | 13E6 PX | DILATION OF CORONARY ARTERY, TWO ARTERIES, BIFURCATION, WITH TWO INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH |
| <b>5.1.4</b> History of surgical or percutaneous 027 coronary revascularization procedure | 13EZ PX | DILATION OF CORONARY ARTERY, TWO ARTERIES WITH TWO INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH |
| <b>5.1.4</b> History of surgical or percutaneous 027 coronary revascularization procedure | 13F6 PX | DILATION OF CORONARY ARTERY, TWO ARTERIES, BIFURCATION, WITH THREE INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH |
| <b>5.1.4</b> History of surgical or percutaneous 027 coronary revascularization procedure | 13FZ PX | DILATION OF CORONARY ARTERY, TWO ARTERIES WITH THREE INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH |
| <b>5.1.4</b> History of surgical or percutaneous 027 coronary revascularization procedure | 13G6 PX | DILATION OF CORONARY ARTERY, TWO ARTERIES, BIFURCATION, WITH FOUR OR MORE INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH |
| <b>5.1.4</b> History of surgical or percutaneous 027 coronary revascularization procedure | 13GZ PX | DILATION OF CORONARY ARTERY, TWO ARTERIES WITH FOUR OR MORE INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH |
| <b>5.1.4</b> History of surgical or percutaneous 027 coronary revascularization procedure | 13T6 PX | DILATION OF CORONARY ARTERY, TWO ARTERIES, BIFURCATION, WITH RADIOACTIVE INTRALUMINAL DEVICE, PERCUTANEOUS APPROACH |
| <b>5.1.4</b> History of surgical or percutaneous 027 coronary revascularization procedure | 13TZ PX | DILATION OF CORONARY ARTERY, TWO ARTERIES WITH RADIOACTIVE INTRALUMINAL DEVICE, PERCUTANEOUS APPROACH |
| <b>5.1.4</b> History of surgical or percutaneous 027 coronary revascularization procedure | 13Z6 PX | DILATION OF CORONARY ARTERY, TWO ARTERIES, BIFURCATION, PERCUTANEOUS APPROACH |
| <b>5.1.4</b> History of surgical or percutaneous 027 coronary revascularization procedure | 13ZZ PX | DILATION OF CORONARY ARTERY, TWO ARTERIES, PERCUTANEOUS APPROACH |
| <b>5.1.4</b> History of surgical or percutaneous 027 coronary revascularization procedure | 1446 PX | DILATION OF CORONARY ARTERY, TWO ARTERIES, BIFURCATION, WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTANEOUS ENDOSCOPIC APPROACH |
| <b>5.1.4</b> History of surgical or percutaneous 027 coronary revascularization procedure | 144Z PX | DILATION OF CORONARY ARTERY, TWO ARTERIES WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTANEOUS ENDOSCOPIC APPROACH |
| <b>5.1.4</b> History of surgical or percutaneous 027 coronary revascularization procedure | 1456 PX | DILATION OF CORONARY ARTERY, TWO ARTERIES, BIFURCATION, WITH TWO DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS ENDOSCOPIC APPROACH |
| <b>5.1.4</b> History of surgical or percutaneous 027 coronary revascularization procedure | 145Z PX | DILATION OF CORONARY ARTERY, TWO ARTERIES WITH TWO DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS ENDOSCOPIC APPROACH |
| <b>5.1.4</b> History of surgical or percutaneous 027 coronary revascularization procedure | 1466 PX | DILATION OF CORONARY ARTERY, TWO ARTERIES, BIFURCATION, WITH THREE DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS ENDOSCOPIC APPROACH |
| <b>5.1.4</b> History of surgical or percutaneous 027 coronary revascularization procedure | 146Z PX | DILATION OF CORONARY ARTERY, TWO ARTERIES WITH THREE DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS ENDOSCOPIC APPROACH |
| <b>5.1.4</b> History of surgical or percutaneous 027 coronary revascularization procedure | 1476 PX | DILATION OF CORONARY ARTERY, TWO ARTERIES, BIFURCATION, WITH FOUR OR MORE DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS ENDOSCOPIC APPROACH |
| <b>5.1.4</b> History of surgical or percutaneous coronary revascularization procedure | 147Z PX | DILATION OF CORONARY ARTERY, TWO ARTERIES WITH FOUR OR MORE DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS ENDOSCOPIC APPROACH |


| <b>5.1.4</b> History of surgical or percutaneous coronary revascularization procedure | 23ZZ PX | EXTIRPATION OF MATTER FROM CORONARY ARTERY, THREE ARTERIES, PERCUTANEOUS APPROACH |
|---|---|---|
| <b>5.1.4</b> History of surgical or percutaneous coronary revascularization procedure | 24Z6 PX | EXTIRPATION OF MATTER FROM CORONARY ARTERY, THREE ARTERIES, BIFURCATION, PERCUTANEOUS ENDOSCOPIC APPROACH |
| <b>5.1.4</b> History of surgical or percutaneous coronary revascularization procedure | 24ZZ PX | EXTIRPATION OF MATTER FROM CORONARY ARTERY, THREE ARTERIES, PERCUTANEOUS ENDOSCOPIC APPROACH |
| <b>5.1.4</b> History of surgical or percutaneous coronary revascularization procedure | 30Z6 PX | EXTIRPATION OF MATTER FROM CORONARY ARTERY, FOUR OR MORE ARTERIES, BIFURCATION, OPEN APPROACH |
| <b>5.1.4</b> History of surgical or percutaneous coronary revascularization procedure | 30ZZ PX | EXTIRPATION OF MATTER FROM CORONARY ARTERY, FOUR OR MORE ARTERIES, OPEN APPROACH |
| <b>5.1.4</b> History of surgical or percutaneous coronary revascularization procedure | 33Z6 PX | EXTIRPATION OF MATTER FROM CORONARY ARTERY, FOUR OR MORE ARTERIES, BIFURCATION, PERCUTANEOUS APPROACH |
| <b>5.1.4</b> History of surgical or percutaneous coronary revascularization procedure | 33ZZ PX | EXTIRPATION OF MATTER FROM CORONARY ARTERY, FOUR OR MORE ARTERIES, PERCUTANEOUS APPROACH |
| <b>5.1.4</b> History of surgical or percutaneous coronary revascularization procedure | 34Z6 PX | EXTIRPATION OF MATTER FROM CORONARY ARTERY, FOUR OR MORE ARTERIES, BIFURCATION, PERCUTANEOUS ENDOSCOPIC APPROACH |
| <b>5.1.4</b> History of surgical or percutaneous o2C3 coronary revascularization procedure | 34ZZ PX | EXTIRPATION OF MATTER FROM CORONARY ARTERY, FOUR OR MORE ARTERIES, PERCUTANEOUS ENDOSCOPIC APPROACH |
| <b>5.1.4</b> History of surgical or percutaneous 02Q/coronary revascularization procedure | AOZZ PX | REPAIR HEART, OPEN APPROACH |
| <b>5.1.4</b> History of surgical or percutaneous 02Q/coronary revascularization procedure | A3ZZ PX | REPAIR HEART, PERCUTANEOUS APPROACH |
| <b>5.1.4</b> History of surgical or percutaneous 02Q/coronary revascularization procedure | A4ZZ PX | REPAIR HEART, PERCUTANEOUS ENDOSCOPIC APPROACH |
| <b>5.1.4</b> History of surgical or percutaneous coronary revascularization procedure | BOZZ PX | REPAIR RIGHT HEART, OPEN APPROACH |
| <b>5.1.4</b> History of surgical or percutaneous 02QE coronary revascularization procedure | B3ZZ PX | REPAIR RIGHT HEART, PERCUTANEOUS APPROACH |
| <b>5.1.4</b> History of surgical or percutaneous 02QE coronary revascularization procedure | B4ZZ PX | REPAIR RIGHT HEART, PERCUTANEOUS ENDOSCOPIC APPROACH |
| <b>5.1.4</b> History of surgical or percutaneous 02QG coronary revascularization procedure | COZZ PX | REPAIR LEFT HEART, OPEN APPROACH |
| <b>5.1.4</b> History of surgical or percutaneous 02QG coronary revascularization procedure | C3ZZ PX | REPAIR LEFT HEART, PERCUTANEOUS APPROACH |
| <b>5.1.4</b> History of surgical or percutaneous 02QG coronary revascularization procedure | C4ZZ PX | REPAIR LEFT HEART, PERCUTANEOUS ENDOSCOPIC APPROACH |
| <b>5.1.4</b> History of surgical or percutaneous coronary revascularization procedure | 10 PX | TRANSMYOCARDIAL LASER REVASCULARIZATION, BY THORACOTOMY; (SEPARATE PROCEDURE) |
| <b>5.1.4</b> History of surgical or percutaneous coronary revascularization procedure | PX | TRANSMYOCARDIAL LASER REVASCULARIZATION, BY THORACOTOMY; PERFORMED AT THE TIME OF OTHER OPEN CARDIAC PROCEDURE(S) (LIST SEPARATELY IN ADDITION TO CODE FOR PRIMARY PROCEDURE) |
| <b>5.1.4</b> History of surgical or percutaneous coronary revascularization procedure | 10 PX | CORONARY ARTERY BYPASS, VEIN ONLY; SINGLE CORONARY VENOUS GRAFT |


| <b>5.1.4</b> History of surgical or percutaneous coronary revascularization procedure | | PERCUTANEOUS TRANSLUMINAL CORONARY ATHERECTOMY, WITH CORONARY ANGIOPLASTY WHEN PERFORMED; EACH ADDITIONAL BRANCH OF A MAJOR CORONARY ARTERY (LIST SEPARATELY IN ADDITION TO CODE FOR PRIMARY PROCEDURE) |
|---|---|---|
| <b>5.1.4</b> History of surgical or percutaneous coronary revascularization procedure | | PERCUTANEOUS TRANSCATHETER PLACEMENT OF INTRACORONARY STENT(S), WITH CORONARY ANGIOPLASTY WHEN PERFORMED; SINGLE MAJOR CORONARY ARTERY OR BRANCH |
| <b>5.1.4</b> History of surgical or percutaneous coronary revascularization procedure | | PERCUTANEOUS TRANSCATHETER PLACEMENT OF INTRACORONARY STENT(S), WITH CORONARY ANGIOPLASTY WHEN PERFORMED; EACH ADDITIONAL BRANCH OF A MAJOR CORONARY ARTERY (LIST SEPARATELY IN ADDITION TO CODE FOR PRIMARY PROCEDURE) |
| <b>5.1.4</b> History of surgical or percutaneous coronary revascularization procedure | 33 PX | PERCUTANEOUS TRANSLUMINAL CORONARY ATHERECTOMY, WITH INTRACORONARY STENT, WITH CORONARY ANGIOPLASTY WHEN PERFORMED; SINGLE MAJOR CORONARY ARTERY OR BRANCH |
| <b>5.1.4</b> History of surgical or percutaneous coronary revascularization procedure | | PERCUTANEOUS TRANSLUMINAL CORONARY ATHERECTOMY, WITH INTRACORONARY STENT, WITH CORONARY ANGIOPLASTY WHEN PERFORMED; EACH ADDITIONAL BRANCH OF A MAJOR CORONARY ARTERY (LIST SEPARATELY IN ADDITION TO CODE FOR PRIMARY PROCEDURE) |
| <b>5.1.4</b> History of surgical or percutaneous coronary revascularization procedure | 37 PX | PERCUTANEOUS TRANSLUMINAL REVASCULARIZATION OF OR THROUGH CORONARY ARTERY BYPASS GRAFT (INTERNAL MAMMARY, FREE ARTERIAL, VENOUS), ANY COMBINATION OF INTRACORONARY STENT, ATHERECTOMY AND ANGIOPLASTY, INCLUDING DISTAL PROTECTION WHEN PERFORMED; SINGLE VESSEL |
| <b>5.1.4</b> History of surgical or percutaneous coronary revascularization procedure | 38 PX | PERCUTANEOUS TRANSLUMINAL REVASCULARIZATION OF OR THROUGH CORONARY ARTERY BYPASS GRAFT (INTERNAL MAMMARY, FREE ARTERIAL, VENOUS), ANY COMBINATION OF INTRACORONARY STENT, ATHERECTOMY AND ANGIOPLASTY, INCLUDING DISTAL PROTECTION WHEN PERFORMED; EACH ADDITIONAL BRANCH SUBTENDED BY THE BYPASS GRAFT (LIST SEPARATELY IN ADDITION TO CODE FOR PRIMARY PROCEDURE) |
| <b>5.1.4</b> History of surgical or percutaneous 9294 coronary revascularization procedure | 41 PX | PERCUTANEOUS TRANSLUMINAL REVASCULARIZATION OF ACUTE TOTAL/SUBTOTAL OCCLUSION DURING ACUTE MYOCARDIAL INFARCTION, CORONARY ARTERY OR CORONARY ARTERY BYPASS GRAFT, ANY COMBINATION OF INTRACORONARY STENT, ATHERECTOMY AND ANGIOPLASTY, INCLUDING ASPIRATION THROMBECTOMY WHEN PERFORMED, SINGLE VESSEL |
| <b>5.1.4</b> History of surgical or percutaneous coronary revascularization procedure | | PERCUTANEOUS TRANSLUMINAL REVASCULARIZATION OF CHRONIC TOTAL OCCLUSION, CORONARY ARTERY, CORONARY ARTERY BRANCH, OR CORONARY ARTERY BYPASS GRAFT, ANY COMBINATION OF INTRACORONARY STENT, ATHERECTOMY AND ANGIOPLASTY: SINGLE VESSEL |
| <b>5.1.4</b> History of surgical or percutaneous 9294 coronary revascularization procedure | 44 PX | PERCUTANEOUS TRANSLUMINAL REVASCULARIZATION OF CHRONIC TOTAL OCCLUSION, CORONARY ARTERY, CORONARY ARTERY BRANCH, OR CORONARY ARTERY BYPASS GRAFT, ANY COMBINATION OF INTRACORONARY STENT, ATHERECTOMY AND ANGIOPLASTY; EACH ADDITIONAL CORONARY ARTERY, CORONARY ARTERY BRANCH, OR BYPASS GRAFT (LIST SEPARATELY IN ADDITION TO CODE FOR PRIMARY PROCEDURE) |
| <b>5.1.4</b> History of surgical or percutaneous coronary revascularization procedure | 73 PX | PERCUTANEOUS TRANSLUMINAL CORONARY THROMBECTOMY MECHANICAL (LIST SEPARATELY IN ADDITION TO CODE FOR PRIMARY PROCEDURE) |
| <b>5.1.4</b> History of surgical or percutaneous coronary revascularization procedure | | TRANSCATHETER PLACEMENT OF AN INTRACORONARY STENT(S), PERCUTANEOUS, WITH OR WITHOUT OTHER THERAPEUTIC INTERVENTION, ANY METHOD; SINGLE VESSEL |
| <b>5.1.4</b> History of surgical or percutaneous coronary revascularization procedure | | TRANSCATHETER PLACEMENT OF AN INTRACORONARY STENT(S), PERCUTANEOUS, WITH OR WITHOUT OTHER THERAPEUTIC INTERVENTION, ANY METHOD; EACH ADDITIONAL VESSEL (LIST SEPARATELY IN ADDITION TO CODE FOR PRIMARY PROCEDURE) |
| <b>5.1.4</b> History of surgical or percutaneous coronary revascularization procedure | 82 PX | PERCUTANEOUS TRANSLUMINAL CORONARY BALLOON ANGIOPLASTY; SINGLE VESSEL |
| <b>5.1.4</b> History of surgical or percutaneous coronary revascularization procedure | | PERCUTANEOUS TRANSLUMINAL CORONARY BALLOON ANGIOPLASTY; EACH ADDITIONAL VESSEL (LIST SEPARATELY IN ADDITION TO CODE FOR PRIMARY PROCEDURE) |
| <b>5.1.4</b> History of surgical or percutaneous coronary revascularization procedure | | PERCUTANEOUS TRANSLUMINAL CORONARY ATHERECTOMY, BY MECHANICAL OR OTHER METHOD, WITH OR WITHOUT BALLOON ANGIOPLASTY; SINGLE VESSEL |
| <b>5.1.4</b> History of surgical or percutaneous coronary revascularization procedure | | PERCUTANEOUS TRANSLUMINAL CORONARY ATHERECTOMY, BY MECHANICAL OR OTHER METHOD, WITH OR WITHOUT BALLOON ANGIOPLASTY; EACH ADDITIONAL VESSEL (LIST SEPARATELY IN ADDITION TO CODE FOR PRIMARY PROCEDURE) |
| <b>5.1.4</b> History of surgical or percutaneous coronary revascularization procedure | 1 DX | PRESENCE OF AORTOCORONARY BYPASS GRAFT |
| <b>5.1.4</b> History of surgical or percutaneous coronary revascularization procedure | 5 DX | PRESENCE OF CORONARY ANGIOPLASTY IMPLANT AND GRAFT |
| <b>5.1.4</b> History of surgical or percutaneous coronary revascularization procedure | 61 DX | CORONARY ANGIOPLASTY STATUS |


| brachial index < 0.9 5.31 Intermittent claudication and anklebrachial index < 0.9 5.32 Intermittent claudication and anklebrachial index < 0.9 5.33 Intermittent claudication and anklebrachial index < 0.9 5.34 Intermittent claudication and anklebrachial index < 0.9 5.35 Intermittent claudication and ankle | ERAL LEGS R EXTREMITY ECIFIED EXTREMITY CLAUDICATION, RIGHT LEG CLAUDICATION, LEFT LEG CLAUDICATION, CLAUDICATION, OTHER CLAUDICATION, HT LEG |
|---|---|
| 5.3.1 Intermittent claudication and anklebrachial index <0.9 5.3.2 Intermittent claudication and anklebrachial index <0.9 5.3.3 Intermittent claudication and anklebrachial index <0.9 5.3.4 Intermittent claudication and anklebrachial index <0.9 5.3.5 Intermittent claudication and anklebrachial index <0.9 5.3.1 Intermittent claudication and anklebrachial index <0.9 5.3.2 Intermittent claudication and anklebrachial index <0.9 | R EXTREMITY CLAUDICATION, RIGHT LEG CLAUDICATION, LEFT LEG CLAUDICATION, CLAUDICATION, OTHER CLAUDICATION, HT LEG |
| 5.3.1 Intermittent claudication and anklebrachial index < 0.9 5.3.2 Intermittent claudication and anklebrachial index < 0.9 5.3.3 Intermittent claudication and anklebrachial index < 0.9 5.3.4 Intermittent claudication and anklebrachial index < 0.9 5.3.5 Intermittent claudication and anklebrachial index < 0.9 5.3.6 Intermittent claudication and anklebrachial index < 0.9 5.3.7 Intermittent claudication and anklebrachial index < 0.9 5.3.8 Intermittent claudication and anklebrachial index < 0.9 5.3.9 Intermittent claudication and anklebrachial index < 0.9 5.3.1 Intermittent claudication and anklebrachial index < 0.9 5.3.2 Intermittent claudication and anklebrachial index < 0.9 5.3.3 Intermittent claudication and anklebrachial index < 0.9 5.3.4 Intermittent claudicatio | CLAUDICATION, RIGHT LEG CLAUDICATION, LEFT LEG CLAUDICATION, CLAUDICATION, OTHER CLAUDICATION, HT LEG |
| 5.3.1 Intermittent claudication and anklebrachial index < 0.9 5.3.2 Intermittent claudication and anklebrachial index < 0.9 5.3.3 Intermittent claudication and anklebrachial index < 0.9 5.3.4 Intermittent claudication and anklebrachial index < 0.9 5.3.2 Intermittent claudicatio | CLAUDICATION, RIGHT LEG CLAUDICATION, LEFT LEG CLAUDICATION, CLAUDICATION, OTHER CLAUDICATION, HT LEG |
| brachial index <0.9 5.31 Intermittent claudication and ankle-brachial index <0.9 | CLAUDICATION, LEFT LEG CLAUDICATION, CLAUDICATION, OTHER CLAUDICATION, HT LEG |
| 5.3.1 Intermittent claudication and anklebrachial index <0.9 DX ATHEROSCLEROSIS OF AUTOLOGOUS VEIN BYPASS GRAFT(S) OF THE EXTREMITIES WITH INTERMITTENT OF ATHEROSCLEROSIS OF AUTOLOGOUS VEIN BYPASS GRAFT(S) OF THE EXTREMITIES WITH INTERMITTENT OF UNSPECIFIED EXTREMITY | CLAUDICATION, CLAUDICATION, OTHER CLAUDICATION, HT LEG |
| 5.3.1 Intermittent claudication and anklebrachial index < 0.9 5.3.1 Intermittent claudicatio | CLAUDICATION, OTHER CLAUDICATION, HT LEG |
| brachial index < 0.9 EXTREMITY 5.3.1 Intermittent claudication and ankle- 170.419 DX ATHEROSCLEROSIS OF AUTOLOGOUS VEIN BYPASS GRAFT(S) OF THE EXTREMITIES WITH INTERMITTENT OF UNSPECIFIED EXTREMITY | CLAUDICATION,<br>HT LEG |
| brachial index < 0.9 UNSPECIFIED EXTREMITY | HTLEG<br>TLEG |
| | TLEG |
| 5.3.1 Intermittent claudication and ankle- I70.421 DX ATHEROSCLEROSIS OF AUTOLOGOUS VEIN BYPASS GRAFT(S) OF THE EXTREMITIES WITH REST PAIN, RIGH brachial index < 0.9 | |
| 5.3.1 Intermittent claudication and ankle- I70.422 DX ATHEROSCLEROSIS OF AUTOLOGOUS VEIN BYPASS GRAFT(S) OF THE EXTREMITIES WITH REST PAIN, LEFT brachial index < 0.9 | ATERAL LEGS |
| 5.3.1 Intermittent claudication and ankle- I70.423 DX ATHEROSCLEROSIS OF AUTOLOGOUS VEIN BYPASS GRAFT(S) OF THE EXTREMITIES WITH REST PAIN, BILA brachial index < 0.9 | |
| 5.3.1 Intermittent claudication and ankle- I70.428 DX ATHEROSCLEROSIS OF AUTOLOGOUS VEIN BYPASS GRAFT(S) OF THE EXTREMITIES WITH REST PAIN, OTHE brachial index < 0.9 | IER EXTREMITY |
| 5.3.1 Intermittent claudication and ankle- I70.429 DX ATHEROSCLEROSIS OF AUTOLOGOUS VEIN BYPASS GRAFT(S) OF THE EXTREMITIES WITH REST PAIN, UNSI brachial index < 0.9 | SPECIFIED EXTREMITY |
| 5.3.1 Intermittent claudication and ankle- I70.431 DX ATHEROSCLEROSIS OF AUTOLOGOUS VEIN BYPASS GRAFT(S) OF THE RIGHT LEG WITH ULCERATION OF The brachial index < 0.9 | HIGH |
| 5.3.1 Intermittent claudication and ankle- I70.432 DX ATHEROSCLEROSIS OF AUTOLOGOUS VEIN BYPASS GRAFT(S) OF THE RIGHT LEG WITH ULCERATION OF CA brachial index < 0.9 | ALF |
| 5.3.1 Intermittent claudication and ankle- I70.433 DX ATHEROSCLEROSIS OF AUTOLOGOUS VEIN BYPASS GRAFT(S) OF THE RIGHT LEG WITH ULCERATION OF AN brachial index < 0.9 | NKLE |
| 5.3.1 Intermittent claudication and ankle- I70.434 DX ATHEROSCLEROSIS OF AUTOLOGOUS VEIN BYPASS GRAFT(S) OF THE RIGHT LEG WITH ULCERATION OF HE brachial index < 0.9 | EEL AND MIDFOOT |
| 5.3.1 Intermittent claudication and ankle- I70.435 DX ATHEROSCLEROSIS OF AUTOLOGOUS VEIN BYPASS GRAFT(S) OF THE RIGHT LEG WITH ULCERATION OF OT brachial index < 0.9 | THER PART OF FOOT |
| 5.3.1 Intermittent claudication and ankle- I70.438 DX ATHEROSCLEROSIS OF AUTOLOGOUS VEIN BYPASS GRAFT(S) OF THE RIGHT LEG WITH ULCERATION OF OT brachial index < 0.9 | THER PART OF LOWER LEG |
| 5.3.1 Intermittent claudication and ankle- I70.439 DX ATHEROSCLEROSIS OF AUTOLOGOUS VEIN BYPASS GRAFT(S) OF THE RIGHT LEG WITH ULCERATION OF UNbrachial index < 0.9 | NSPECIFIED SITE |
| 5.3.1 Intermittent claudication and ankle- I70.441 DX ATHEROSCLEROSIS OF AUTOLOGOUS VEIN BYPASS GRAFT(S) OF THE LEFT LEG WITH ULCERATION OF THI brachial index < 0.9 | IIGH |
| 5.3.1 Intermittent claudication and ankle- I70.442 DX ATHEROSCLEROSIS OF AUTOLOGOUS VEIN BYPASS GRAFT(S) OF THE LEFT LEG WITH ULCERATION OF CAI brachial index < 0.9 | ιLF |
| 5.3.1 Intermittent claudication and ankle- I70.443 DX ATHEROSCLEROSIS OF AUTOLOGOUS VEIN BYPASS GRAFT(S) OF THE LEFT LEG WITH ULCERATION OF ANI brachial index < 0.9 | IKLE |
| 5.3.1 Intermittent claudication and ankle- I70.444 DX ATHEROSCLEROSIS OF AUTOLOGOUS VEIN BYPASS GRAFT(S) OF THE LEFT LEG WITH ULCERATION OF HEE brachial index < 0.9 | EL AND MIDFOOT |
| 5.3.1 Intermittent claudication and ankle- I70.445 DX ATHEROSCLEROSIS OF AUTOLOGOUS VEIN BYPASS GRAFT(S) OF THE LEFT LEG WITH ULCERATION OF OTHe brachial index < 0.9 | HER PART OF FOOT |
| 5.3.1 Intermittent claudication and ankle- I70.448 DX ATHEROSCLEROSIS OF AUTOLOGOUS VEIN BYPASS GRAFT(S) OF THE LEFT LEG WITH ULCERATION OF OTHe brachial index < 0.9 | HER PART OF LOWER LEG |
| 5.3.1 Intermittent claudication and ankle- I70.449 DX ATHEROSCLEROSIS OF AUTOLOGOUS VEIN BYPASS GRAFT(S) OF THE LEFT LEG WITH ULCERATION OF UNSbrachial index < 0.9 | ISPECIFIED SITE |
| 5.3.1 Intermittent claudication and ankle- I70.45 DX ATHEROSCLEROSIS OF AUTOLOGOUS VEIN BYPASS GRAFT(S) OF OTHER EXTREMITY WITH ULCERATION brachial index < 0.9 | |
| 5.3.1 Intermittent claudication and ankle- I70.461 DX ATHEROSCLEROSIS OF AUTOLOGOUS VEIN BYPASS GRAFT(S) OF THE EXTREMITIES WITH GANGRENE, RIGI brachial index < 0.9 | HTLEG |


| OPEN APPROACH | JBSTITUTE, ICD-10-PCS |
|---|---|
| 17 Cardiovascular event or intervention < 60 days prior to screening 05190KY PX BYPASS RIGHT BRACHIAL VEIN TO UPPER VEIN WITH NONAUTOLOG SUBSTITUTE. OPEN APPROACH | OUS TISSUE ICD-10-PCS |
| 17 Cardiovascular event or intervention <60 days prior to screening 05190ZY PX BYPASS RIGHT BRACHIAL VEIN TO UPPER VEIN, OPEN APPROACH | ICD-10-PCS |
| 17 Cardiovascular event or intervention <60 days prior to screening 051947Y PX BYPASS RIGHT BRACHIAL VEIN TO UPPER VEIN WITH AUTOLOGOUS SUBSTITUTE, PERCUTANEOUS ENDOSCOPIC APPROACH | |
| 17 Cardiovascular event or intervention <60 days prior to screening 051949Y PX BYPASS RIGHT BRACHIAL VEIN TO UPPER VEIN WITH AUTOLOGOUS TISSUE, PERCUTANEOUS ENDOSCOPIC APPROACH | S VENOUS ICD-10-PCS |
| 17 Cardiovascular event or intervention <60 days prior to screening O5194AY PX BYPASS RIGHT BRACHIAL VEIN TO UPPER VEIN WITH AUTOLOGOUS TISSUE, PERCUTANEOUS ENDOSCOPIC APPROACH | S ARTERIAL ICD-10-PCS |
| 17 Cardiovascular event or intervention <60 days prior to screening O5194JY PX BYPASS RIGHT BRACHIAL VEIN TO UPPER VEIN WITH SYNTHETIC SU PERCUTANEOUS ENDOSCOPIC APPROACH | UBSTITUTE, ICD-10-PCS |
| 17 Cardiovascular event or intervention <60 days prior to screening 05194KY PX BYPASS RIGHT BRACHIAL VEIN TO UPPER VEIN WITH NONAUTOLOG SUBSTITUTE, PERCUTANEOUS ENDOSCOPIC APPROACH | OUS TISSUE ICD-10-PCS |
| 17 Cardiovascular event or intervention <60 days prior to screening O5194ZY PX BYPASS RIGHT BRACHIAL VEIN TO UPPER VEIN, PERCUTANEOUS EN APPROACH | NDOSCOPIC ICD-10-PCS |
| 17 Cardiovascular event or intervention <60 days prior to screening 051A07Y PX BYPASS LEFT BRACHIAL VEIN TO UPPER VEIN WITH AUTOLOGOUS TO SUBSTITUTE. OPEN APPROACH | TISSUE ICD-10-PCS |
| 17 Cardiovascular event or intervention <60 days prior to screening 051A09Y PX BYPASS LEFT BRACHIAL VEIN TO UPPER VEIN WITH AUTOLOGOUS VEIN TISSUE, OPEN APPROACH | VENOUS ICD-10-PCS |
| 17 Cardiovascular event or intervention <60 days prior to screening 051A0AY PX BYPASS LEFT BRACHIAL VEIN TO UPPER VEIN WITH AUTOLOGOUS AT TISSUE. OPEN APPROACH | ARTERIAL ICD-10-PCS |
| 17 Cardiovascular event or intervention <60 days prior to screening 051A0JY PX BYPASS LEFT BRACHIAL VEIN TO UPPER VEIN WITH SYNTHETIC SUB- | BSTITUTE, ICD-10-PCS |
| OPEN APPROACH 17 Cardiovascular event or intervention <60 days prior to screening 051A0KY PX BYPASS LEFT BRACHIAL VEIN TO UPPER VEIN WITH NONAUTOLOGO SUBSTITUTE. OPEN APPROACH | OUS TISSUE ICD-10-PCS |
| 17 Cardiovascular event or intervention <60 days prior to screening 051A0ZY PX BYPASS LEFT BRACHIAL VEIN TO UPPER VEIN, OPEN APPROACH | ICD-10-PCS |
| 17 Cardiovascular event or intervention <60 days prior to screening 051A47Y PX BYPASS LEFT BRACHIAL VEIN TO UPPER VEIN WITH AUTOLOGOUS | TISSUE ICD-10-PCS |
| 17 Cardiovascular event or intervention <60 days prior to screening O51A49Y PX SUBSTITUTE, PERCUTANEOUS ENDOSCOPIC APPROACH BYPASS LEFT BRACHIAL VEIN TO UPPER VEIN WITH AUTOLOGOUS VEIN COMMON APPROACH ENDOSCOPIC APPROACH | VENOUS ICD-10-PCS |
| TISSUE, PERCUTANEOUS ENDOSCOPIC APPROACH 17 Cardiovascular event or intervention <60 days prior to screening 051A4AY PX HENDOSCOPIC APPROACH TISSUE, PERCUTANEOUS ENDOSCOPIC APPROACH TISSUE, PERCUTANEOUS ENDOSCOPIC APPROACH | ARTERIAL ICD-10-PCS |
| 17 Cardiovascular event or intervention <60 days prior to screening 051A4JY PX BYPASS LEFT BRACHIAL VEIN TO UPPER VEIN WITH SYNTHETIC SUB- | BSTITUTE, ICD-10-PCS |
| PERCUTANEOUS ENDOSCOPIC APPROACH 17 Cardiovascular event or intervention <60 days prior to screening 051A4KY PX BYPASS LEFT BRACHIAL VEIN TO UPPER VEIN WITH NONAUTOLOGO SUBSTITUTE, PERCUTANEOUS ENDOSCOPIC APPROACH | OUS TISSUE ICD-10-PCS |
| 17 Cardiovascular event or intervention <60 days prior to screening 051A4ZY PX BYPASS LEFT BRACHIAL VEIN TO UPPER VEIN, PERCUTANEOUS ENL APPROACH | DOSCOPIC ICD-10-PCS |
| 17 Cardiovascular event or intervention <60 days prior to screening 051B07Y PX BYPASS RIGHT BASILIC VEIN TO UPPER VEIN WITH AUTOLOGOUS TI SUBSTITUTE. OPEN APPROACH | ISSUE ICD-10-PCS |
| 17 Cardiovascular event or intervention <60 days prior to screening 051B09Y PX BYPASS RIGHT BASILIC VEIN TO UPPER VEIN WITH AUTOLOGOUS VE | ENOUS ICD-10-PCS |
| TISSUE, OPEN APPROACH 17 Cardiovascular event or intervention <60 days prior to screening 051B0AY PX BYPASS RIGHT BASILIC VEIN TO UPPER VEIN WITH AUTOLOGOUS AI BYPASS RIGHT BASILIC VEIN TO UPPER VEIN WITH AUTOLOGOUS AI | RTERIAL ICD-10-PCS |
| TISSUE, OPEN APPROACH 17 Cardiovascular event or intervention <60 days prior to screening 051B0JY PX BYPASS RIGHT BASILIC VEIN TO UPPER VEIN WITH SYNTHETIC SUBS | STITUTE, ICD-10-PCS |
| 17 Cardiovascular event or intervention <60 days prior to screening 051B0KY PX 051B0KY PX BYPASS RIGHT BASILIC VEIN TO UPPER VEIN WITH NONAUTOLOGOL | US TISSUE ICD-10-PCS |
| SUBSTITUTE, OPEN APPROACH | 100 40 000 |
| 17 Cardiovascular event or intervention <60 days prior to screening 051B0ZY PX BYPASS RIGHT BASILIC VEIN TO UPPER VEIN, OPEN APPROACH 17 Cardiovascular event or intervention <60 days prior to screening 051B47Y PX BYPASS RIGHT BASILIC VEIN TO UPPER VEIN WITH AUTOLOGOUS TI | ICD-10-PCS<br>ISSUE ICD-10-PCS |
| SUBSTITUTE, PERCUTANEOUS ENDOSCOPIC APPROACH | 330E 10D-10-1 C3 |
| 17 Cardiovascular event or intervention <60 days prior to screening 051B49Y PX BYPASS RIGHT BASILIC VEIN TO UPPER VEIN WITH AUTOLOGOUS VEIN TISSUE, PERCUTANEOUS ENDOSCOPIC APPROACH | ENOUS ICD-10-PCS |
| 17 Cardiovascular event or intervention <60 days prior to screening 051B4AY PX BYPASS RIGHT BASILIC VEIN TO UPPER VEIN WITH AUTOLOGOUS AI TISSUE, PERCUTANEOUS ENDOSCOPIC APPROACH | RTERIAL ICD-10-PCS |
| 17 Cardiovascular event or intervention <60 days prior to screening O51B4JY PX BYPASS RIGHT BASILIC VEIN TO UPPER VEIN WITH SYNTHETIC SUBSTANCE OF SUBSTANCE O | STITUTE, ICD-10-PCS |
| 17 Cardiovascular event or intervention <60 days prior to screening 051B4KY PX BYPASS RIGHT BASILIC VEIN TO UPPER VEIN WITH NONAUTOLOGOL SUBSTITUTE, PERCUTANEOUS ENDOSCOPIC APPROACH | US TISSUE ICD-10-PCS |
| 17 Cardiovascular event or intervention <60 days prior to screening 051B4ZY PX BYPASS RIGHT BASILIC VEIN TO UPPER VEIN, PERCUTANEOUS ENDO APPROACH | OSCOPIC ICD-10-PCS |
| 17 Cardiovascular event or intervention <60 days prior to screening 051C07Y PX BYPASS LEFT BASILIC VEIN TO UPPER VEIN WITH AUTOLOGOUS TIS SUBSTITUTE, OPEN APPROACH | SSUE ICD-10-PCS |
| 17 Cardiovascular event or intervention <60 days prior to screening 051C09Y PX BYPASS LEFT BASILIC VEIN TO UPPER VEIN WITH AUTOLOGOUS VEINT TISSUE. OPEN APPROACH | NOUS ICD-10-PCS |
| 17 Cardiovascular event or intervention <60 days prior to screening 051C0AY PX BYPASS LEFT BASILIC VEIN TO UPPER VEIN WITH AUTOLOGOUS AR TISSUE, OPEN APPROACH | RTERIAL ICD-10-PCS |


#### Appendix 3. Flowchart for cohort assembly

| | Excluded Patients | Remaining Patients |
|---|---|---|
| Patients in dataset | | 96,791,997 |
| Patients meeting cohort entry criteria | | 705,899 |
| Excluded due to insufficient enrollment | -198,502 (28%) | 507,397 |
| Excluded due to prior use of referent | -137,947 (27%) | 369,450 |
| Excluded due to prior use of exposure | -268,183 (73%) | 101,267 |
| Excluded because patient qualified in >1 exposure category | -11 (<1%) | 101,256 |
| Excluded based on 1 - Age | -3,583 (4%) | 97,673 |
| Excluded based on 1 - Gender | -11 (<1%) | 97,662 |
| Excluded based on 2 - Type 2 diabetes mellitus | -10,623 (11%) | 87,039 |
| Excluded based on 4 - BMI ≥ 25kg/m2 (ICD-10) | -17,659 (20%) | 69,380 |
| Excluded based on 4 - BMI ≥ 25kg/m2 (Truncated) | -582 (<1%) | 68,798 |
| Excluded based on 5 - Established atherosclerotic cardiovascular disease | -16,249 (24%) | 52,549 |
| Excluded based on 7 - Planning treatment for diabetic retinopathy and/or macular edema | -786 (1%) | 51,763 |
| Excluded based on 8 - Hospitalized for chronic heart failure within 2 months prior to screening | -191 (<1%) | 51,572 |
| Excluded based on 11 - History of chronic or acute pancreatitis | -302 (<1%) | 51,270 |
| Excluded based on 12 - Known clinically significant gastric emptying abnormality or bariatric surgery | -2,942 (6%) | 48,328 |
| Excluded based on 13 - Liver disease (not including non-alcoholic fatty liver disease [NAFLD]) or ALT level ≥3X the ULN | -314 (<1%) | 48,014 |
| Excluded based on 14 - eGFR <15 mL/Min/1.73 m2 or on chronic dialysis | -381 (<1%) | 47,633 |
| Excluded based on 15 - Family or personal history of multiple endocrine neoplasia or medullary thyroid carcinoma | -79 (<1%) | 47,554 |
| Excluded based on 17 - Cardiovascular event or intervention < 60 days prior to screening | -221 (<1%) | 47,333 |
| Excluded based on 18 - GLP-1-RA or pramlintide treatment within 3 months prior to Visit 1 | -3,735 (8%) | 43,598 |
| Excluded based on 19 - Women who are pregnant or breastfeeding | -2 (<1%) | 43,596 |
| Patients in Exposure Group | | 29,761 |
| Patients in Referent Group | | 13,835 |
| Total Patients | | 43,596 |

| MARKETSCAN (May 13, 2022 to Dec 31, 2023) | Evaluded Patients | Remaining Patients |
|---|---|---|
| Patients in dataset | Excluded Fatients | 126.118.01 |
| Patients meeting cohort entry criteria | | 292.14 |
| Excluded due to insufficient enrollment | -53.707 (18%) | 238,440 |
| Excluded due to prior use of referent | -91.632 (38%) | 146.80 |
| Excluded due to prior use of exposure | -105,424 (72%) | 41,38- |
| Excluded because patient qualified in >1 exposure category | -7 (<1%) | 41,37 |
| Excluded based on 1 - Age | -4,046 (10%) | 37,33 |
| Excluded based on 1 - Gender | -0 (<1%) | 37,33 |
| Excluded based on 2 - Type 2 diabetes mellitus | -5,682 (15%) | 31,64 |
| Excluded based on 4 - BMI ≥ 25kg/m2 | -8,718 (28%) | 22,93 |
| Excluded based on 5 - Established atherosclerotic cardiovascular disease | -10,471 (46%) | 12,460 |
| Excluded based on 7 - Planning treatment for diabetic retinopathy and/or macular edema | -204 (2%) | 12,25 |
| Excluded based on 8 - Hospitalized for chronic heart failure within 2 months prior to screening | -69 (<1%) | 12,18 |
| Excluded based on 11 - History of chronic or acute pancreatitis | -60 (<1%) | 12,12 |
| Excluded based on 12 - Known clinically significant gastric emptying abnormality or bariatric surgery | -764 (6%) | 11,36 |
| Excluded based on 13 - Liver disease (not including non-alcoholic fatty liver disease (NAFLDI)) or ALT level ≥3X the ULN | -62 (<1%) | 11,30 |
| Excluded based on 14 - eGFR <15 mL/Min/1.73 m2 or on chronic dialysis | -72 (<1%) | 11,22 |
| Excluded based on 15 - Family or personal history of multiple endocrine neoplasia or medullary thyroid carcinoma | -36 (<1%) | 11,19: |
| Excluded based on 17 - Cardio vascular event or intervention < 60 days prior to screening | -69 (<1%) | 11,12 |
| Excluded based on 18 - GLP-1-RA or pramlintide treatment within 3 months prior to Visit 1 | -1,678 (15%) | 9,44 |
| Excluded based on 19 - Women who are pregnant or breastfeeding | -4 (<1%) | 9,442 |
| Patients in Exposure Group | | 5,610 |
| Patients in Referent Group | | 3,83 |
| Total Patients | | 9,442 |

#### Appendix 4.1st Feasibility Assessment

#### Table of Contents

- A. Patient characteristics by treatment group
- B. Summary Parameters of Study Population
- C. Median Follow up Time in Overall Study Population
- D. Reasons for Censoring in Overall Study Population
- E. Initial Power Assessment
- F. Aetion report link
- G. Review by Principal Investigator

In order to complete the initial power analysis, a dummy outcome of a 90-day gap in database enrollment was used. This outcome is used to ensure that no information on the comparative risks of the outcomes of interest are available at this stage. We completed a PS overlap weighted comparative analysis using this outcome. The PS included only 3 covariates: age, sex, and combined comorbidity index. Power calculations are based on the formulas from Chow et al. (2008).

OPTUM: Study period from May 13, 2022 to May 31, 2025 MARKETSCAN: Study period from May 13, 2022 to Dec 31, 2023

#### A. Patient characteristics by treatment group (follow-up start is 1 days after CED, so few patients and dropped, hence table 1 could include sightly fewer patients than the attrition table)

| Before weighting | | Optum | | Marketscan | | |
|---|---|---|---|---|---|---|
| Variable | Reference: Dulaglutide | Exposure: Tirzepatide | Difference | Reference: Dulaglutide | Exposure: Tirzepatide | Difference |
| Number of patients | 13,793 | 29,744 | - (-, -) | 5,329 | 5,116 | - (-, -) |
| Age | | | | | | |
| mean (sd) | 73.95 (7.67) | 66.65 (9.20) | 7.30 (7.13, 7.46) | 63.74 (10.60) | 59.86 (9.36) | 3.88 (3.50, 4.26) |
| median [IQR] | 74.00 [69.00, 79.00] | 68.00 [61.00, 73.00] | - (-, -) | 63.00 [56.00, 72.00] | 59.00 [53.00, 65.00] | - (-, -) |
| Gender | | | | | | |
| Male; n (%) | 6,699 (48.6%) | 14,518 (48.8%) | -0.2% (-1.3%, 0.8%) | 2,885 (54.1%) | 2,538 (49.6%) | 4.5% (2.6%, 6.5%) |
| CCI (365 days) | | | | | | |
| mean (sd) | 3.64 (3.09) | 2.84 (2.66) | 0.81 (0.75, 0.87) | 2.34 (2.50) | 1.78 (2.02) | 0.57 (0.48, 0.65) |
| median [IQR] | 3.00 [1.00, 5.00] | 2.00 [1.00, 4.00] | - (-, -) | 2.00 [1.00, 3.00] | 1.00 [0.00, 3.00] | - (-, -) |

### B. Summary Parameters of Overall Study Population (Step 1)

| | Optum | Marketscan |
|-----------------------------------------------------|----------|------------|
| Variable | Value | Value |
| Number of patients in full cohort | 43,596 | 9,442 |
| Number of patients dropped as incomplete cases | 0 | 0 |
| Number of patients that did not begin follow-up | 59 | 8 |
| Number of patients in analytic cohort | 43,537 | 9,434 |
| Number of events | 322 | 88 |
| Number of person-years | 22,000,1 | 4,052.00 |
| Number of patients in group: Reference: Sitagliptin | 13,793 | 3,825 |
| Number of patients in group: Exposure: Tirzepatide | 29,744 | 5,609 |

#### C. Median Follow up Time in Overall Study Population (Step 1)

| | Optum | Marketscan |
|----------------------------|-------------------|-------------------|
| Patient Group | Median Follow-Up | Median Follow-Up |
| ratient di oup | Time (Days) [IQR] | Time (Days) [IQR] |
| Overall Patient Population | 145 [75, 297] | 133 [71, 231] |

### D. Reasons for Censoring in Overall Study Population (Step 1)

| | Optum | Marketscan |
|---|---|---|
| Overall | Value | Value |
| Outcome | 322 (0.7%) | 88 (0.9%) |
| Start of an additional exposure | 341 (0.8%) | 97 (1.0%) |
| End of index exposure | 16,757 (38.5%) | 2,397 (25.4%) |
| Maximum follow-up time | 8,118 (18.6%) | 773 (8.2%) |
| Specified date reached | 10,456 (24.0%) | 4,917 (52.1%) |
| End of patient data | 0 (0.0%) | 0 (0.0%) |
| End of patient enrollment | 4,150 (9.5%) | 563 (6.0%) |
| Switch to other GLP-1-RA (for censoring) / Nursing home admission | 3,029 (7.0%) | 577 (6.1%) |

#### E. Power Assessment

| Superiority Analysis | Optum | Marketscan | Pooled |
|---------------------------|--------|------------|--------|
| Number of patients | | | |
| Reference | 9,834 | 2,442 | 12,276 |
| Exposed | 15,677 | 3,375 | 19,052 |
| Risk per 1,000 patients | 14.64 | 21.72 | 15.89 |
| Expected HR | 0.75 | 0.75 | 0.75 |
| Alpha (2-sided) | 0.05 | 0.05 | 0.05 |
| Number of events expected | 373 | 126 | 498 |
| Power | 0.79 | 0.37 | 0.89 |

## F. Aetion report link

Optum Step 1: https://bwh-dope.aetion.com/project/2951/rwrs/142679 Marketscan Step 1: https://bwh-dope.aetion.com/project/2950/rwrs/142680

## F. Review by principal investigator

Stop analyses until feasibility and power are reviewed by primary investigators.

| Reviewed by PI: | Nils Krüger | Date reviewed: | September 25, 2025 |
|-----------------|-------------|----------------|--------------------|

## Appendix 5. 2nd Feasibility Assessment

### **Table of Contents**

- A. Median Follow up Time by Treatment Group
- B. Reasons for Censoring by Treatment Group
- C. Final Power Assessment
- D. Aetion report link
- E. Review by Principal Investigator

In order to complete the feasibility analysis, a dummy outcome of a 90-day gap in database enrollment was used. This outcome is used to ensure that no information on the comparative risks of the outcomes of interest are available at this stage. We completed a PS overlap weighted comparative analysis using this outcome. The PS included all prespecified covariates listed in the protocol. Power calculations are based on the formulas from Chow et al. (2008).

# A. Median Follow Up Time by Treatment Group

| Patient Group | Median Follow-Up Time (Days) [IQR] | Median Follow-Up<br>Time (Days) [IQR] |
|---|---|---|
| Overall Patient Population | 145 [75, 297] | 133 [71, 231] |

# B. Reasons for Censoring in Overall Study Population

| | Optum | Marketscan |
|---|---|---|
| Overall | Value | Value |
| Outcome | 322 (0.7%) | 88 (0.9%) |
| Start of an additional exposure | 341 (0.8%) | 97 (1.0%) |
| End of index exposure | 16,757 (38.5%) | 2,397 (25.4%) |
| Maximum follow-up time | 8,118 (18.6%) | 773 (8.2%) |
| Specified date reached | 10,456 (24.0%) | 4,917 (52.1%) |
| End of patient data | 0 (0.0%) | 0 (0.0%) |
| End of patient enrollment | 4,150 (9.5%) | 563 (6.0%) |
| Switch to other GLP-1-RA (for censoring) / Nursing home admission | 3,029 (7.0%) | 577 (6.1%) |

### C. Power Assessment

| Superiority Analysis | Optum | Marketscan | Pooled |
|---------------------------|--------|------------|--------|
| Number of patients | | | |
| Reference | 9,834 | 2,442 | 12,276 |
| Exposed | 15,677 | 3,375 | 19,052 |
| Risk per 1,000 patients | 14.64 | 21.72 | 15.89 |
| Expected HR | 0.75 | 0.75 | 0.75 |
| Alpha (2-sided) | 0.05 | 0.05 | 0.05 |
| Number of events expected | 373 | 126 | 498 |
| Power | 0.79 | | |

# D. Aetion report link

Optum Step 1: https://bwh-dope.aetion.com/project/2951/rwrs/142679

Marketscan Step 1: https://bwh-dope.aetion.com/project/2950/rwrs/142680

# E. Review by principal investigator

Stop analyses until feasibility and power are reviewed by primary investigators.

| Reviewed by PI: | Nils Krüger | Date reviewed: | September 25, 2025 |
|-----------------|-------------|----------------|--------------------|

## Appendix 6. Balance Assessment - PS Distribution and C-Statistic

### C-statistics unadjusted, OPTUM: 0.823



### C-statistics adjusted after overlap weighing on the PS, OPTUM: 0.505



## C-statistics unadjusted, MARKETSCAN: 0.822



## C-statistics adjusted after overlap weighing on the PS, MARKETSCAN: 0.505



### Appendix 7. Balance Assessment - Table 1

| OPTUM | | | | I |
|---|---|---|---|---|
| Variable | Reference: Sitagliptin | Exposure: Tirzepatide | Reference: Sitagliptin | Exposure: Tirzepatide |
| Number of patients | 13.970 | | 13.793 | 29.744 |
| Sum of weights | 13,970 | 20,263 | 6,027.46 | 6,027.46 |
| Effective sample size | | | 9,834 | 15,677 |
| Age | | | 3,834 | 15,077 |
| mean (sd) | 73.95 (7.67) | 66.65 (9.20) | 71.37 (7.77) | 71.37 (7.57) |
| Gender (male); n (%) | 6.699 (48.6%) | 14.518 (48.8%) | 2,899.0 (48.1%) | 2,899.0 (48.1%) |
| Race | 0,033 (48:0%) | 14,518 (48.8%) | 2,833.0 (48.1%) | 2,899.0 (48.1%) |
| White; n (%) | 8,030 (58.2%) | 18,967 (63.8%) | 3,751.3 (62.2%) | 3,751.3 (62.2%) |
| Black: n (%) | 2.806 (20.3%) | 4.186 (14.1%) | 1.073.5 (17.8%) | 1.073.5 (17.8%) |
| Unknown / Missing; n (%) | 2,478 (18.0%) | 6,134 (20.6%) | 1,063.0 (17.6%) | 1,063.0 (17.6%) |
| Others: n (%) | 479 (3.5%) | 457 (1.5%) | 139.7 (2.3%) | 139.7 (2.3%) |
| Region/ State | 47 3 (3.370) | 437 (1.370) | 155.7 (2.570) | 155.7 (2.570) |
| Northest; n (%) | 1,855 (13.4%) | 2,523 (8.5%) | 645.4 (10.7%) | 645.4 (10.7%) |
| Midwest / North central; n (%) | 2,152 (15.6%) | 5,933 (19.9%) | 1,039.3 (17.2%) | 1,039.3 (17.2%) |
| South; n (%) | 7,684 (55.7%) | 17,385 (58.4%) | 3,472.4 (57.6%) | 3,472.4 (57.6%) |
| West; n(%) | 2,092 (15.2%) | 3,884 (13.1%) | 866.1 (14.4%) | 866.1 (14.4%) |
| Missing; n (%) | 10 (0.1%) | 19 (0.1%) | 4.2 (0.1%) | 4.2 (0.1%) |
| Smoking/Tobacco use; n (%) | 3.847 (27.9%) | 8.616 (29.0%) | 1.732.4 (28.7%) | 1.732.4 (28.7%) |
| Weight | 3,047 (27.370) | 0,010 (23.0 /0) | 1,1 32.7 (20.1 /0) | 1,1 32.7 (20.1 /0) |
| Overweight; n (%) | 3,104 (22.5%) | 1,893 (6.4%) | 808.3 (13.4%) | 808.3 (13.4%) |
| Class 1 Obesity; n (%) | 4,150 (30.1%) | 5,950 (20.0%) | 1,647.7 (27.3%) | 1,647.7 (27.3%) |
| Class 2 Obesity; n (%) | 3,720 (27.0%) | 10,508 (35.3%) | 1,960.3 (32.5%) | 1,960.3 (32.5%) |
| Class 3 Obesity; n(%) | 1,443 (10.5%) | 7,750 (26.1%) | 935.1 (15.5%) | 935.1 (15.5%) |
| Unspecified Obesity; n(%) | 1,376 (10.0%) | 3,643 (12.2%) | 676.0 (11.2%) | 676.0 (11.2%) |
| Diabetic retinopathy; n (%) | 1,759 (12.8%) | 3.319 (11.2%) | 738.0 (12.2%) | 738.0 (12.2%) |
| Diabetic neuropathy; n (%) | 5,337 (38.7%) | 9.824 (33.0%) | 2,226.9 (37.0%) | 2.226.9 (37.0%) |
| Diabetic nephropathy: n (%) | 5.198 (37.7%) | 8.040 (27.0%) | 2,004.3 (33.3%) | 2,004.3 (33.3%) |
| Diabetes with other ophthalmic complications; n (%) | 1,043 (7.6%) | 1,376 (4.6%) | 386.2 (6.4%) | 386.2 (6.4%) |
| Diabetes with peripheral circulatory disorders; n (%) | 3.722 (27.0%) | 6,013 (20.2%) | 1,447.6 (24.0%) | 1,447.6 (24.0%) |
| Diabetic foot; n(%) | 587 (4.3%) | 1.201 (4.0%) | 249.7 (4.1%) | 249.7 (4.1%) |
| Erectile dysfunction; n (%) | 642 (4.7%) | 1,722 (5.8%) | 310.0 (5.1%) | 310.0 (5.1%) |
| Hypoglycemia; n (%) | 4,267 (30.9%) | 8,127 (27.3%) | 1,763.1 (29.3%) | 1,763.1 (29.3%) |
| Hyperglycemia/DKA/HONK; n (%) | 7,494 (54.3%) | 15,277 (51.4%) | 3,196.7 (53.0%) | 3,196.7 (53.0%) |
| Skin infections; n (%) | 1,580 (11.5%) | 3,699 (12.4%) | 711.4 (11.8%) | 711.4 (11.8%) |
| Stable angina; n (%) | 1.275 (9.2%) | 2.946 (9.9%) | 580.1 (9.6%) | 580.1 (9.6%) |
| Unstable angina; n (%) | 593 (4.3%) | 1,342 (4.5%) | 262.4 (4.4%) | 262.4 (4.4%) |
| Hypertension; n (%) | 13,088 (94.9%) | 27,506 (92.5%) | 5,681.7 (94.3%) | 5,681.7 (94.3%) |
| Hypotension; n (%) | 883 (6.4%) | 1,287 (4.3%) | 320.8 (5.3%) | 320.8 (5.3%) |
| Hyperlipidemia; n (%) | 12,534 (90.9%) | 26,680 (89.7%) | 5,469.4 (90.7%) | 5,469.4 (90.7%) |
| Atrial fibrillation; n (%) | 2,611 (18.9%) | 5,104 (17.2%) | 1,099.6 (18.2%) | 1,099.6 (18.2%) |
| Cardiac conduction disorder; n (%) | 1,552 (11.3%) | 2,828 (9.5%) | 630.9 (10.5%) | 630.9 (10.5%) |
| Previous cardiac procedure (CABG, PTCA, Stent); n (%) | 334 (2.4%) | 824 (2.8%) | 157.0 (2.6%) | 157.0 (2.6%) |
| Ischemic stroke; n(%) | 217 (1.6%) | 280 (0.9%) | 73.3 (1.2%) | 73.3 (1.2%) |
| PVD diagnosis or surgery; n (%) | 3,375 (24.5%) | 5,515 (18.5%) | 1,313.2 (21.8%) | 1,313.2 (21.8%) |
| Other cardiac dysrhythmia; n (%) | 4,215 (30.6%) | 8,680 (29.2%) | 1,785.7 (29.6%) | 1,785.7 (29.6%) |
| Cardiomyopathy; n (%) | 1,236 (9.0%) | 2,549 (8.6%) | 534.5 (8.9%) | 534.5 (8.9%) |
| Valve disorders; n (%) | 2,870 (20.8%) | 5,355 (18.0%) | 1,191.3 (19.8%) | 1,191.3 (19.8%) |
| Valve replacement; n (%) | 347 (2.5%) | 672 (2.3%) | 151.5 (2.5%) | 151.5 (2.5%) |
| TIA; n(%) | 530 (3.8%) | 857 (2.9%) | 201.3 (3.3%) | 201.3 (3.3%) |
| Edema; n (%) | 2,564 (18.6%) | 5,387 (18.1%) | 1,101.5 (18.3%) | 1,101.5 (18.3%) |
| Venous thromboembolism / Pulmonary embolism; n (%) | 702 (5.1%) | 1,387 (4.7%) | 285.4 (4.7%) | 285.4 (4.7%) |
| Pulmonary hypertension; n (%) | 787 (5.7%) | 1,424 (4.8%) | 314.3 (5.2%) | 314.3 (5.2%) |
| Implantable cardioverter defibrillator; n (%) | 53 (0.4%) | 146 (0.5%) | 27.1 (0.4%) | 27.1 (0.4%) |
| Hyperkalemia; n (%) | 852 (6.2%) | 1,184 (4.0%) | 304.4 (5.1%) | 304.4 (5.1%) |
| Coronary atherosclerosis; n (%) | 6,176 (44.8%) | 13,983 (47.0%) | 2,785.0 (46.2%) | 2,785.0 (46.2%) |
| Cerebrovascular procedure; n (%) | 40 (0.3%) | 60 (0.2%) | 14.8 (0.2%) | 14.8 (0.2%) |
| Insertion of pacemakers / removal of cardiac lead; n (%) | 64 (0.5%) | 74 (0.2%) | 21.3 (0.4%) | 21.3 (0.4%) |

| CKD Stage 1-2; n (%) | 1.256 (9.1%) | 2.025 (6.8%) | 505.9 (8.4%) | 505.9 (8.4%) |
|---|---|---|---|---|
| CKD Stage 3-4; n(%) | 4,247 (30.8%) | 6,403 (21.5%) | 1,638.6 (27.2%) | 1,638.6 (27.2%) |
| Unspecified CKD; n (%) | 1.800 (13.1%) | 2,543 (8.5%) | 654.1 (10.9%) | 654.1 (10.9%) |
| Acute kidney injury: n (%) | 1.862 (13.5%) | 2,387 (8.0%) | 635.4 (10.5%) | 635.4 (10.5%) |
| Hypertensive nephropathy; n (%) | 3,582 (26.0%) | 5,317 (17.9%) | 1,365.5 (22.7%) | 1,365.5 (22.7%) |
| Urinary tract infections; n (%) | 2,902 (21.0%) | 4,703 (15.8%) | 1,123.9 (18.7%) | 1,123.9 (18.7%) |
| Genital infections; n (%) | 406 (2.9%) | 720 (2.4%) | 166.3 (2.8%) | 166.3 (2.8%) |
| Urolithiasis (Kidney and urinary stone); n (%) | 832 (6.0%) | 1,606 (5.4%) | 356.9 (5.9%) | 356.9 (5.9%) |
| COPD; n (%) | 2,762 (20.0%) | 5,169 (17.4%) | 1,180.6 (19.6%) | 1,180.6 (19.6%) |
| Asthma; n (%) | 1,511 (11.0%) | 4,043 (13.6%) | 733.0 (12.2%) | 733.0 (12.2%) |
| Obstructive sleep apnea; n (%) | 3.212 (23.3%) | 12,358 (41.5%) | 1.830.6 (30.4%) | 1.830.6 (30.4%) |
| Serious bacterial infections; n (%) | 840 (6.1%) | 995 (3.3%) | 272.9 (4.5%) | 272.9 (4.5%) |
| Pneumonia; n (%) | 1,079 (7.8%) | 1,674 (5.6%) | 402.1 (6.7%) | 402.1 (6.7%) |
| Liver disease; n(%) | 2.698 (19.6%) | 5,752 (19.3%) | 1.164.5 (19.3%) | 1.164.5 (19.3%) |
| MASH/MASLD; n(%) | 1,034 (7.5%) | 3.105 (10.4%) | 525.2 (8.7%) | 525.2 (8.7%) |
| Fractures / Falls; n (%) | 1,486 (10.8%) | 1,901 (6.4%) | 515.4 (8.6%) | 515.4 (8.6%) |
| Osteoporosis; n(%) | 1,035 (7.5%) | 1,573 (5.3%) | 402.6 (6.7%) | 402.6 (6.7%) |
| Osteoarthritis: n (%) | 4.808 (34.9%) | 10,144 (34.1%) | 2,089.7 (34.7%) | 2,089.7 (34.7%) |
| Depression: n (%) | 2.718 (19.7%) | 6.289 (21.1%) | 1.201.7 (19.9%) | 1.201.7 (19.9%) |
| Dementia; n (%) | 1,752 (12.7%) | 1,292 (4.3%) | 1,201.7 (19.9%)<br>465.8 (7.7%) | 1,201.7 (19.9%)<br>465.8 (7.7%) |
| | , , , , , | | | |
| Delirium or psychosis; n (%) | 394 (2.9%) | 389 (1.3%) | 117.3 (2.0%) | 117.3 (2.0%) |
| Anxiety; n (%) | 2,526 (18.3%) | 6,755 (22.7%) | 1,181.1 (19.6%) | 1,181.1 (19.6%) |
| Sleep disorders; n(%) | 4,942 (35.8%) | 11,677 (39.3%) | 2,236.1 (37.1%) | 2,236.1 (37.1%) |
| Anemia; n (%) | 4,280 (31.0%) | 6,827 (23.0%) | 1,625.9 (27.0%) | 1,625.9 (27.0%) |
| Influenza; n (%) | 265 (1.9%) | 633 (2.1%) | 121.2 (2.0%) | 121.2 (2.0%) |
| COVID; n (%) | 1,596 (11.6%) | 3,110 (10.5%) | 650.3 (10.8%) | 650.3 (10.8%) |
| Hyperthyroidism and other thyroid gland disorders; n (%) | 4,096 (29.7%) | 8,920 (30.0%) | 1,799.1 (29.8%) | 1,799.1 (29.8%) |
| Hypothyroidism; n (%) | 3,283 (23.8%) | 7,054 (23.7%) | 1,433.7 (23.8%) | 1,433.7 (23.8%) |
| Nephrotic syndrome; n (%) | 4 (0.0%) | 34 (0.1%) | 2.5 (0.0%) | 2.5 (0.0%) |
| Urinary incontinence; n (%) | 1,267 (9.2%) | 2,086 (7.0%) | 504.0 (8.4%) | 504.0 (8.4%) |
| Biliary disease; n (%) | 27 (0.2%) | 39 (0.1%) | 10.4 (0.2%) | 10.4 (0.2%) |
| Pancreatitis; n (%) | 4 (0.0%) | 11 (0.0%) | 2.3 (0.0%) | 2.3 (0.0%) |
| Bowel obstruction; n (%) | 26 (0.2%) | 53 (0.2%) | 10.1 (0.2%) | 10.1 (0.2%) |
| Gastroparesis; n (%) | 130 (0.9%) | 281 (0.9%) | 61.5 (1.0 %) | 61.5 (1.0%) |
| Number of antidiabetic drugs on CED | | | | |
| mean (sd) | 1.25 (0.90) | 1.09 (0.97) | 1.22 (0.91) | 1.22 (0.97) |
| Concomitant use or initiation of Metformin; n (%) | 7,516 (54.5%) | 12,987 (43.7%) | 3,074.9 (51.0%) | 3,074.9 (51.0%) |
| Concomitant use or initiation of Insulins; n (%) | 2,085 (15.1%) | 6,749 (22.7%) | 1,122.5 (18.6%) | 1,122.5 (18.6%) |
| Concomitant use or initiation of Sulfonylureas; n (%) | 3,880 (28.1%) | 4,591 (15.4%) | 1,425.5 (23.7%) | 1,425.5 (23.7%) |
| Concomitant use or initiation of DPP-4i; n (%) | 124 (0.9%) | 610 (2.1%) | 67.6 (1.1%) | 67.6 (1.1%) |
| Concomitant use or initiation of SGLT-2i; n (%) | 2,575 (18.7%) | 5,937 (20.0%) | 1,234.8 (20.5%) | 1,234.8 (20.5%) |
| Concomitant use or initiation of Any other glucose-lowering drugs; n (%) | 1,038 (7.5%) | 1,666 (5.6%) | 437.7 (7.3%) | 437.7 (7.3%) |
| Past use of Metformin; n (%) | 8,755 (63.5%) | 17,105 (57.5%) | 3,763.2 (62.4%) | 3,763.2 (62.4%) |
| Past use of Insulins; n (%) | 2,900 (21.0%) | 8,822 (29.7%) | 1,525.8 (25.3%) | 1,525.8 (25.3%) |
| Past use of Sulfonylureas; n (%) | 5,079 (36.8%) | 6,256 (21.0%) | 1,878.1 (31.2%) | 1,878.1 (31.2%) |
| Past use of DPP-4i; n (%) | 373 (2.7%) | 1,004 (3.4%) | 163.7 (2.7%) | 163.7 (2.7%) |
| Past use of SGLT-2i; n (%) | 3,791 (27.5%) | 8,329 (28.0%) | 1,792.7 (29.7%) | 1,792.7 (29.7%) |
| Past use of Any other glucose-lowering drugs; n (%) | 1,462 (10.6%) | 2,407 (8.1%) | 622.1 (10.3%) | 622.1 (10.3%) |
| ACE-is/ARB's; n (%) | 10,334 (74.9%) | 21,664 (72.8%) | 4,516.0 (74.9%) | 4,516.0 (74.9%) |
| ARNI; n (%) | 416 (3.0%) | 1,038 (3.5%) | 199.2 (3.3%) | 199.2 (3.3%) |
| Thiazides; n (%) | 4,354 (31.6%) | 10,043 (33.8%) | 1,983.4 (32.9%) | 1,983.4 (32.9%) |
| Beta-blockers; n (%) | 8,224 (59.6%) | 16,912 (56.9%) | 3,563.0 (59.1%) | 3,563.0 (59.1%) |
| Calcium channel blockers; n (%) | 5,855 (42.4%) | 10,905 (36.7%) | 2,432.9 (40.4%) | 2,432.9 (40.4%) |
| Digoxin / Digitoxin; n (%) | 174 (1.3%) | 267 (0.9%) | 71.2 (1.2%) | 71.2 (1.2%) |
| Loop diuretics; n (%) | 3,598 (26.1%) | 7,919 (26.6%) | 1,610.4 (26.7%) | 1,610.4 (26.7%) |
| Other diuretics; n (%) | 1,318 (9.6%) | 3,641 (12.2%) | 646.1 (10.7%) | 646.1 (10.7%) |
| Intravenous diuretics; n (%) | 301 (2.2%) | 592 (2.0%) | 122.9 (2.0%) | 122.9 (2.0%) |
| Nitrates; n(%) | 1,579 (11.4%) | 3,536 (11.9%) | 717.3 (11.9%) | 717.3 (11.9%) |
| Anti-arrhythmics; n (%) | 537 (3.9%) | 1,285 (4.3%) | 254.8 (4.2%) | 254.8 (4.2%) |
| Statins; n (%) | 11,936 (86.5%) | 24,562 (82.6%) | 5,195.0 (86.2%) | 5,195.0 (86.2%) |
| PCSK9 inhibitors and other lipid-lowering drugs; n (%) | 2,228 (16.2%) | 5,648 (19.0%) | 1,080.3 (17.9%) | 1,080.3 (17.9%) |

| COPPDARTMENT COPP | Oral anticoagulants; n (%) | 2,500 (18.1%) | 4,944 (16.6%) | 1,052.2 (17.5%) | 1,052.2 (17.5%) |
|---|---|---|---|---|---|
| NSADS (n/s) | | | | | |
| Control (Control (C | | | | | |
| Oktooprovise segents forch bisphosophoratesin (Phi) Oktoophosis (Phi) Oktoophosi | | | | | |
| Quadra (PM) | | | | | |
| Anti-depressants (%) Anti-depressants (%) Anti-depressants (%) (674,999) (1228,413%) (2254,437,44%) 2254,437,44%) 2254,4437,44%) 2254,4437,44%) 2254,444% Antiolytic Physroptics berages (%) 2357,844%) 2357,844,844%) 2357,844%) 2357,844%) 2357,844%) 2357,844%) 2357,844%) 2357,844%) 2357,844% 2357,844%) 2357,844% | | | | | |
| Antipoyrontos, n°69 (255) (43%) (255) (44%) (255) (44% | | | | | |
| Amolyptics Improvises Improvises (199) 2,537 (8.44%) 5,966 (5.07%) 5,961 (5.99%) 5,96 | | | | | |
| Demential medications; n (%) | | | | | |
| Ultimary fractimeterions ambinistics; n(%) \$23 (8.8%) \$2.56 (6.507.8%) \$3.00.47 (49.9%) \$3.00.47 (49.9%) \$3.00.47 (49.9%) \$3.30.47 (49.9%) \$3.30.47 (49.9%) \$3.30.47 (49.9%) \$3.30.47 (49.9%) \$3.30.47 (49.9%) \$3.00.47 ( | | | | | |
| Lasthews, n(s) 523 (38%) 1259 (4.3%) 247 0 (4.1%) 247 0 (4.1%) Lasthews, n(s) 155 (6.57) 16.30 (7.11) 16.29 (6.71) Lasthews of latinct medications 15.50 (6.57) 16.30 (7.11) 16.29 (6.71) Lasthews of latinct works 10.78 (7.30) 11.53 (7.55) 11.23 (7.66) 11.23 (7.14) Lasthews of latinct works 10.78 (7.30) 11.53 (7.55) 11.23 (7.66) 11.23 (7.14) Lasthews of latinct works 12.30 (7.66) 12.30 (7.17) Lasthews of latinct works 12.30 (7.66) 12.30 (7.17) Lasthews of latinct works 12.30 (7.66) 12.30 (7.17) Lasthews of latinct works 12.30 (7.67) 12.30 (7.77) Lasthews of latinct works 12.30 (7.77) 12.30 (7.77) Lasthews of latinct works 12.30 (7.77) 12.30 (7.77) Lasthews of latinct works 12.30 (7.77) 12.30 (7.77) Lasthews of latinct works 12.30 (7.79) 12.30 (7.77) Lasthews of latinct works 12.30 (7.79) 12.30 (7.73) Lasthews of latinct works 12.30 (7.79) 12.30 (7.73) Lasthews of latinct works 12.30 (7.79) 12.30 (7.73) Lasthews of latinct works 12.30 (7.73) Lasthews of latinct works 12.30 (7.73) | | | | | |
| Number of distinct medications | | | | | |
| | | 323 (3.370) | 1,203 (1.370) | 2 17.0 (1.170) | 2 17.0 (1.170) |
| Number of office visits | | 15.85 (6.57) | 16 30 (7 11) | 1629 (676) | 1629 (671) |
| Info@sign Info | | 13.33 (6.37) | 10.50 (7.11) | 10.23 (0.7 0) | 10.23 (0.71) |
| Number of endocrinologist vivists | | 10.78 (7.30) | 11 53 <i>(</i> 7 55) | 11 23 (7 66) | 11 23 (7 14) |
| Description | | 10.7 0 (7.50) | 11.03 (7.00) | 11.23 (7.00) | 11.23 (7.11) |
| Number of cardiologist visits | | 0.42 (1.69) | 0.56 (1.57) | 0.44 (1.70) | 0.44 (1.34) |
| | | 0.12 (1.00) | 0.00 (1.07) | J. 1 1 (1.7 J) | 3.11(2.01) |
| Number of Internal/family medicine visits 994 (11.47) 7.64 (8.32) 8.79 (9.46) 8.79 (9.86) | | 2 65 (4 43) | 2.66 (4.09) | 2.62 (4.17) | 2.62 (4.08) |
| .mean (sd) 994 (1147) 7-64 (8.32) 8-79 (9.74) 8-79 (9.66) .mean (sd) 1.47 (2.01) 1.33 (8.77) 1.38 (1.90) 1.38 (1.88) .mean (sd) 0.46 (0.77) 0.45 (0.77) 0.45 (0.77) 0.45 (0.74) .mean (sd) 0.46 (0.77) 0.45 (0.77) 0.45 (0.74) 0.45 (0.75) .mean (sd) 0.46 (0.77) 0.45 (0.77) 0.45 (0.74) .mean (sd) 0.46 (0.77) 0.45 (0.77) 0.45 (0.74) .mean (sd) 0.46 (0.77) 0.45 (0.77) .mean (sd) 0.45 (0.78) .mean (sd) 0.46 (0.78) .mean (sd) 0.46 (0.78) .mean (sd) 0.46 (0.78) .mean (sd) 0.45 (0.78) .mean (sd) | | 2.00 (1.10) | 2.55 ( 1.55) | 2.02 ( / | 2.02 ( 3) |
| Number of electrocardiograms (ECG/EKG) | | 9.94 (11.47) | 7.64 (8.32) | 8.79 (9.74) | 8.79 (9.86) |
| mean(sd) | | 0.0 . (22 / | (0.02) | J., 0 (0., 1) | =:/ 0 (0.00) |
| Number of echocardiograms | | 1.47 (2.01) | 1.33 (1.87) | 1.38 (1.90) | 1.38 (1.88) |
| mean(sd) | | 1 (2.01) | 1100 (1107) | 2.00 (2.00) | 1.00 (1.00) |
| Out-of-pocket medication cost | | 0.46(0.77) | 0.45 (0.77) | 0.45 (0.74) | 0.45 (0.75) |
| mean(sd) | | 0.10(0.77) | 0.10 (0.1.7 | 0.10(0) | 0.10 (011 0) |
| Unique prand medicines | | 617.36 (799.68) | 710.57 (960.32) | 659.83 (853.88) | 659.83 (748.45) |
| | | | | (223.22) | |
| Unique generic medicines | | 16.12 (6.79) | 16.57 (7.33) | 16.56 (6.97) | 16.56 (6.93) |
| | | | | | , |
| Colonoscopy Sigmoildoscopy, n(%) 1,327 (9.6%) 3,581 (12.0%) 653.7 (10.8%) 653.7 (10.8%) 653.7 (10.8%) 1,942.5 (32.2%) 1,94 | | 15.85 (6.57) | 16.30 (7.11) | 16.29 (6.76) | 16.29 (6.71) |
| FluPneumococcal vaccine; n (%) | | | | | |
| Pap smear, n(%) 374 (2.7%) 1617 (5.4%) 220.4 (3.7%) 220. | | | | | |
| PSA test n (%) Fecal occult blood test; n (%) Fecal occult blood test; n (%) Fecal occult blood test; n (%) 872 (6.3%) 1183 (8.6%) 1263 (8.8%) 1283 (4.0%) 1324.0 (5.4%) 324.0 (5.4%) 324. | | | | | |
| Bone mineral density tests; n (%) | PSA test; n(%) | | | | 1,601.9 (26.6%) |
| Bone mineral density tests; n (%) | | | | | |
| Telemedicine; n(%) 1,236.9 (20.5%) 1,249 (1.38) 1,26 (1.28) 1,26 (1.28) 1,26 (1.28) 1,26 (1.28) 1,26 (1.28) 1 | Bone mineral density tests; n (%) | | | | |
| HbAlc tests | Mammograms; n(%) | | | | |
| HbAlc tests | Telemedicine; n (%) | 2,855 (20.7%) | 6,957 (23.4%) | 1,236.9 (20.5%) | 1,236.9 (20.5%) |
| Lipid panelsmean(sd) | HbA1c tests | | | | |
| Lipid panels L C mean (sd) 1.72 (1.22) 1.76 (1.23) 1.75 (1.21) 1.75 (1.21) Creatinine tests mean (sd) 3.88 (3.36) 3.42 (3.41) 3.73 (3.11) 3.73 (4.17) Natriuretic peptide tests mean (sd) 0.26 (0.78) 0.26 (0.81) 0.25 (0.76) 0.25 (0.75) Limean (sd) 1.44 (1.92) 1.23 (1.80) 1.36 (1.85) 1.36 (1.89) Combined comorbidity score mean (sd) 1.44 (1.92) 1.23 (1.80) 1.36 (1.85) 1.36 (1.89) Limean (sd) 3.64 (3.09) 2.84 (2.66) 3.26 (2.82) 3.26 (2.89) Frailty Score mean (sd) 0.20 (0.07) 0.18 (0.06) 0.19 (0.06) 0.19 (0.06) mean (sd) 0.20 (0.07) 0.18 (0.06) 0.19 (0.06) 0.19 (0.06) mean (sd) 0.42 (1.05) 0.23 (0.67) 0.30 (0.82) 0.30 (0.81) mean (sd) 0.42 (1.05) 0.23 (0.67) 0.30 (0.82) 0.30 (0.81) mean (sd) 0.42 (1.05) 0.23 (0.67) 0.30 (0.82) 0.30 (0.81) mean (sd) 0.42 (1.05) 0.23 (0.67) 0.30 | mean (sd) | 2.48 (1.34) | 2.41 (1.37) | 2.49 (1.33) | 2.49 (1.38) |
| Creatinine tests 3.88 (3.36) 3.42 (3.41) 3.73 (3.11) 3.73 (4.17) Natriuretic peptide tests 0.26 (0.78) 0.26 (0.81) 0.25 (0.76) 0.25 (0.75) Lyrine tests 1 1 1.23 (1.80) 1.36 (1.85) 1.36 (1.89) Combined comorbidity score 1 1.23 (1.80) 1.36 (1.85) 1.36 (1.89) Lyrine tests 1 1.23 (1.80) 1.36 (1.85) 1.36 (1.89) Combined comorbidity score 1 1.23 (1.80) 1.36 (1.85) 1.36 (1.89) Lyrine tests 1 1.23 (1.80) 1.36 (1.85) 1.36 (1.89) Combined comorbidity score 1.23 (1.80) 1.36 (1.85) 1.36 (1.89) Lyrine tests 1.36 (1.89) 2.84 (2.66) 3.26 (2.82) 3.26 (2.89) Frailty Score 1.36 (1.89) 2.84 (2.66) 3.26 (2.82) 3.26 (2.89) Lyrine tests 1.36 (1.89) 0.18 (0.06) 0.19 | Lipid panels | | | | |
| mean(sd) 3.88 (3.36) 3.42 (3.41) 3.73 (3.11) 3.73 (4.17) Natriuretic peptide tests | mean (sd) | 1.72 (1.22) | 1.76 (1.23) | 1.75 (1.21) | 1.75 (1.21) |
| mean(sd) 3.88 (3.36) 3.42 (3.41) 3.73 (3.11) 3.73 (4.17) Natriuretic peptide tests | Creatinine tests | | | | |
| mean(sd) 0.26 (0.78) 0.26 (0.81) 0.25 (0.76) 0.25 (0.75) Urine tests | | 3.88 (3.36) | 3.42 (3.41) | 3.73 (3.11) | 3.73 (4.17) |
| Urine tests Langer (sd) Last (1.89) Last (1.85) Last (1.89) Combined comorbidity score Last (1.92) Last (1.80) Last (1.85) Last (1.89) mean (sd) 3.64 (3.09) 2.84 (2.66) 3.26 (2.82) 3.26 (2.89) Frailty Score Earth (1.85) Last (1.85) Last (1.85) Last (1.85) 1.36 (1.89) mean (sd) 0.20 (0.07) 0.18 (0.06) 0.19 (0.06) 0.19 (0.06) 0.19 (0.06) Number of Hospitalizations 0.42 (1.05) 0.23 (0.67) 0.30 (0.82) 0.30 (0.81) Any hospitalization within prior 91 days; n (%) 1,307 (9.5%) 1,190 (4.0%) 366.2 (6.1%) 366.2 (6.1%) Any hospitalization within prior 92-365 days; n (%) 2,336 (16.9%) 3,757 (12.6%) 886.0 (14.7%) Number of hospitalizations (0,1,2 or more) 10,738 (77.9%) 25,280 (85.0%) 4,931.8 (81.8%) 4,931.8 (81.8%) | Natriuretic peptide tests | | | | |
| mean(sd) | mean (sd) | 0.26 (0.78) | 0.26 (0.81) | 0.25 (0.76) | 0.25 (0.75) |
| Combined comorbidity score 3.64 (3.09) 2.84 (2.66) 3.26 (2.82) 3.26 (2.89) Frailty Score 5.20 (0.07) 0.18 (0.06) 0.19 (0.06) 0.19 (0.06) Number of Hospitalizations 5.20 (0.07) 0.20 (0.07) 0.18 (0.06) 0.19 (0.06) Number of Hospitalization within prior 91 days; n (%) 0.42 (1.05) 0.23 (0.67) 0.30 (0.82) 0.30 (0.81) Any hospitalization within prior 91 days; n (%) 1,307 (9.5%) 1,190 (4.0%) 366.2 (6.1%) 366.2 (6.1%) Number of hospitalizations (0,1,2 or more) 2,336 (16.9%) 3,757 (12.6%) 886.0 (14.7%) Number of hospitalizations (0,1,2 or more) 10,738 (77.9%) 25,280 (85.0%) 4,931.8 (81.8%) 4,931.8 (81.8%) | | | | | |
| mean(sd) 3.64 (3.09) 2.84 (2.66) 3.26 (2.82) 3.26 (2.89) Frailty Scoremean (sd) 0.20 (0.07) 0.18 (0.06) 0.19 (0.06) 0.19 (0.06) Number of Hospitalizationsmean(sd) 0.42 (1.05) 0.23 (0.67) 0.30 (0.82) 0.30 (0.81) Any hospitalization within prior 91 days; n (%) 1,307 (9.5%) 1,190 (4.0%) 366.2 (6.1%) 366.2 (6.1%) Any hospitalization within prior 92-365 days; n (%) 2,336 (16.9%) 3,757 (12.6%) 886.0 (14.7%) Number of hospitalizations (0,1,2 or more) 2,338 (77.9%) 25,280 (85.0%) 4,931.8 (81.8%) 4,931.8 (81.8%) | mean (sd) | 1.44 (1.92) | 1.23 (1.80) | 1.36 (1.85) | 1.36 (1.89) |
| Frailty Score 0.20 (0.07) 0.18 (0.06) 0.19 (0.06) 0.19 (0.06) Number of Hospitalizations 0.42 (1.05) 0.23 (0.67) 0.30 (0.82) 0.30 (0.81) mean (sd) 0.42 (1.05) 0.23 (0.67) 0.30 (0.82) 0.30 (0.81) Any hospitalization within prior 91 days; n (%) 1,307 (9.5%) 1,190 (4.0%) 366.2 (6.1%) 366.2 (6.1%) Any hospitalization within prior 92-365 days; n (%) 2,336 (16.9%) 3,757 (12.6%) 886.0 (14.7%) 886.0 (14.7%) Number of hospitalizations (0, 1, 2 or more) 10,738 (77.9%) 25,280 (85.0%) 4,931.8 (81.8%) 4,931.8 (81.8%) | Combined comorbidity score | | | | |
| mean (sd) 0.20 (0.07) 0.18 (0.06) 0.19 | mean (sd) | 3.64 (3.09) | 2.84 (2.66) | 3.26 (2.82) | 3.26 (2.89) |
| Number of Hospitalizations 0.42 (1.05) 0.23 (0.67) 0.30 (0.82) 0.30 (0.81) Any hospitalization within prior 91 days; n (%) 1,307 (9.5%) 1,190 (4.0%) 366.2 (6.1%) 366.2 (6.1%) Any hospitalization within prior 92-365 days; n (%) 2,336 (16.9%) 3,757 (12.6%) 886.0 (14.7%) Number of hospitalizations (0, 1, 2 or more) 10,738 (77.9%) 25,280 (85.0%) 4,931.8 (81.8%) 4,931.8 (81.8%) | Frailty Score | | | | |
| Number of Hospitalizations 0.42 (1.05) 0.23 (0.67) 0.30 (0.82) 0.30 (0.81) Any hospitalization within prior 91 days; n (%) 1,307 (9.5%) 1,190 (4.0%) 366.2 (6.1%) 366.2 (6.1%) Any hospitalization within prior 92-365 days; n (%) 2,336 (16.9%) 3,757 (12.6%) 886.0 (14.7%) Number of hospitalizations (0, 1, 2 or more) 10,738 (77.9%) 25,280 (85.0%) 4,931.8 (81.8%) 4,931.8 (81.8%) | mean (sd) | 0.20 (0.07) | 0.18 (0.06) | 0.19 (0.06) | 0.19 (0.06) |
| Any hospitalization within prior 91 days; n (%) 1,307 (9.5%) 1,190 (4.0%) 366.2 (6.1%) 366.2 (6.1%) Any hospitalization within prior 92-365 days; n (%) 2,336 (16.9%) 3,757 (12.6%) 886.0 (14.7%) 886.0 (14.7%) Number of hospitalizations (0,1,2 or more) 10,738 (77.9%) 25,280 (85.0%) 4,931.8 (81.8%) 4,931.8 (81.8%) | Number of Hospitalizations | | | | |
| Any hospitalization within prior 92-365 days; n (%) Number of hospitalizations (0,1,2 or more) <1; n (%) 2,336 (16.9%) 3,757 (12.6%) 886.0 (14.7%) 886.0 (14.7%) 886.0 (14.7%) 4,931.8 (81.8%) 4,931.8 (81.8%) | mean (sd) | 0.42 (1.05) | 0.23 (0.67) | 0.30 (0.82) | 0.30 (0.81) |
| Number of hospitalizations (0,1,2 or more) | Any hospitalization within prior 91 days; n (%) | 1,307 (9.5%) | 1,190 (4.0%) | 366.2 (6.1%) | 366.2 (6.1%) |
| <1; n (%) 10,738 (77.9%) 25,280 (85.0%) 4,931.8 (81.8%) 4,931.8 (81.8%) | Any hospitalization within prior 92-365 days; n (%) | 2,336 (16.9%) | 3,757 (12.6%) | 886.0 (14.7%) | 886.0 (14.7%) |
| <1; n (%) 10,738 (77.9%) 25,280 (85.0%) 4,931.8 (81.8%) 4,931.8 (81.8%) | Number of hospitalizations (0,1,2 or more) | | | | |
| 1 - <2; n(%) | | 10,738 (77.9%) | 25,280 (85.0%) | 4,931.8 (81.8%) | 4,931.8 (81.8%) |
| | 1 - <2; n (%) | 1,709 (12.4%) | 3,139 (10.6%) | 693.2 (11.5%) | 693.2 (11.5%) |

| >= 2; n (%) | 1,346 (9.8%) | 1,325 (4.5%) | 402.4 (6.7%) | 402.4 (6.7%) |
|---|---|---|---|---|
| Heart failure hospitalization; n (%) | 978 (7.1%) | 1,473 (5.0%) | 355.2 (5.9%) | 355.2 (5.9%) |
| ED visit; n (%) | 6,077 (44.1%) | 10,116 (34.0%) | 2,419.8 (40.2%) | 2,419.8 (40.2%) |
| Acute MI; n (%) | 242 (1.8%) | 467 (1.6%) | 98.8 (1.6%) | 98.8 (1.6%) |
| Old MI; n (%) | 1,160 (8.4%) | 2,392 (8.0%) | 493.3 (8.2%) | 493.3 (8.2%) |
| Heart failure; n (%) | 3,490 (25.3%) | 6,804 (22.9%) | 1,474.1 (24.5%) | 1,474.1 (24.5%) |
| Acute heart failure; n (%) | 848 (6.1%) | 1,448 (4.9%) | 330.4 (5.5%) | 330.4 (5.5%) |
| Microalbuminuria or proteinuria; n (%) | 1,107 (8.0%) | 2,260 (7.6%) | 467.9 (7.8%) | 467.9 (7.8%) |
| Ratio of brand to generic medications | | | | |
| mean (sd) | 1.02 (0.04) | 1.01(0.03) | 1.01 (0.04) | 1.01 (0.03) |
| CED | | | | |
| 2022 | 3,157 (22.9%) | 1,553 (5.2%) | 651.5 (10.8%) | 651.5 (10.8%) |
| 2023 | 4,846 (35.1%) | 9,004 (30.3%) | 2,160.0 (35.8%) | 2,160.0 (35.8%) |
| 2024 | 4,522 (32.8%) | 13,188 (44.3%) | 2,418.1 (40.1%) | 2,418.1 (40.1%) |
| 2025 | 1,268 (9.2%) | 5,999 (20.2%) | 797.9 (13.2%) | 797.9 (13.2%) |

| MARKETSCAN | | | | |
|---|---|---|---|---|
| Variable | Reference: Sitagliptin | Exposure: Tirzepatide | Reference: Sitagliptin | Exposure: Tirzepatide |
| Number of patients | 3,825 | 5,609 | 3,825 | 5,609 |
| Sum of weights | | | 1,413.43 | 1,413.43 |
| Effective sample size | | | 2,442 | 3,375 |
| Age | | | | |
| mean (sd) | 68.34 (11.44) | 59.43 (9.10) | 63.13 (10.46) | 63.13 (9.54) |
| Gender (male); n (%) | 2,110 (55.2%) | 2,813 (50.2%) | 760.0 (53.8%) | 760.0 (53.8%) |
| Region/State | | | | |
| Northeast; n (%) | 710 (18.6%) | 571 (10.2%) | 193.6 (13.7%) | 193.6 (13.7%) |
| Widwest / North central: n(%) | 1.526 (39.9%) | 1.476 (26.3%) | 459.6 (32.5%) | 459.6 (32.5%) |
| South; n (%) | 1,432 (37.4%) | 3,261 (58.1%) | 692.9 (49.0%) | 692.9 (49.0%) |
| West: n(%) | 152 (4.0%) | 295 (5.3%) | 65.5 (4.6%) | 65.5 (4.6%) |
| Missing; n(%) | 5 (0.1%) | 6 (0.1%) | 1.8 (0.1%) | 1.8 (0.1%) |
| Smoking / Tobacco use; n (%) | 529 (13.8%) | 742 (13.2%) | 193.4 (13.7%) | 193.4 (13.7%) |
| Weight | 020 (201070) | (10.2 / 0) | 10011 (1011 70) | 100.1 (101.70) |
| Overweight; n(%) | 1,097 (28.7%) | 443 (7.9%) | 206.1 (14.6%) | 206.1 (14.6%) |
| Class 1 Obesity; n (%) | 500 (13.1%) | 457 (8.1%) | 166.4 (11.8%) | 166.4 (11.8%) |
| Class 2 Obesity; n (%) | 193 (5.0%) | 385 (6.9%) | 93.5 (6.6%) | 93.5 (6.6%) |
| Class 3 Obesity; n(%) | 547 (14.3%) | 1,102 (19.6%) | 256.2 (18.1%) | 256.2 (18.1%) |
| Unspecified Obesity; n (%) | 1,488 (38.9%) | 3,222 (57.4%) | 691.2 (48.9%) | 691.2 (48.9%) |
| Diabetic retinopathy; n (%) | 402 (10.5%) | 494 (8.8%) | 125.8 (8.9%) | 125.8 (8.9%) |
| Diabetic neuropathy; n (%) | 1,175 (30.7%) | 1,261 (22.5%) | 370.7 (26.2%) | 370.7 (26.2%) |
| Diabetic nephropathy; n(%) | 994 (26.0%) | 870 (15.5%) | 273.9 (19.4%) | 273.9 (19.4%) |
| Diabetes with other opthalmic complications; n (%) | 160 (4.2%) | 115 (2.1%) | 40.5 (2.9%) | 40.5 (2.9%) |
| Diabetes with peripheral circulatory disorders; n (%) | 642 (16.8%) | 700 (12.5%) | 196.9 (13.9%) | 196.9 (13.9%) |
| Diabetic foot: n(%) | 115 (3.0%) | 150 (2.7%) | 38.0 (2.7%) | 38.0 (2.7%) |
| Erectile dysfunction; n (%) | 182 (4.8%) | 263 (4.7%) | 65.7 (4.7%) | 65.7 (4.7%) |
| Hypoglycemia; n (%) | 748 (19.6%) | 1,102 (19.6%) | 273.4 (19.3%) | 273.4 (19.3%) |
| Hyperglycemia/DKA/HONK; n (%) | 1,954 (51.1%) | 2,858 (51.0%) | 720.5 (51.0%) | 720.5 (51.0%) |
| Skininfections; n(%) | 413 (10.8%) | 598 (10.7%) | 147.3 (10.4%) | 147.3 (10.4%) |
| Stable angina; n (%) | 282 (7.4%) | 347 (6.2%) | 95.5 (6.8%) | 95.5 (6.8%) |
| | 155 (4.1%) | 188 (3.4%) | 50.1 (3.6%) | 50.1 (3.6%) |
| Unstable angina; n (%) | 3,474 (90.8%) | 4,960 (88.4%) | 1,256.9 (88.9%) | 1,256.9 (88.9%) |
| Hypertension; n (%) | 156 (4.1%) | 119 (2.1%) | 36.1 (2.6%) | 36.1 (2.6%) |
| Hypotension; n (%) | | | | |
| Hyperlipidemia; n (%) | 3,345 (87.5%) | 4,853 (86.5%) | 1,235.0 (87.4%) | 1,235.0 (87.4%) |
| Atrial fibrillation; n (%) | 625 (16.3%) | 605 (10.8%) | 178.9 (12.7%) | 178.9 (12.7%) |
| Cardiac conduction disorder; n (%) | 317 (8.3%) | 282 (5.0%) | 83.8 (5.9%) | 83.8 (5.9%) |
| Previous cardiac procedure (CABG, PTCA, Stent); n (%) | 102 (2.7%) | 134 (2.4%) | 38.5 (2.7%) | 38.5 (2.7%) |
| Ischemic stroke; n (%) | 115 (3.0%) | 67 (1.2%) | 23.9 (1.7%) | 23.9 (1.7%) |
| PVD diagnosis or surgery; n (%) | 693 (18.1%) | 658 (11.7%) | 206.0 (14.6%) | 206.0 (14.6%) |
| Other cardiac dysrhythmia; n (%) | 1,004 (26.2%) | 1,291 (23.0%) | 327.5 (23.2%) | 327.5 (23.2%) |
| Cardiomyopathy; n (%) | 303 (7.9%) | 362 (6.5%) | 94.3 (6.7%) | 94.3 (6.7%) |
| Valve disorders; n (%) | 641 (16.8%) | 636 (11.3%) | 190.9 (13.5%) | 190.9 (13.5%) |
| Valve replacement; n (%) | 56 (1.5%) | 44 (0.8%) | 15.0 (1.1%) | 15.0 (1.1%) |
| TIA; n(%) | 160 (4.2%) | 128 (2.3%) | 39.2 (2.8%) | 39.2 (2.8%) |
| Edema; n (%) | 518 (13.5%) | 655 (11.7%) | 173.3 (12.3%) | 173.3 (12.3%) |
| Venous thromboembolism / Pulmonary embolism; n (%) | 172 (4.5%) | 191 (3.4%) | 51.6 (3.7%) | 51.6 (3.7%) |
| Pulmonary hypertension; n (%) | 138 (3.6%) | 112 (2.0%) | 30.6 (2.2%) | 30.6 (2.2%) |
| Implantable cardioverter defibrillator; n (%) | 14 (0.4%) | 18 (0.3%) | 4.4 (0.3%) | 4.4 (0.3%) |
| Hyperkalemia; n (%) | 142 (3.7%) | 85 (1.5%) | 30.4 (2.2%) | 30.4 (2.2%) |
| Coronary atherosclerosis; n (%) | 1,612 (42.1%) | 2,022 (36.0%) | 559.8 (39.6%) | 559.8 (39.6%) |
| Cerebrovascular procedure; n (%) | 8 (0.2%) | 6 (0.1%) | 2.2 (0.2%) | 2.2 (0.2%) |
| Insertion of pacemakers / removal of cardiac lead; n (%) | 11 (0.3%) | 4 (0.1%) | 1.7 (0.1%) | 1.7 (0.1%) |
| CKD stage 1-2; n (%) | 145 (3.8%) | 165 (2.9%) | 50.7 (3.6%) | 50.7 (3.6%) |
| CKD stage 3-4; n(%) | 689 (18.0%) | 493 (8.8%) | 170.0 (12.0%) | 170.0 (12.0%) |
| Unspecified CKD; n (%) | 246 (6.4%) | 170 (3.0%) | 58.5 (4.1%) | 58.5 (4.1%) |
| Acute kidney injury; n (%) | 358 (9.4%) | 213 (3.8%) | 78.0 (5.5%) | 78.0 (5.5%) |

| Hypertensive nephropathy; n (%) | 573 (15.0%) | 446 (8.0%) | 143.7 (10.2%) | 143.7 (10.2%) |
|---|---|---|---|---|
| Urinary tract infections; n (%) | 609 (15.9%) | 641 (11.4%) | 176.8 (12.5%) | 176.8 (12.5%) |
| Genital infections; n (%) | 130 (3.4%) | 167 (3.0%) | 45.7 (3.2%) | 45.7 (3.2%) |
| Urolithiasis (Kidney and urinary stone); n (%) | 207 (5.4%) | 245 (4.4%) | 69.5 (4.9%) | 69.5 (4.9%) |
| COPD: n(%) | 478 (12.5%) | 476 (8.5%) | 146.3 (10.4%) | 146.3 (10.4%) |
| Asthma: n (%) | 344 (9.0%) | 591 (10.5%) | 140.8 (10.0%) | 140.8 (10.0%) |
| Obstructive sleep apnea; n (%) | 1,001 (26.2%) | 2,193 (39.1%) | 459.1 (32.5%) | 459.1 (32.5%) |
| Serious bacterial infections; n(%) | 250 (6.5%) | 190 (3.4%) | 62.4 (4.4%) | 62.4 (4.4%) |
| Pneumonia; n (%) | 269 (7.0%) | 224 (4.0%) | 68.0 (4.8%) | 68.0 (4.8%) |
| Liver disease; n(%) | 575 (15.0%) | 879 (15.7%) | 206.8 (14.6%) | 206.8 (14.6%) |
| MASH/MASLD; n (%) | 217 (5.7%) | 501 (8.9%) | 101.2 (7.2%) | 101.2 (7.2%) |
| Fractures / Falls; n(%) | 294 (7.7%) | 206 (3.7%) | 67.5 (4.8%) | 67.5 (4.8%) |
| | 150 (3.9%) | 103 (1.8%) | | 37.9 (2.7%) |
| Osteoporosis; n (%) | 976 (25.5%) | | 37.9 (2.7%) | |
| Osteoarthritis; n (%) | | 1,354 (24.1%) | 330.4 (23.4%) | 330.4 (23.4%) |
| Depression; n (%) | 497 (13.0%) | 878 (15.7%) | 187.2 (13.3%) | 187.2 (13.3%) |
| Dementia; n (%) | 272 (7.1%) | 90 (1.6%) | 39.9 (2.8%) | 39.9 (2.8%) |
| Delirium or psychosis; n (%) | 41 (1.1%) | 26 (0.5%) | 9.3 (0.7%) | 9.3 (0.7%) |
| Anxiety; n(%) | 540 (14.1%) | 1,175 (20.9%) | 228.6 (16.2%) | 228.6 (16.2%) |
| Sleep disorders; n(%) | 939 (24.5%) | 1,593 (28.4%) | 366.3 (25.9%) | 366.3 (25.9%) |
| Anemia; n (%) | 1,009 (26.4%) | 1,094 (19.5%) | 301.8 (21.3%) | 301.8 (21.3%) |
| Influenza; n (%) | 62 (1.6%) | 142 (2.5%) | 29.3 (2.1%) | 29.3 (2.1%) |
| COVID; n (%) | 533 (13.9%) | 809 (14.4%) | 190.9 (13.5%) | 190.9 (13.5%) |
| Hyperthyroidism and other thyroid gland disorders; n (%) | 1,001 (26.2%) | 1,498 (26.7%) | 353.3 (25.0%) | 353.3 (25.0%) |
| Hypothyroidism; n (%) | 774 (20.2%) | 1,148 (20.5%) | 275.7 (19.5%) | 275.7 (19.5%) |
| Nephrotic syndrome; n (%) | 4 (0.1%) | 2 (0.0%) | 0.7 (0.1%) | 0.7 (0.1%) |
| Urinary incontinence; n (%) | 222 (5.8%) | 191 (3.4%) | 59.2 (4.2%) | 59.2 (4.2%) |
| Biliary disease; n (%) | 15 (0.4%) | 12 (0.2%) | 2.8 (0.2%) | 2.8 (0.2%) |
| Pancreatitis; n (%) | 1 (0.0%) | 4 (0.1%) | 0.8 (0.1%) | 0.8 (0.1%) |
| Bowel obstruction; n (%) | 15 (0.4%) | 11 (0.2%) | 3.0 (0.2%) | 3.0 (0.2%) |
| Gastroparesis; n (%) | 25 (0.7%) | 49 (0.9%) | 12.2 (0.9%) | 12.2 (0.9%) |
| Number of antidiabetic drugs on CED | | | | |
| mean (sd) | 1.17 (0.87) | 1.06 (0.94) | 1.17 (0.86) | 1.17 (0.94) |
| Concomitant use or initiation of Metformin; n (%) | 2,198 (57.5%) | 2,557 (45.6%) | 777.2 (55.0%) | 777.2 (55.0%) |
| Concomitant use or initiation of Insulins; n (%) | 488 (12.8%) | 1,145 (20.4%) | 226.6 (16.0%) | 226.6 (16.0%) |
| Concomitant use or initiation of Sulfonylureas; n (%) | 821 (21.5%) | 576 (10.3%) | 231.0 (16.3%) | 231.0 (16.3%) |
| Concomitant use or initiation of DPP-4i; n (%) | 35 (0.9%) | 77 (1.4%) | 16.2 (1.2%) | 16.2 (1.2%) |
| Concomitant use or initiation of SGLT-2i; n (%) | 753 (19.7%) | 1,345 (24.0%) | 332.6 (23.5%) | 332.6 (23.5%) |
| Concomitant use or initiation of Any other glucose-lowering drugs; n (%) | 186 (4.9%) | 221 (3.9%) | 68.1 (4.8%) | 68.1 (4.8%) |
| Past use of Metformin; n (%) | 2,620 (68.5%) | 3,503 (62.5%) | 959.2 (67.9%) | 959.2 (67.9%) |
| Past use of Insulins; n (%) | 739 (19.3%) | 1,495 (26.7%) | 315.6 (22.3%) | 315.6 (22.3%) |
| Past use of Sulfonylureas; n (%) | 1,197 (31.3%) | 887 (15.8%) | 333.2 (23.6%) | 333.2 (23.6%) |
| Past use of DPP-4i; n (%) | 98 (2.6%) | 112 (2.0%) | 30.3 (2.2%) | 30.3 (2.2%) |
| Past use of SGLT-2i; n (%) | 1,053 (27.5%) | 1,749 (31.2%) | 441.4 (31.2%) | 441.4 (31.2%) |
| Past use of Any other glucose-lowering drugs; n (%) | 285 (7.5%) | 309 (5.5%) | 92.2 (6.5%) | 92.2 (6.5%) |
| ACE-is/ARB's; n (%) | 2,833 (74.1%) | 3,963 (70.7%) | 1,035.3 (73.3%) | 1,035.3 (73.3%) |
| ARNI; n (%) | 104 (2.7%) | 183 (3.3%) | 37.0 (2.6%) | 37.0 (2.6%) |
| Thiazides; n (%) | 1,178 (30.8%) | 1,946 (34.7%) | 458.2 (32.4%) | 458.2 (32.4%) |
| Beta-blockers; n (%) | 2,149 (56.2%) | 2,931 (52.3%) | 765.6 (54.2%) | 765.6 (54.2%) |
| Calcium channel blockers; n (%) | 1,544 (40.4%) | 1,783 (31.8%) | 502.2 (35.5%) | 502.2 (35.5%) |
| Digoxin / Digitoxin; n (%) | 41 (1.1%) | 43 (0.8%) | 13.5 (1.0%) | 13.5 (1.0%) |
| Loop diuretics; n (%) | 791 (20.7%) | 1,019 (18.2%) | 263.9 (18.7%) | 263.9 (18.7%) |
| Other diuretics; n (%) | 331 (8.7%) | 586 (10.4%) | 127.5 (9.0%) | 127.5 (9.0%) |
| Intravenous diuretics; n (%) | 53 (1.4%) | 54 (1.0%) | 15.2 (1.1%) | 15.2 (1.1%) |
| Nitrates; n (%) | 424 (11.1%) | 543 (9.7%) | 147.2 (10.4%) | 147.2 (10.4%) |
| Anti-arrhythmics; n (%) | 136 (3.6%) | 190 (3.4%) | 49.2 (3.5%) | 49.2 (3.5%) |
| Statins; n(%) | 3,165 (82.7%) | 4,325 (77.1%) | 1,144.6 (81.0%) | 1,144.6 (81.0%) |
| PCSK9 inhibitors and other lipid-lowering drugs; n (%) | 622 (16.3%) | 985 (17.6%) | 243.0 (17.2%) | 243.0 (17.2%) |
| Antiplatelet medications; n (%) | 821 (21.5%) | 1,004 (17.9%) | 285.2 (20.2%) | 285.2 (20.2%) |
| Oral anticoagulants: n (%) | 663 (17 3%) | 713 (12 7%) | 2045 (145%) | 2045 (145%) |
| Oral anticoagulants; n (%) COPD/Asthma medications; n (%) | 663 (17.3%)<br>1,262 (33.0%) | 713 (12.7%)<br>2,160 (38.5%) | 204.5 (14.5%)<br>513.0 (36.3%) | 204.5 (14.5%)<br>513.0 (36.3%) |

| NSAIDS; n (%) | 1,077 (28.2%) | 1,891 (33.7%) | 436.3 (30.9%) | 436.3 (30.9%) |
|---|---|---|---|---|
| Oral corticosteroids; n (%) | 938 (24.5%) | 1,738 (31.0%) | 382.8 (27.1%) | 382.8 (27.1%) |
| Osteoporosis agents (incl. bisphosphonates); n (%) | 90 (2.4%) | 89 (1.6%) | 28.4 (2.0%) | 28.4 (2.0%) |
| Opioids; n (%) | 748 (19.6%) | 1,198 (21.4%) | 294.1 (20.8%) | 294.1 (20.8%) |
| Anti-depressants; n (%) | 1,090 (28.5%) | 2,150 (38.3%) | 458.2 (32.4%) | 458.2 (32.4%) |
| Antipsychotics; n(%) | 127 (3.3%) | 186 (3.3%) | 42.7 (3.0%) | 42.7 (3.0%) |
| Anxiolytics / hypnotics, benzos; n (%) | 612 (16.0%) | 1,294 (23.1%) | 276.5 (19.6%) | 276.5 (19.6%) |
| Dementia medications; n (%) | 146 (3.8%) | 34 (0.6%) | 19.1 (1.4%) | 19.1 (1.4%) |
| Jrinary tract infections antibiotics; n (%) | 1,757 (45.9%) | 2,750 (49.0%) | 658.8 (46.6%) | 658.8 (46.6%) |
| -axatives; n(%) | 115 (3.0%) | 195 (3.5%) | 44.9 (3.2%) | 44.9 (3.2%) |
| Number of distinct medications | 113 (3.0 70) | 133 (3.370) | +4.5 (S.2 70) | 44.5 (5.2 70) |
| mean (sd) | 14.08 (6.15) | 15.02 (6.65) | 14.37 (6.47) | 14.37 (6.17) |
| Number of office visits | 14.08 (0.13) | 15.02 (6.65) | 14.57 (0.47) | 14.37 (0.17) |
| | 10 F1 (7.12) | 10.05 (0.00) | 10.33 (7.10) | 10.22 (0.77) |
| .mean (sd) | 10.51 (7.12) | 10.65 (6.99) | 10.33 (7.18) | 10.33 (6.77) |
| Number of endocrinologist visits | 2.42.4.20 | 0.51.4.00) | 0.45.4.5.0 | 0.45.46.00 |
| .mean (sd) | 0.46 (1.61) | 0.51 (1.39) | 0.45 (1.54) | 0.45 (1.29) |
| Number of cardiologist visits | | | | |
| .mean (sd) | 2.54 (4.18) | 1.99 (3.41) | 2.11 (3.66) | 2.11 (3.48) |
| Number of internal/family medicine visits | | | | |
| .mean (sd) | 6.70 (7.91) | 5.41 (5.75) | 5.73 (6.20) | 5.73 (6.25) |
| Number of Electrocardiograms (ECG/EKG) | | | | |
| mean (sd) | 1.50 (1.99) | 1.20 (1.72) | 1.29 (1.71) | 1.29 (1.85) |
| Number of Echocardiograms | · /=/ | , , , | , , , | / |
| mean (sd) | 0.54 (0.93) | 0.42 (0.79) | 0.45 (0.80) | 0.45 (0.83) |
| Out-of-pocket medication cost | 0.54 (0.55) | 0.42 (0.73) | 0.43 (0.00) | 0.43 (0.83) |
| mean (sd) | 525.86 (1,080.34) | 603.48 (1,048.58) | 554.16 (1,206.55) | 554.16 (913.40) |
| | 323.80 (1,080.34) | 003.48 (1,048.38) | 334.10 (1,200.33) | 554.10 (915.40) |
| Jnique brand medicines | 1424(020) | 15 20 (6 04) | 14.63 (6.60) | 14 (2) (6 22) |
| .mean (sd) | 14.34 (6.36) | 15.28 (6.84) | 14.63 (6.69) | 14.62 (6.33) |
| Jnique generic medicines | | | | |
| mean (sd) | 14.08 (6.15) | 15.02 (6.65) | 14.37 (6.47) | 14.37 (6.17) |
| Colonoscopy Sigmoidoscopy; n (%) | 393 (10.3%) | 723 (12.9%) | 160.9 (11.4%) | 160.9 (11.4%) |
| Flu Pneumococcal vaccine; n (%) | 1,242 (32.5%) | 1,562 (27.8%) | 426.2 (30.2%) | 426.2 (30.2%) |
| Pap smear; n (%) | 181 (4.7%) | 554 (9.9%) | 97.8 (6.9%) | 97.8 (6.9%) |
| PSA test; n(%) | 1,046 (27.3%) | 1,546 (27.6%) | 404.9 (28.6%) | 404.9 (28.6%) |
| Fecal occult blood test; n(%) | 180 (4.7%) | 233 (4.2%) | 63.5 (4.5%) | 63.5 (4.5%) |
| Bone mineral density tests; n (%) | 188 (4.9%) | 285 (5.1%) | 70.5 (5.0%) | 70.5 (5.0%) |
| Mammograms: n (%) | 702 (18.4%) | 1,473 (26.3%) | 323.2 (22.9%) | 323.2 (22.9%) |
| Telemedicine; n (%) | 969 (25.3%) | 1,736 (31.0%) | 389.1 (27.5%) | 389.1 (27.5%) |
| HbA1C tests | 303 (23.370) | 1,7 30 (31.0 70) | 303.1 (27.370) | 303.1 (27.370) |
| mean (sd) | 2.14 (1.52) | 2.30 (1.81) | 2.26 (1.50) | 2.26 (1.52) |
| Lipid panels | 2.14 (1.32) | 2.50 (1.81) | 2.20(1.30) | 2.20 (1.32) |
| | 1 FF (1 21) | 172 (124) | 1.00 (1.22) | 1.00 (1.20) |
| mean (sd) | 1.55 (1.31) | 1.72 (1.34) | 1.66 (1.32) | 1.66 (1.29) |
| Creatinine tests | 0.00 (0.44) | 0.04(0.07) | 0.00(0.00) | 0.06 (0.33) |
| mean (sd) | 0.08 (0.44) | 0.04 (0.27) | 0.06 (0.34) | 0.06 (0.32) |
| Natriuretic peptide tests | | | | |
| .mean (sd) | 0.20 (0.80) | 0.20 (0.99) | 0.20 (0.86) | 0.20 (0.93) |
| Jrine tests | | | | |
| .mean (sd) | 1.23 (1.91) | 1.08 (1.88) | 1.13 (1.74) | 1.13 (1.84) |
| Combined comorbidity score | | | | |
| .mean (sd) | 2.64 (2.81) | 1.70 (2.01) | 1.98 (2.30) | 1.98 (2.23) |
| Frailty Score | ì | , | | |
| mean (sd) | 0.18 (0.06) | 0.16 (0.04) | 0.17 (0.05) | 0.17 (0.05) |
| Number of Hospitalizations | === (0.00) | | (5/ | () |
| .mean (sd) | 11.51 (35.04) | 5.80 (24.31) | 7.25 (25.65) | 7.25 (27.50) |
| | | | | 60.5 (4.3%) |
| Any hospitalization within prior 91 days; n (%) | 272 (7.1%) | 160 (2.9%) | 60.5 (4.3%) | |
| Any hospitalization within prior 92-365 days; n (%) | 548 (14.3%) | 486 (8.7%) | 140.7 (10.0%) | 140.7 (10.0%) |
| | 0.004 (0.0.00): | E 0.4 E (0.0 40() | | |
| .<1; n(%) | 3,091 (80.8%) | 5,017 (89.4%) | 1,229.0 (87.0%) | 1,229.0 (87.0%) |
| Number of hospitalizations (0,1,2 or more)<br><1; n (%)<br>1 - <2; n (%)<br>>= 2; n (%) | 3,091 (80.8%)<br>32 (0.8%)<br>702 (18.4%) | 5,017 (89.4%)<br>30 (0.5%)<br>562 (10.0%) | 1,229.0 (87.0%)<br>9.1 (0.7%)<br>175.3 (12.4%) | 1,229.0 (87.0%)<br>9.1 (0.7%)<br>175.3 (12.4%) |

| Heart failure hospitalization; n (%) | 247 (6.5%) | 164 (2.9%) | 54.8 (3.9%) | 54.8 (3.9%) |
|---|---|---|---|---|
| ED visit; n(%) | 1,601 (41.9%) | 2,012 (35.9%) | 518.1 (36.7%) | 518.1 (36.7%) |
| Acute MI; n (%) | 90 (2.4%) | 97 (1.7%) | 28.6 (2.0%) | 28.6 (2.0%) |
| Old MI; n (%) | 169 (4.4%) | 212 (3.8%) | 60.2 (4.3%) | 60.2 (4.3%) |
| Heart failure; n (%) | 704 (18.4%) | 665 (11.9%) | 194.8 (13.8%) | 194.8 (13.8%) |
| Acute heart failure; n (%) | 192 (5.0%) | 149 (2.7%) | 47.1 (3.3%) | 47.1 (3.3%) |
| Microalbuminuria or proteinuria; n (%) | 190 (5.0%) | 208 (3.7%) | 62.1 (4.4%) | 62.1 (4.4%) |
| Ratio of brand to generic medications | | | | |
| mean (sd) | 1.02 (0.04) | 1.02 (0.04) | 1.02 (0.04) | 1.02 (0.04) |
| CED | | | | |
| 2022 | 1,611 (42.1%) | 940 (16.8%) | 399.6 (28.3%) | 399.6 (28.3%) |
| 2023 | 2,214 (57.9%) | 4,669 (83.2%) | 1,013.9 (71.7%) | 1,013.9 (71.7%) |

Variable\_name Algorithm sources Age Gender Race If region not available, from State, https://www2.census.gov/geo/pdfs/maps-Region data/maps/reference/us\_regdiv.pdf Investigator review of codes based on: https://dev.sentinelsystem.org/projects/AP/repos/sentinelanalytic-packages/browse?at=refs%2Fheads%2Fcder\_mpl2p\_wp015, https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analyticpackages/browse?at=refs%2Fheads%2Fcder\_sir\_wp002, https://pubmed.ncbi.nlm.nih.gov/34953068/, https://www.ncbi.nlm.nih.gov/pmc/articles/PMC9154288/, Smoking / Tobacco use https://www.ncbi.nlm.nih.gov/pmc/articles/PMC3721171/ Underweight Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34338404/ Normal weight, if BMI is 20.0-24.9 Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34338404/ Overweight, if BMI is 25.0 to 29.9 Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34338404/ Class 1 (low-risk) obesity, if BMI is 30.0 to 34.9 Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34338404/ Class 2 (moderate-risk) obesity, if BMI is 35.0 to 39.9 Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34338404/ Class 3 (high-risk) obesity if BMI is equal to or greater than 40 Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34338404/ Unspecified obesity Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34338404/ Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34953068/, Diabetic retinopathy https://pubmed.ncbi.nlm.nih.gov/35043165/ Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34953068/, Diabetic neuropathy https://pubmed.ncbi.nlm.nih.gov/35043165/ Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/35043165/ Diabetic nephropathy Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34953068/, ICD9 to ICD10 Diabetes with other opthalmic complications conversion Investigator review of codes based on: https://www.ncbi.nlm.nih.gov/books/NBK368403/table/sb203.t5/, https://www.health.mil/Reference-Center/Publications/2016/03/01/Diabetes-Mellitus, http://www.icd9data.com/2014/Volume1/240-Diabetes with peripheral circulatory disorders 279/249-259/250/default.htm, https://www.icd10data.com/ICD10CM/Codes/E00-E89/E08-E13/E11-Diabetic foot Investigator review of codes based on: (modified codes) https://pubmed.ncbi.nlm.nih.gov/36102675/ Investigator review of codes based on: the paper then used ICD9/ICD10 website to expand it, https://www.icd10data.com/ICD10CM/Codes/N00-N99/N40-N53/N52-, Erectile dysfuntion https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4857901/ Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34953068/, https://pubmed.ncbi.nlm.nih.gov/35043165/ Hypoglycemia Investigator review of codes based on: Hyperglycemia: https://pubmed.ncbi.nlm.nih.gov/34953068/, https://pubmed.ncbi.nlm.nih.gov/35043165/ DKA: https://pubmed.ncbi.nlm.nih.gov/29773640/, https://pubmed.ncbi.nlm.nih.gov/38262528/ HONK: https://dam.assets.ohio.gov/image/upload/medicaid.ohio.gov/Providers/PaymentInnovation/DEF/DK Hyperglycemia/DKA/HONK Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34953068/ , ICD9 to ICD10 Skin infections conversion Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/19337843/, https://pmc.ncbi.nlm.nih.gov/articles/PMC9172873/ Stable angina Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/19337843/, Unstable angina https://pmc.ncbi.nlm.nih.gov/articles/PMC9172873/ Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/35043165/, https://www.ncbi.nlm.nih.gov/pmc/articles/PMC8929186/ Hypertension Hypotension Investigator review of codes based on: https://pmc.ncbi.nlm.nih.gov/articles/PMC8064679/ Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/35043165/, https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analyticpackages/browse?at=refs%2Fheads%2Fcder\_sir\_wp002, https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analyticpackages/browse?at=refs%2Fheads%2Fcder\_mpl2p\_wp015 Hyperlipidemia Atrial fibrillation Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/31933524/ Acute myocardial infarction Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/24682186/ Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/24682186/ Old myocardial infarction Investigator review of codes based on: https://stacks.cdc.gov/view/cdc/31381/cdc\_31381\_DS8.pdf, https://www.health.ny.gov/health\_care/medicaid/redesign/dsrip/vbp\_library/docs/arrblk.pdf,

https://www.cdc.gov/dhdsp/maps/atlas/data-sources.html,

to ICD10 conversion

Cardiac conduction disorder

https://www.cms.gov/medicare/coding/icd10/downloads/icd10clinicalconceptscardiology1.pdf, ICD9

Previous cardiac procedure (CABG, PTCA, Stent) Modified codes based on eligibility criteria, here we implement any care setting, any diagnosis position Modified codes based on eligibility criteria, here we implement any care setting, any diagnosis position Ischemic stroke Investigator review of codes, https://www.icd10data.com/ PVD diagnosis or surgery  $Investigator\ review\ of\ codes\ based\ on:\ https://stacks.cdc.gov/view/cdc/31381/cdc\_31381\_DS8.pdf,$ https://www.health.ny.gov/health\_care/medicaid/redesign/dsrip/vbp\_library/docs/arrblk.pdf, https://www.cdc.gov/dhdsp/maps/atlas/data-sources.html, https://www.cms.gov/medicare/coding/icd10/downloads/icd10clinicalconceptscardiology1.pdf, ICD9 Other cardiac dysrhythmia to ICD10 conversion Heart failure Investigator review of codes Acute heart failure Investigator review of codes Microalbuminuria/proteinuria Modified codes based on inclusion criteria, here we implement any care setting, any diagnosis position Investigator review of codes based on: https://dev.sentinelsystem.org/projects/AP/repos/sentinel-Cardiomyopathy analytic-packages/browse?at=refs%2Fheads%2Fcder\_mpl2p\_wp015 Investigator review of codes based on: https://stacks.cdc.gov/view/cdc/31381/cdc\_31381\_DS8.pdf, https://pubmed.ncbi.nlm.nih.gov/38440888/, https://www.ncbi.nlm.nih.gov/pmc/articles/PMC8751938/, https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analyticpackages/browse?at=refs%2Fheads%2Fcder\_mpl2p\_wp015 https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-Valve disorders packages/browse?at=cder\_mpl2p\_wp009 Valve replacement Modified codes based on eligibility criteria, here we implement any care setting, any diagnosis position TIA Modified codes based on eligibility criteria, here we implement any care setting, any diagnosis position Investigator review of codes based on: https://www.cms.gov/medicare-coveragedatabase/view/article.aspx?articleid=52993&ver=45& Edema Investigator review of codes based on: https://www.sciencedirect.com/science/article/pii/S2666572723000251 Venous thromboembolism/ pulmonary embolsim Pulmonary hypertension Investigator review of codes Implantable cardioverter defibrillator Modified codes based on eligibility criteria, here we implement any care setting, any diagnosis position Hyperkalemia https://pmc.ncbi.nlm.nih.gov/articles/PMC4399109/ Coronary atherosclerosis Investigator review of codes based on: https://pmc.ncbi.nlm.nih.gov/articles/PMC10251803/ Cerebrovascular procedure Investigator review of codes, https://www.icd10data.com/ Modified codes based on eligibility criteria, here we implement any care setting, any diagnosis position Insertion of pacemakers / removal of cardiac lead CKD stage 1-2 Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/35043165/ CKD stage 3-4 Investigator review of codes based on: https://pmc.ncbi.nlm.nih.gov/articles/PMC2978782/ Unspecified CKD Investigator review of codes based on: https://pmc.ncbi.nlm.nih.gov/articles/PMC5888226/ Acute kidney injury Investigator review of codes based on: https://www.ncbi.nlm.nih.gov/pmc/articles/PMC8929186/ Investigator review of codes based on: https://nccd.cdc.gov/ckd/Methods.aspx?Qnum=Q637, https://www.kidneymedicinejournal.org/cms/10.1016/j.xkme.2022.100414/attachment/5e29ab67-7a7d-4621-9af3-81bd071bbc67/mmc1.pdf, https://www.icd10data.com/ICD10CM/Codes/I00-I99 Hypertensive nephropathy Investigator reviewed code based on: https://pmc.ncbi.nlm.nih.gov/articles/PMC7558992/#app1-Urinary tract infections antibiotics-09-00536 Genital infections Investigator reviewed codes based on: https://pubmed.ncbi.nlm.nih.gov/30207042/

Urolithiasis (kidney or urinary stones)

COPD

Asthma

Obstructive sleep apnea

Serious bacterial infections

Pneumonia

Investigator review of codes based on: https://pmc.ncbi.nlm.nih.gov/articles/PMC7793999/

Investigator review of codes based on: https://www.ncbi.nlm.nih.gov/pmc/articles/PMC10203971/

Investigator review of codes based on: https://www.ncbi.nlm.nih.gov/pmc/articles/PMC10203971/, modified CCW algorithm (any care setting, any diagnosis position)

Investigator review of codes based on: https://www.ncbi.nlm.nih.gov/pmc/articles/PMC8636332/, https://www.ncbi.nlm.nih.gov/pmc/articles/PMC7927325/

https://pubmed.ncbi.nlm.nih.gov/29921683/, https://pubmed.ncbi.nlm.nih.gov/17346615/,

https://pubmed.ncbi.nlm.nih.gov/23335588/

Investigator review of codes based on: https://www.ncbi.nlm.nih.gov/pmc/articles/PMC10203971/

https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-

packages/browse?at=refs%2Fheads%2Fcder\_sir\_wp002,

https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-

packages/browse?at=refs%2Fheads%2Fcder\_mpl2p\_wp015, Modified algorightm from

https://pubmed.ncbi.nlm.nih.gov/34256144/, Modified CCW algorithm Investigator review of codes: https://pubmed.ncbi.nlm.nih.gov/32300995/\_

https://pubmed.ncbi.nlm.nih.gov/39316292/

https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-packages/browse?at=refs%2Fheads%2Fcder\_mpl2p\_wp015, https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-packages/browseppengages/bro

packages/browse?at=cder\_mpl2p\_wp009,

https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-packages/browse?at=refs%2Fheads%2Fcder\_mpl2p\_wp015, https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-

packages/browse?at=cder mpl2p wp010

https://www.ncbi.nlm.nih.gov/pmc/articles/PMC8202643/,

https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-packages/browse?at=refs%2Fheads%2Fcder\_sir\_wp002, CCW Algorithms

Modified CCW algorithm

https://pubmed.ncbi.nlm.nih.gov/35043165/, CCW Algorithms

https://pubmed.ncbi.nlm.nih.gov/35043165/,

https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-packages/browse?at=refs%2Fheads%2Fcder\_mpl2p\_wp015

https://pubmed.ncbi.nlm.nih.gov/28485014/, https://pubmed.ncbi.nlm.nih.gov/35043165/

https://pubmed.ncbi.nlm.nih.gov/35043165/

Investigator review of codes based on https://www.verywellhealth.com/sleeping-disorders-list-and-

diagnostic-codes-3014779

Modified codes based on eligibility criteria, here we implement any care setting, any diagnosis position

Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/38556924/

https://pubmed.ncbi.nlm.nih.gov/34913208/,

https://www.ncbi.nlm.nih.gov/pmc/articles/PMC8427377/

 $\underline{Investigator\ review\ of\ codes\ based\ on:\ https://www.cms.gov/icd10m/version37-fullcode-particles.}$ 

cms/fullcode\_cms/P0244.html

Investigator review of codes based on: https://pmc.ncbi.nlm.nih.gov/articles/PMC10478599/

Investigator review of codes based on: https://nccd.cdc.gov/ckd/Methods.aspx?Qnum=Q637, https://www.cms.gov/icd10m/FY2024-nprmversion41.0-fullcode-cms/fullcode\_cms/P2401.html <a href="mailto:lnvestigator.review.of.codes">lnvestigator.review.of.codes</a> based on: https://pubmed.ncbi.nlm.nih.gov/38527324/

Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/37796527/,

 $Investigator\ review\ of\ codes: \underline{https://pubmed.ncbi.nlm.nih.gov/36222554/,}$ 

https://pubmed.ncbi.nlm.nih.gov/30287807/, https://pubmed.ncbi.nlm.nih.gov/22262606/ Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/36798959/, https://pubmed.ncbi.nlm.nih.gov/28438588/, https://pubmed.ncbi.nlm.nih.gov/31095068/

Investigator review of codes: https://pubmed.ncbi.nlm.nih.gov/34624355/

Investigator review of codes

Investigator review of codes, https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK518983/
Investigator review of codes, https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK278938/
Investigator review of codes, https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK513225/

Investigator review of codes, https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK542331/

Investigator review of codes, https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK576405/

Investigator review of codes, https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK551656/, https://pmc.ncbi.nlm.nih.gov/articles/PMC4882495/,

https://www.ncbi.nlm.nih.gov/books/NBK557848/

Investigator review of codes, https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK518983/ Investigator review of codes. https://www.drugs.com.

https://www.ncbi.nlm.nih.gov/books/NBK278938/ Investigator review of codes, https://www.drugs.com,

https://www.ncbi.nlm.nih.gov/books/NBK513225/

Liver disease

MASH/MASLD

Fractures / Falls

Osteoporosis Osteoarthritis Depression

Dementia

Delirium or psychosis

Anxiety

Sleep disorder

Anemia Influenza

COVID-19

Hyperthyroidism and other thyroid gland disorders

Hypothyroidism

Nephrotic syndrome Urinary incontinence

Biliary disease

Pancreatitis

Bowel obstruction

Gastroparesis Number of antidiabetic drugs on CED

Number of articulabetic drugs of CED

Concomitant use or initiation of metformin

Concomitant use or initiation of insulin

Concomitant use or initiation of sulfonylureas

Concomitant use or initiation of DPP4i except sitagliptin

Concomitant use or initiation of SGLT2i

Concomitant use or initiation of other glucose-lowering drugs

Past use of metformin

Past use of insulin

Past use of sulfonylureas

Past use of DPP4i except sitagliptin https://www.ncbi.nlm.nih.gov/books/NBK542331/

Investigator review of codes, https://www.drugs.com,
Past use of SGLT2i https://www.ncbi.nlm.nih.gov/books/NBK576405/

https://www.ncbi.nlm.nih.gov/books/NBK576405/ Investigator review of codes, https://www.drugs.com,

> https://www.ncbi.nlm.nih.gov/books/NBK551656/, https://pmc.ncbi.nlm.nih.gov/articles/PMC4882495/,

Investigator review of codes, https://www.drugs.com.

Past use of other glucose-lowering drugs https://www.ncbi.nlm.nih.gov/books/NBK557848/

Investigator review of codes, https://www.drugs.com,

ACEI / ARB https://www.ncbi.nlm.nih.gov/books/NBK9626/table/A66/ Investigator review of codes, https://www.drugs.com,

ARNI https://www.ncbi.nlm.nih.gov/books/NBK507904/ Investigator review of codes, https://www.drugs.com,

Thiazides https://www.ncbi.nlm.nih.gov/books/NBK9626/table/A66/ Investigator review of codes, https://www.drugs.com,

Beta-Blockers https://www.ncbi.nlm.nih.gov/books/NBK9626/table/A66/
Investigator review of codes, https://www.drugs.com.

Calcium channel blockers https://www.ncbi.nlm.nih.gov/books/NBK9626/table/A66/lnvestigator review of codes, https://www.drugs.com,

Investigator review of codes, https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK556025/

Digoxin / Digitoxin https://pubchem.ncbi.nlm.nih.gov/compound/441207 Investigator review of codes, https://www.drugs.com,
Loop diuretics https://www.ncbi.nlm.nih.gov/books/NBK9626/table/A66/

Investigator review of codes, https://www.drugs.com,
Other diuretics https://www.ncbi.nlm.nih.gov/books/NBK9626/table/A66/
Intravenous diuretics Investigator review of codes

Investigator review of codes, https://www.drugs.com,

Nitrates https://www.ncbi.nlm.nih.gov/books/NBK9626/table/A66/
Investigator review of codes, https://www.drugs.com,

https://www.ncbi.nlm.nih.gov/books/NBK482322/ (using class I and class II as class 2 is beta blockers

and class 4 is calcium channel blockers)

Investigator review of codes, https://www.drugs.com, https://www.heart.org/en/health-topics/cholesterol/prevention-and-treatment-of-high-cholesterol-hyperlipidemia/cholesterol-

Statins medications

Investigator review of codes, https://www.drugs.com, https://www.heart.org/en/health-topics/cholesterol/prevention-and-treatment-of-high-cholesterol-hyperlipidemia/cholesterol-

PCSK9 inhibitors and other lipid-lowering drugs medications

Investigator review of codes, https://www.drugs.com,
Antiplatelet agents https://www.ncbi.nlm.nih.gov/books/NBK537062/
Investigator review of codes, https://www.drugs.com,

Oral anticoagulants https://www.ahajournals.org/doi/full/10.1161/JAHA.120.017559

Investigator review of codes, https://www.copdfoundation.org/Learn-More/I-am-a-Person-with-

COPD/Asthma medication COPD/Treatments-Medications.aspx, https://getasthmahelp.org/medications-list.aspx Investigator review of codes, https://www.drugs.com,

NSAIDs https://www.ncbi.nlm.nih.gov/books/NBK547742/

Investigator review of codes, https://www.drugs.com, https://www.aaaai.org/tools-for-the-public/drug-

Oral corticosteroids guide/oral-corticosteroid-medications

Investigator review of codes based on: https://www.drugs.com,

Osteoporosis agents (incl. bisphosphonates) https://www.ncbi.nlm.nih.gov/books/NBK470248/
Investigator review of codes, https://www.drugs.com.

https://pubmed.ncbi.nlm.nih.gov/31643200/#:~:text=They%20can%20also%20be%20informally,%2

Opioids C%20codeine%2C%20oxycodone%2C%20hydrocodone%2C Investigator review of codes, https://www.drugs.com,

Anti-depressants https://www.ncbi.nlm.nih.gov/books/NBK538182/
Antipsychotics Investigator review of codes, https://www.drugs.com

Investigator review of codes, https://www.drugs.com, https://www.dea.gov/sites/default/files/2020-

06/Benzodiazepenes-2020.pdf, https://www.ncbi.nlm.nih.gov/books/NBK470159/,

Anxiolytics/hypnotics, benzodiazepines <a href="https://www.drugs.com">https://www.drugs.com</a>

Investigator review of codes based on: https://www.drugs.com,

https://www.ncbi.nlm.nih.gov/pmc/articles/PMC7462122/, https://go.drugbank.com/drugs/DB00382

https://pubmed.ncbi.nlm.nih.gov/35790044/

Investigator review of codes, https://www.drugs.com

N/A

https://www.cms.gov/files/document/mm13473-how-use-office-and-outpatient-evaluation-and-management-visit-complexity-add-code-g2211.pdf, https://www.cms.gov/files/document/physician-fee-schedule-pfs-payment-officeoutpatient-evaluation-and-management-em-visits-fact-sheet.pdf

Number of distinct medications, median (iqr), mean (sd)

Medication for dementia

Urinary tract infections antibiotics

Anti-arrhythmics

Number of office visits median (iqr), mean (sd)

Data dictionary of Optum, Marketscan and https://www.cms.gov/Medicare/Provider-Enrollment-and-

Certification/MedicareProviderSupEnroll/downloads/taxonomy.pdf,

https://www.cms.gov/medicare/provider-enrollment-and-

certification/medicareprovidersupenroll/downloads/taxonomycrosswalk.pdf Number of endocrinologist visits, median (igr), mean (sd)

Data dictionary of Optum, Marketscan and https://www.cms.gov/Medicare/Provider-Enrollment-and-

Certification/MedicareProviderSupEnroll/downloads/taxonomv.pdf.

https://www.cms.gov/medicare/provider-enrollment-and-

Number of cardiologist visits, median (iqr), mean (sd) certification/medicareprovidersupenroll/downloads/taxonomycrosswalk.pdf

Data dictionary of Optum, Marketscan and https://www.cms.gov/Medicare/Provider-Enrollment-and-

Certification/Medicare Provider Sup Enroll/downloads/taxonomy.pdf,

https://www.cms.gov/medicare/provider-enrollment-and-

Number of internal medicine/family medicine visits, median (iqr), mean (sd. certification/medicareprovidersupenroll/downloads/taxonomycrosswalk.pdf

https://www.cms.gov/medicare-coverage-database/view/article.aspx?articleId=57326,

https://firstcoastbillinggroup.com/ekg-billing-and-reimbursement/.

https://www.aapc.com/codes/coding-newsletters/my-cardiology-coding-alert/cpt-answer-5-common-

ecg-coding-questions-175952-article Number of electrocardiograms, median (iqr), mean (sd)

https://www.ncbi.nlm.nih.gov/pmc/articles/PMC8511132/,

https://pubmed.ncbi.nlm.nih.gov/34778785/, https://www.cms.gov/medicare-coverage-

database/view/article.aspx?articleid=56625&ver=27&,

Number of echocardiograms, median (igr), mean (sd) https://www.medicalbillgurus.com/echocardiogram-cpt-code/

Pharmacy out-of-pocket cost, median (iqr), mean (sd)

Unique brand medications Investigator review of codes, https://www.drugs.com Investigator review of codes, https://www.drugs.com Unique generic medications Ratio of unique brand to generic medications Investigator review of codes, https://www.drugs.com

https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-

packages/browse?at=refs%2Fheads%2Fcder\_sir\_wp002 Colonoscopy/ Sigmoidoscopy

https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-

packages/browse?at=refs%2Fheads%2Fcder\_sir\_wp002, https://www.cms.gov/medicare-coverage-

database/view/article.aspx?articleId=54767&DocID=A54767, https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-

packages/browse?at=refs%2Fheads%2Fcder\_sir\_wp002, https://www.cms.gov/medicare-coverage-

Flu vaccine / Pneumococcal vaccine database/view/article.aspx?articleId=54767&DocID=A54767

https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-

packages/browse?at=refs%2Fheads%2Fcder\_sir\_wp002,

http://www.icd9data.com/2012/Volume1/V01-V91/V70-V82/V72/default.htm, http://www.icd9data.com/2012/Volume1/V01-V91/V70-V82/V76/default.htm

https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-

PSA test packages/browse?at=refs%2Fheads%2Fcder\_sir\_wp002

Fecal occult blood test Investigator review of codes

Bone mineral density tests

Pap smear test

Investigator review of codes based on: https://dev.sentinelsystem.org/projects/AP/repos/sentinel-

analytic-packages/browse?at=refs%2Fheads%2Fcder\_sir\_wp002, https://www.cms.gov/medicare-

coverage-database/view/article.aspx?articleid=56448&ver=16&bc=0,

http://www.icd9data.com/2012/Volume1/V01-V91/V70-V82/V76/default.htm Mammograms

Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/33151319/,

https://www.cms.gov/newsroom/fact-sheets/medicare-telemedicine-health-care-provider-factsheet, https://www.aafp.org/family-physician/practice-and-career/getting-paid/coding/coding-

Telemedicine telehealth-audio-virtual-digital-visits.html

Number of HbA1c tests, median (igr), mean (sd) https://pubmed.ncbi.nlm.nih.gov/34953068/ Number of lipid panels, median (igr), mean (sd) https://pubmed.ncbi.nlm.nih.gov/34953068/ https://pubmed.ncbi.nlm.nih.gov/34953068/ Number of creatinine tests, median (igr), mean (sd)

Number of natriuretic peptide tests, median (igr), mean (sd) Investigator review of codes Number of urine tests, median (iqr), mean (sd) Investigator review of codes

HbA1c N/A Glucose N/A Creatinine N/A Systolic blood pressure N/A Heart rate N/A вмі N/A eGFR N/A LDL N/A HDL N/A Total cholesterol N/Δ Triglycerides

A combined comorbidity score predicted mortality in elderly patients better than existing scores,

https://pubmed.ncbi.nlm.nih.gov/21208778/

Measuring Frailty in Medicare Data: Development and Validation of a Claims-Based Frailty Index,

https://pubmed.ncbi.nlm.nih.gov/29244057/

Number of any hospitalization, median (igr), mean (sd) N/A Any hospitalization within prior 90 days; n (%) N/A

Combined comorbidity score

Any hospitalization within prior 91-365 days; n (%) 0, 1, >1 hospitalizations (any)

Hospitalization for heart failure; n (%)

N/A N/A N/A

Different in all 3 databases and measure already created in all 3 as well;

ED visit (Medicare): Revenue center codes: 0450, 0451, 0452, 0456, 0459, 0981; Place of service:

ED visit (Optum): Place of service: 23

 $ED\ visit\ (Marketscan): Service\ sub-category\ codes: 10120, 10220, 10320, 10420, 10520, 12220,$ 20120, 20220, 21120, 21220, 22120, 22320, 30120, 30220, 30320, 30420, 30520, 30620, 31120,

31220, 31320, 31420, 31520, 31620; Place of service: 23

Number of emergency department visit median (iqr), mean (sd) Calendar year